CLINICAL TRIAL: NCT01186744
Title: A Phase 3, Multi-Site, Randomized, Mixed-Blind, Parallel-Group Treatment Withdrawal And Re-Treatment Study Of The Efficacy And Safety Of 2 Oral Doses Of CP-690,550 In Subjects With Moderate To Severe Chronic Plaque Psoriasis
Brief Title: A Study To Evaluate The Effects And Safety Of Treatment, Treatment Withdrawal, Followed By Re-Treatment With CP-690,550 In Subjects With Moderate To Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921111
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Psoriasis
Keywords: OPT Retreatment; OPT; chronic; moderate; severe; treatment; safety; treatment withdrawal; retreatment; retreatment withdrawal; CP-690,550; Psoriasis Vulgaris; Plaque Psoriasis; tofacitinib; Xeljanz; nail psoriasis; Jak-inhibitor; oral treatment; Pruritus; Itch; DLQI; rebound; intermittent; retreat
MeSH Terms: conditions — Psoriasis; Bronchiolitis Obliterans Syndrome; Lymphoma, Follicular; Pruritus | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active Treatment (10 mg) BID / Placebo BID (Experimental): Continuous active treatment (CP-690,550) for 24 weeks, followed by treatment withdrawal (placebo treatment) for 4-16 weeks, followed by active treatment (CP-690,550) for 16-28 weeks
  Interventions: Drug: CP-690,550
- Active Treatment (10 mg) BID (Experimental): Continuous active treatment (CP-690,550) for 56 weeks
  Interventions: Drug: CP-690,550
- Active Treatment (5 mg) BID / Placebo BID (Experimental): Continuous active treatment (CP-690,550) for 24 weeks, followed by treatment withdrawal (placebo treatment) for 4-16 weeks, followed by active treatment (CP-690,550) for 16-28 weeks
  Interventions: Drug: CP-690,550
- Active Treatment (5 mg) BID (Experimental): Continuous active treatment (CP-690,550) for 56 weeks
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — 10 mg of CP-690,550 oral BID or placebo oral BID, as appropriate based on treatment withdrawal/retreatment design
  Arms: Active Treatment (10 mg) BID / Placebo BID
Drug: CP-690,550 — 10 mg oral BID
  Arms: Active Treatment (10 mg) BID
Drug: CP-690,550 — 5 mg of CP-690,550 oral BID or Placebo oral BID, as appropriate based on treatment withdrawal/retreatment design
  Arms: Active Treatment (5 mg) BID / Placebo BID
Drug: CP-690,550 — 5 mg oral BID
  Arms: Active Treatment (5 mg) BID

SUMMARY:
The primary objectives of the study are to 1) compare the efficacy responses of CP 690,550 (5 mg BID and 10 mg BID) versus placebo following 24 weeks of CP 690,550 treatment and subsequent withdrawal of active treatment at various timepoints during the 16 week double blind active or placebo treatment period; 2) evaluate the regain of efficacy responses of CP 690,550 (5 mg BID and 10 mg BID) following 4 -16 weeks of CP 690,550 treatment withdrawal and subsequent re treatment; and 3) evaluate the safety and tolerability of CP 690,550 (5 mg BID and 10 mg BID) in subjects with moderate to severe chronic plaque psoriasis who are candidates for systemic therapy or phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with diagnosis of plaque-type psoriasis (psoriasis vulgaris) for at least 12 months prior to first dose of study drug;
* Psoriasis Area and Severity Index (PASI) score of 12 or greater, AND Physician's Global Assessment (PGA) score of 3 (moderate) or 4 (severe); Psoriasis covering at least 10% of body surface area;
* No evidence of active or latent or inadequately treated infection with Tuberculosis or other serious infections.

Exclusion Criteria:

* Non-plaque or drug induced forms of psoriasis;
* Cannot discontinue current oral, injectable or topical therapy for psoriasis or cannot discontinue phototherapy (Psoralen Ultraviolet A; Ultraviolet B).
* Any uncontrolled significant medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (87):
- United States (50):
  - Horizon Research Group, Inc., Mobile, Alabama
  - Radiant Research, Inc., Tucson, Arizona
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Associates In Research, Inc., Fresno, California
  - Dermatology Research Associates, Los Angeles, California
  - Expresscare Medical, Los Angeles, California
  - Dermatology Specialists, Inc., Oceanside, California
  - University of California San Francisco, San Francisco, California
  - Longmont Clinic, PC, Longmont, Colorado
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Florida Academic Dermatology Center, Miami, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Park Avenue Dermatology, PA, Orange Park, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Miami Research Associates, South Miami, Florida
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Springfield Clinic, LLP, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - DMIA, Louisville, Kentucky
  - DermResearch, PLLC, Louisville, Kentucky
  - Quest Diagnostics, Louisville, Kentucky
  - Northeast Dermatology Associates, Beverly, Massachusetts
  - ActivMed Practices and Research, Inc., Haverhill, Massachusetts
  - Michigan Center for Research Corporation dba Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Dermatology Consulting Services, High Point, North Carolina
  - Dermatology Associates, Wilmington, North Carolina
  - New Hanover Medical Group, PA, Wilmington, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - PMG Research of Wilmington LLC, Wilmington, North Carolina
  - Piedmont Imaging, Winston-Salem, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Triad Dermatology, PA, Winston-Salem, North Carolina
  - Jewish Hospital, Cincinnati, Ohio
  - Radiant Research, Inc., Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical Research South, LLC, Charleston, South Carolina
  - Office of Marta T. Hampton, MD, Charleston, South Carolina
  - Dermatology & Laser Center of Charleston, Charleston, South Carolina
  - Office of John Michael Humeniuk, MD, Greer, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - Dermatology Research Associates, Nashville, Tennessee
  - Office of Stephen Miller, MD, PA, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Argentina (3):
  - Centro de Investigaciones Dermatologicas, Buenos Aires, C1114aap
  - Centro de Investigaciones Dermatologicas, Buenos Aires
  - IMAI (Instituto Medico de Asistencia e Investigaciones), Buenos Aires
- Australia (6):
  - Dr. Glenn & Partners, Kogarah, New South Wales
  - Premier Dermatology, Kogarah, New South Wales
  - Skin and Cancer Foundation, Carlton, Victoria
  - Uniradiology, Carlton, Victoria
  - Malvern Diagnostic Imaging, Malvern, Victoria
  - Emeritus Research, Malvern East, Victoria
- Brazil (2):
  - Instituto de Dermatologia e Est�ca do Brasil LTDA - IDERJ, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
- Bulgaria (5):
  - Universitetska Mnogoprofilna Bolnitsa Za Aktivno Lechenie- Dr Georgi Stranski- Pleven, Pleven
  - Tsentar za kozhno-venericheski zaboliavania� EOOD, Sofia
  - Mnogoprofilna Bolnitsa Za Aktivno Lechenie- Tokuda Bolnitsa Sofia- Sofia, Sofia
  - Universitetska mnogoprofilna bolnitsa za aktivno lechenie- Alexandrovska- Sofia, Sofia
  - MBAL na Voennomeditsinska akademia- Sofia, Sofia
- Canada (8):
  - Derm Research @ 888 Inc., Vancouver, British Columbia
  - UBC Department of Dermatology and Skin Science, Vancouver, British Columbia
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - NewLab Clinical Research Inc., St. John's, Newfoundland and Labrador
  - Dermatrials Research, Hamilton, Ontario
  - Windsor Clinical Research, Windsor, Ontario
  - Innovaderm Research Inc, Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec, Quebec
- Denmark (3):
  - Department of Dermatology, Aarhus University Hospital, Aarhus C
  - Gentofte Hospital, Hellerup
  - Hudklinikken, Svendborg
- Tampere University Hospital, Department of Dermatology and Venreology, Tampere, Finland
- Greece (3):
  - Dermatology Department, Andreas Sygros Hospital, Aathens
  - University Hospital of Ioannina/Dermatology Department, Ioannina
  - "Papageorgiou" General Hospital / B' Dermatology and Venereology Clinic of University of Thessalonik, Thessaloniki
- PT & R, Beek, Netherlands
- Slovakia (2):
  - Univerzitna Nemocnica, Bratislava, Bratislava
  - Fakultna Nemocnica Trnava, Trnava
- United Kingdom (3):
  - Whipps Cross University Hospital, Department of Dermatology, London, Leytonstone
  - Department of Dermatology, Nuneaton, Warwickshire
  - Salford Royal NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Bissonnette R, Iversen L, Sofen H, Griffiths CE, Foley P, Romiti R, Bachinsky M, Rottinghaus ST, Tan H, Proulx J, Valdez H, Gupta P, Mallbris L, Wolk R. Tofacitinib withdrawal and retreatment in moderate-to-severe chronic plaque psoriasis: a randomized controlled trial. Br J Dermatol. 2015;172(5):1395-406. doi: 10.1111/bjd.13551. Epub 2015 Apr 2. PMID 25418186
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921111&StudyName=A%20Phase%203%2C%20Multi-Site%2C%20Randomized%2C%20Mixed-Blind%2C%20Parallel-Group%20Treatment%20Withdrawal%20And%20Re-Treatment%20Study%20Of%20The%20Efficacy%20And%20Safety%20Of%202%20Oral%20Doses%20Of%20CP-690%2C550%20In%20Subjects%20With%20Moderate%20To%20Severe%20Chronic%20Plaque%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 5 mg BID (Period A): Participants received CP-690,550 5 milligram (mg) tablets orally twice daily (BID) for up to 24 continuous weeks during Period A (Initial Treatment)
- CP-690,550 10 mg BID (Period A): Participants received CP-690,550 10 mg tablets orally BID for up to 24 continuous weeks during Period A (Initial Treatment)
- CP-690,550 5 mg/CP-690,550 5 mg/CP-690,550 5 mg: Participants received CP-690,550 5 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by CP-690,550 5 mg tablets orally BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 5 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- CP-690,550 5 mg/Placebo/CP-690,550 5 mg: Participants received CP-690,550 5 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 5 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- CP-690,550 10 mg/CP-690,550 10 mg/CP-690,550 10 mg: Participants received CP-690,550 10 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by CP-690,550 10 mg tablets orally BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 10 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- CP-690,550 10 mg / Placebo / CP-690,550 10 mg: Participants received CP-690,550 10 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 10 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
Period: Overall Study
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A) | CP-690,550 5 mg/CP-690,550 5 mg/CP-690,550 5 mg | CP-690,550 5 mg/Placebo/CP-690,550 5 mg | CP-690,550 10 mg/CP-690,550 10 mg/CP-690,550 10 mg | CP-690,550 10 mg / Placebo / CP-690,550 10 mg
Started | 218 | 157 | 31 | 82 | 45 | 133
Completed | 10 | 5 | 25 | 70 | 39 | 107
Not Completed | 208 | 152 | 6 | 12 | 6 | 26
Not completed — Lack of Efficacy | 156 | 99 | 0 | 2 | 2 | 5
Not completed — Protocol Violation | 1 | 2 | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 15 | 16 | 2 | 1 | 1 | 4
Not completed — Screen failure | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 14 | 10 | 2 | 5 | 0 | 6
Not completed — Study terminated by Sponsor | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 9 | 10 | 1 | 2 | 1 | 5
Not completed — Adverse Event | 10 | 14 | 1 | 0 | 1 | 4
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized at baseline and received at least one dose of the randomized investigational drug (CP-690,550 5 mg BID or 10 mg BID) during Period A.
Groups:
- CP-690,550 5 mg BID (Period A): Participants received CP-690,550 5 milligram (mg) tablets orally twice daily (BID) for 24 continuous weeks during Period A (Initial Treatment)
- CP-690,550 10 mg BID (Period A): Participants received CP-690,550 10 mg tablets orally BID for 24 continuous weeks during Period A (Initial Treatment)
- CP-690,550 10 mg / Placebo / CP-690,550 10 mg: Participants received CP-690,550 10 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 10 mg tablets orally BID or up to 28 weeks in Period C (Double-Blind Re-Treatment)
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A) | CP-690,550 5 mg/CP-690,550 5 mg/CP-690,550 5 mg | CP-690,550 5 mg/Placebo/CP-690,550 5 mg | CP-690,550 10 mg/CP-690,550 10 mg/CP-690,550 10 mg | CP-690,550 10 mg / Placebo / CP-690,550 10 mg | Total
Number analyzed (Participants) | 218 | 157 | 31 | 82 | 45 | 133 | 666
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (13.0) | 45.6 (12.6) | 44.3 (13.0) | 45.2 (13.4) | 48.5 (14.8) | 46.1 (13.4) | 44.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 50 | 11 | 27 | 11 | 44 | 208
  Male | 153 | 107 | 20 | 55 | 34 | 89 | 458

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining a Psoriasis Area and Severity Index 75 (PASI75) Response During the Double-Blind Treatment Withdrawal Period (Period B)
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percent of body surface area (BSA) affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI75 response defined as at least a 75 percent (%) reduction in PASI relative to baseline.
Time Frame: Weeks 4, 8 12, and 16 (Period B)
Population: The Period B-Full Analysis Set (FAS-B) included all participants who were re-randomized at the end of Period A and received at least 1dose of investigational drug (CP-690,550 5 mg BID or 10 mg BID) or placebo at the beginning of Period B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CP-690,550 5 mg (Period B): Participants received CP-690,550 5 mg tablets orally BID for 24 continuous weeks during Period A (Initial Treatment) followed by CP690-550 5 mg for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
- Placebo for CP-690,550 5 mg (Period B): Participants received CP-690,550 5 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
- CP-690,550 10 mg (Period B): Participants received CP-690,550 10 mg tablets orally BID for 24 continuous weeks during Period A (Initial Treatment) followed by CP-690,550 10 mg BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
- Placebo for 10 mg CP-690,550: Participants received CP-690,550 10 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
Arm/Group | CP-690,550 5 mg (Period B) | Placebo for CP-690,550 5 mg (Period B) | CP-690,550 10 mg (Period B) | Placebo for 10 mg CP-690,550
Number analyzed (Participants) | 31 | 82 | 45 | 132
percentage of participants
  Week 4 | 90.3 [72.9 to 96.8] | 63.4 [52.0 to 72.8] | 91.1 [78.0 to 96.6] | 61.4 [52.5 to 69.1]
  Week 8 | 70.3 [50.6 to 83.3] | 36.2 [25.8 to 46.7] | 86.6 [72.5 to 93.7] | 39.6 [31.2 to 47.9]
  Week 12 | 63.2 [43.4 to 77.7] | 32.4 [22.4 to 42.7] | 77.2 [61.7 to 87.0] | 33.4 [25.4 to 41.5]
  Week 16 | 56.2 [36.7 to 71.8] | 23.3 [14.7 to 33.1] | 62.3 [45.8 to 75.0] | 26.1 [18.8 to 33.9]
Statistical Analysis 1: Comparison: CP-690,550 5 mg (Period B) vs Placebo for CP-690,550 5 mg (Period B); Test type: Superiority or Other; p = 0.0008, Log Rank
Statistical Analysis 2: Comparison: CP-690,550 10 mg (Period B) vs Placebo for 10 mg CP-690,550; Test type: Superiority or Other; p < 0.0001, Log Rank

2. Primary Outcome: Percentage of Participants Maintaining a Physician's Global Assessment (PGA) Response During the Double-Blind Treatment Withdrawal (Period B)
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response defined as 0 (clear) or 1 (almost clear).
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CP-690,550 5 mg BID (Period B): Participants received CP-690,550 5 mg tablets orally BID for 24 continuous weeks during Period A (Initial Treatment) followed by CP-690,550 5 mg BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
- CP-690,550 10 mg BID (Period B): Participants received CP-690,550 10 mg tablets orally BID for 24 continuous weeks during Period A (Initial Treatment) followed by CP-690,550 10 mg BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for CP-690,550 5 mg (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550
Number analyzed (Participants) | 31 | 82 | 45 | 132
percentage of participants
  Week 4 | 80.6 [61.9 to 90.8] | 57.3 [45.9 to 67.2] | 80.0 [65.1 to 89.1] | 52.3 [43.4 to 60.4]
  Week 8 | 67.7 [48.4 to 81.2] | 34.4 [24.2 to 44.8] | 80.0 [65.1 to 89.1] | 32.5 [24.6 to 40.6]
  Week 12 | 60.6 [41.1 to 75.4] | 26.7 [17.6 to 36.8] | 66.3 [50.4 to 78.1] | 23.8 [16.8 to 31.4]
  Week 16 | 49.9 [31.0 to 66.2] | 22.9 [14.4 to 32.6] | 63.9 [48.0 to 76.1] | 18.0 [11.9 to 25.2]
Statistical Analysis 1: Comparison: CP-690,550 5 mg BID (Period B) vs Placebo for CP-690,550 5 mg (Period B); Test type: Superiority or Other; p = 0.0027, Log Rank
Statistical Analysis 2: Comparison: CP-690,550 10 mg BID (Period B) vs Placebo for 10 mg CP-690,550; Test type: Superiority or Other; p < 0.0001, Log Rank

3. Primary Outcome: Percentage of Participants Achieving a PASI75 Response During CP-690,550 Re-Treatment (Period C) Among Those Who Had a Greater Than (>)50% Reduction of Visit A4/Week 24 PASI Response During Double-Blind Treatment Withdrawal (Period B)
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percent of BSA affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. PASI75 response is defined as at least 75% reduction in PASI relative to Baseline/Day 1. Baseline defined as the last observation up to first dosing date in Period C. PASI responses at each period were relative to Baseline-A, where Baseline-A was defined as the last observation up to first dosing date in Period A.
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CP-690,550 5 mg BID / CP-690,550 5 mg BID; CP-690,550 10 mg BID / CP-690,550 10 mg BID: Participants received CP-690,550 5 mg tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 5 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- Placebo BID / CP-690,550 5 mg BID; Placebo BID / CP-690,550 10 mg BID: Participants placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 5 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 2 | 38 | 3 | 59
percentage of participants
  Baseline | 50.00 [0.00 to 100.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 4 | 100.00 [100.00 to 100.00] | 13.16 [2.41 to 23.91] | 0.00 [0.00 to 0.00] | 40.68 [28.14 to 53.21]
  Week 8 | 100.00 [100.00 to 100.00] | 31.58 [16.80 to 46.36] | 0.00 [0.00 to 0.00] | 49.15 [36.40 to 61.91]
  Week 16 | 50.00 [0.00 to 100.00] | 31.58 [16.80 to 46.36] | 0.00 [0.00 to 0.00] | 50.85 [38.09 to 63.60]

4. Primary Outcome: Percentage of Participants Achieving a PGA Response of Clear or Almost Clear During CP-690,550 Re-treatment (Period C) Among Participants Who Had a PGA of Mild, Moderate, or Severe During Double-Blind Treatment Withdrawal (Period B)
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe).
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: The Period C-Full Analysis Set (FAS-C) included all FAS-B participants who were advanced to the re-treatment period (Period C) during the 16 weeks of Period B and had received at least one dose of investigational drug (CP-690,550 5 mg BID or 10 mg BID) during Period C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo BID / CP-690,550 5 mg BID: Participants received placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 5 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- CP-690,550 10 mg BID / CP-690,550 10 mg BID: Participants received CP-690,550 10 mg tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 10 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- Placebo BID / CP-690,550 10 mg BID: Participants received placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 10 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 13 | 58 | 15 | 98
percentage of participants
  Baseline | 23.08 [0.17 to 45.98] | 5.17 [0.0 to 10.87] | 6.67 [0.0 to 19.29] | 7.14 [2.04 to 12.24]
  Week 4 | 23.08 [0.17 to 45.98] | 25.86 [14.59 to 37.13] | 33.33 [9.48 to 57.19] | 51.02 [41.12 to 60.92]
  Week 8 | 30.77 [5.68 to 55.86] | 39.66 [27.07 to 52.24] | 40.0 [15.21 to 64.79] | 55.10 [45.25 to 64.95]
  Week 16 | 30.77 [5.68 to 55.86] | 41.38 [28.70 to 54.05] | 53.33 [28.09 to 78.58] | 48.98 [39.08 to 58.88]

5. Secondary Outcome: Median Time to PASI75 Response During Initial CP-690,550 Treatment (Period A)
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percent of BSA affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. PASI75 response defined as 75% reduction in PASI relative to baseline.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: The Period A-Full Analysis Set (FAS-A) included all participants who were randomized at baseline and received at least 1 dose of the randomized investigational drug (CP-690,550 5mg BID or 10 mg BID) during Period A.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- CP-690,550 5 mg (Period A): Participants received CP-690,550 5 mg tablets orally BID for 24 continuous weeks during Period A (Initial Treatment)
Arm/Group | CP-690,550 5 mg (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 330 | 333
weeks | 24.3 [24.1 to 24.6] | 8.7 [8.1 to 15.4]

6. Secondary Outcome: Median Time to PGA Response of Clear or Almost Clear During Initial CP-690,550 Treatment (Period A)
Description: as for outcome 2
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 329 | 333
weeks | 24.1 [16.6 to 24.4] | 8.1 [NA to NA] — 95% confidence interval cannot be estimated due to less than (<)50% of events occurring and/or censoring issue.

7. Secondary Outcome: Percentage of Participants Achieving Both a PASI50-75 Response and Dermatology Life Quality Index (DLQI) ≤5 Response During Initial CP-690,550 Treatment (Period A)
Description: PASI50-75 response defined as a reduction of at least 50% but less than 75%. The DLQI is a general dermatology questionnaire that consists of 10 items that assess participant health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment. The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
percentage of participants
  Week 4 | 12.69 [9.10 to 16.27] | 21.19 [16.82 to 25.57]
  Week 8 | 18.73 [14.53 to 22.93] | 19.40 [15.17 to 23.64]
  Week 16 | 18.13 [13.98 to 22.28] | 13.13 [9.52 to 16.75]
  Week 24 | 10.88 [7.52 to 14.23] | 10.15 [6.92 to 13.38]

8. Secondary Outcome: Percentage of Participant Maintaining an Adequate Response During the Double-Blind Treatment Withdrawal (Period B)
Description: Adequate response defined as >50% reduction of the Visit A4/Week 24 (last visit in Period A) PASI response.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CP-690,550 5 mg (Period B): Participants received CP-690,550 5 mg tablets orally BID for 24 continuous weeks during Period A (Initial Treatment) followed by CP-690,550 5 mg BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
- Placebo for 5 mg CP-690,550 (Period B): Participants received CP-690,550 5 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
- Placebo for 10 mg CP-690,550 BID (Period B): Participants received CP-690,550 10 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
Arm/Group | CP-690,550 5 mg (Period B) | Placebo for 5 mg CP-690,550 (Period B) | CP-690,550 10 mg (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 132
percentage of participants
  Week 4 | 100.0 [100.0 to 100.0] | 90.0 [81.0 to 94.9] | 100.0 [100.0 to 100.0] | 85.9 [78.6 to 90.9]
  Week 8 | 96.7 [78.6 to 99.5] | 72.0 [60.6 to 80.6] | 97.7 [84.6 to 99.7] | 68.4 [59.5 to 75.7]
  Week 12 | 96.7 [78.6 to 99.5] | 58.8 [47.0 to 68.8] | 93.0 [79.9 to 97.7] | 58.5 [49.4 to 66.6]
  Week 16 | 92.3 [72.1 to 98.0] | 32.8 [16.3 to 50.4] | 93.0 [79.9 to 97.7] | 42.9 [30.5 to 54.6]

9. Secondary Outcome: Median Time to Loss of Adequate Response During the Double-Blind Treatment Withdrawal (Period B)
Description: Adequate response defined as >50% reduction of the Visit A4/Week 24 (last visit in Period A) PASI response.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg (Period B) | Placebo for 5 mg CP-690,550 (Period B) | CP-690,550 10 mg (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
weeks | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 16.4 [12.6 to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 16.1 [14.1 to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue.

10. Secondary Outcome: Percentage of Participants With PASI Score ≥125% of Baseline-A or New Type of Psoriasis (Pustular, Erythrodermic) During the Period Between Week 24 and Week 32 (Period B)
Description: The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI responses at each period are relative to Baseline-A where Baseline-A was defined as the last observation up to first dosing date in Period A. Weeks 4 and 8 are relative to the Period B baseline and are the same as Weeks 28 and 32, which are relative to Period A baseline. 95% confidence interval is constructed using the normal approximation to the binomial distribution of two-sample proportion.
Time Frame: Weeks 4 and 8 (Period B)
Population: FAS-B; Overall number (n) indicates the total number of participants with PASI Score ≥125% of baseline at least once during Weeks 4 to 8 of Period B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 (Period B) | CP-690,550 10 mg (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 44 | 132
percentage of participants
  Week 4 (n=30,82,43,128) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 8 (n=31,70,43,106) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Overall (n=31,82,44,132) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

11. Secondary Outcome: Percentage of Participants With PASI Score ≥125% of Baseline-A or New Type of Psoriasis (Pustular, Erythrodermic) During the Double-Blind Treatment Withdrawal (Period B)
Description: The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI responses at each period are relative to Baseline-A where Baseline-A was defined as the last observation up to first dosing date in Period A. 95% confidence interval is constructed using the normal approximation to the binomial distribution of two-sample proportion.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; Overall number (n) indicates the total number of participants with PASI Score ≥125% of baseline at least once during Weeks 4 to 16 of Period B.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 (Period B) | CP-690,550 10 mg (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 132
percentage of participants
  Week 4 (n=30,82,43,128) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 8 (n=31,70,43,106) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 12 (n=30,53,43,87) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 1.15 [-3.39 to 1.09]
  Week 16 (n=28,45,38,72) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Overall (n=31,82,45,132) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.76 [0.00 to 0.00]

12. Secondary Outcome: Percentage of Participants Maintaining Adequate PASI Response and Maintaining PGA Response (Clear or Almost Clear) During the Double-Blind Treatment Withdrawal (Period B)
Description: Adequate PASI response defined as less than or equal to 50% reduction of the Visit A4/Week 24 PASI Response.
Time Frame: Week 24 (Period A) and Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo for 5 mg CP-690,550 BID (Period B): Participants received CP-690,550 5 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 132
percentage of participants
  Week 4 | 100.00 [100.0 to 100.0] | 90.0 [81.0 to 94.9] | 100.0 [100.0 to 100.0] | 85.9 [78.6 to 90.9]
  Week 8 | 96.7 [78.6 to 99.5] | 72.0 [60.6 to 80.6] | 97.7 [84.6 to 99.7] | 68.4 [59.5 to 75.7]
  Week 12 | 96.7 [78.6 to 99.5] | 58.8 [47.0 to 68.8] | 93.0 [79.9 to 97.7] | 58.4 [49.3 to 66.5]
  Week 16 | 92.3 [72.1 to 98.0] | 32.8 [16.3 to 50.4] | 93.0 [79.9 to 97.7] | 43.5 [31.0 to 55.3]

13. Secondary Outcome: Median Time to Loss of >50% of the Visit A4/Week 24 PASI Response and Loss of PGA Response (Clear or Almost Clear) During the Double-Blind Treatment Withdrawal (Period B)
Time Frame: Week 24 (Period A) and Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 132
weeks | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 16.4 [12.6 to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 16.1 [14.1 to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue.

14. Secondary Outcome: Percentage of Participants Regaining PASI75 and PGA Response (Clear or Almost Clear) During CP-690,550 Re-Treatment (Period C) Among Participants Who Lost Both PASI75 Response and PGA Response (Clear or Almost Clear) at the Beginning of Period C
Description: PASI75 response defined as at least a 75% reduction in PASI relative to baseline.
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CP-690,550 5 mg BID / CP-690,550 5 mg BID: Participants received CP-690,550 5 mg tablets orally BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 5 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- Placebo BID / CP-690,550 5 mg BID: Participants received placebo tablets orally BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 5 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- CP-690,550 10 mg BID / CP-690,550 10 mg BID: Participants received CP-690,550 10 mg tablets orally BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 10 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- Placebo BID / CP-690,550 10 mg BID: Participants received placebo tablets orally BID for 4, 8, 12, or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 10 mg tablets orally BID for up to 28 weeks in Period C (Double-Blind Re-Treatment)
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 7 | 52 | 7 | 81
percentage of participants
  Week 4 | 14.3 [2.1 to 66.6] | 7.7 [3.0 to 19.2] | 14.3 [2.1 to 66.6] | 37.0 [27.6 to 48.5]
  Week 8 | 28.6 [8.0 to 74.2] | 32.3 [21.2 to 47.3] | 42.9 [16.3 to 82.8] | 48.5 [38.2 to 60.0]
  Week 16 | 64.3 [22.0 to 98.6] | 100.0 [NA to NA] — 95% confidence interval could not be estimated due to censoring. | 42.9 [16.3 to 82.8] | 57.2 [46.2 to 68.8]

15. Secondary Outcome: Median Time to Regain PASI75 and PGA Response (Clear or Almost Clear) During CP-690,550 Re-Treatment (Period C) Among Participants Who Lost Both PASI75 Response and PGA Response (Clear or Almost Clear) at the Beginning of Period C
Description: PASI75 response defined as at least a 75% reduction in PASI relative to baseline.
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 7 | 52 | 7 | 81
weeks | 16.4 [8.6 to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 16.4 [16.1 to 17.3] | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 12.4 [7.6 to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue.

16. Secondary Outcome: Percentage of Participants Regaining PASI75 and PGA Response (PGA of Clear or Almost Clear) During CP-690,550 Re-Treatment (Period C) Who Had Lost Both PASI75 Response and PGA Response at the Beginning of Period C
Description: PASI75 response defined as at least a 75% reduction in PASI relative to baseline. PASI responses at each period are relative to Baseline-A, where Baseline-A is defined as the last observation up to first dosing date in Period A. 95% confidence interval constructed using the normal approximation to the binomial distribution of one-sample proportion.
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 7 | 52 | 7 | 81
percentage of participants
  Baseline | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 4 | 14.29 [0.00 to 40.21] | 7.69 [0.45 to 14.93] | 14.29 [0.00 to 40.21] | 37.04 [26.52 to 47.55]
  Week 8 | 28.57 [0.00 to 62.04] | 28.85 [16.53 to 41.16] | 42.86 [6.2 to 79.52] | 41.98 [31.23 to 52.72]
  Week 16 | 28.57 [0.00 to 62.04] | 21.15 [10.05 to 32.25] | 42.86 [6.20 to 79.52] | 41.98 [31.23 to 52.72]

17. Secondary Outcome: Median Time to PASI75 Response During CP-690,550 Re-Treatment (Period C) For Those Who Had a >50% Reduction of Visit A4/Week 24 PASI Response During Double-Blind Treatment Withdrawal (Period B)
Description: PASI75 response defined as at least a 75% reduction in PASI relative to baseline.
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 2 | 38 | 3 | 59
weeks | 4.5 [4.3 to 4.7] | 16.4 [16.1 to 17.3] | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 8.1 [5.9 to 16.1]

18. Secondary Outcome: Median Time to PGA Response of Clear or Almost Clear During CP-690,550 Re-Treatment (Period C) Among Participants Who Had a PGA of Mild, Moderate, or Severe at the Beginning of Period C
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 10 | 55 | 14 | 91
weeks | 16.3 [16.1 to 16.4] | 16.1 [8.4 to 16.6] | 13.1 [6.0 to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 8.1 [5.0 to 16.1]

19. Secondary Outcome: Percentage of Participants With a PASI75 Response During the Initial CP-690,550 Treatment (Period A)
Description: PASI75 response defined as at least a 75% reduction in PASI relative to baseline. Baseline defined as the last observation up to the first dosing date in Period A. 95% confidence interval is constructed using the normal approximation to the binomial distribution of one-sample proportion.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
percentage of participants
  Week 4 | 7.85 [4.96 to 10.75] | 22.39 [17.92 to 26.85]
  Week 8 | 23.87 [19.27 to 28.46] | 50.45 [45.09 to 55.80]
  Week 16 | 38.07 [32.84 to 43.30] | 60.60 [55.36 to 65.83]
  Week 24 | 38.97 [33.72 to 44.23] | 59.40 [54.14 to 64.66]

20. Secondary Outcome: Percentage of Participants With a PASI75 Response During Double-Blind Withdrawal Treatment (Period B)
Description: PASI75 response defined as at least a 75% reduction in PASI relative to baseline. PASI responses in each period are relative to Baseline-A, where Baseline-A is defined as the last observation until first dosing date in Period A. 95% confidence interval is constructed using the normal approximation to the binomial distribution of one-sample proportion.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
percentage of participants
  Week 4 | 87.10 [7.94 to 39.43] | 63.41 [0.00 to 0.00] | 86.67 [14.29 to 40.24] | 59.40 [0.00 to 0.00]
  Week 8 | 70.97 [17.83 to 55.81] | 34.15 [0.00 to 0.00] | 86.67 [35.40 to 61.24] | 38.35 [0.00 to 0.00]
  Week 12 | 67.74 [18.02 to 56.49] | 30.49 [0.00 to 0.00] | 77.78 [29.38 to 58.51] | 33.83 [0.00 to 0.00]
  Week 16 | 64.52 [20.89 to 59.36] | 24.39 [0.00 to 0.00] | 62.22 [18.32 to 50.49] | 27.82 [0.00 to 0.00]

21. Secondary Outcome: Percentage of Participants With a PASI75 Response During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 20
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
percentage of participants
  Week 4 | 70.37 [53.15 to 87.59] | 34.67 [23.90 to 45.44] | 73.81 [60.51 to 87.11] | 60.83 [52.10 to 69.57]
  Week 8 | 62.96 [44.75 to 81.18] | 48.00 [36.69 to 59.31] | 66.67 [52.41 to 80.92] | 68.33 [60.01 to 76.66]
  Week 16 | 55.56 [36.81 to 74.30] | 45.33 [34.07 to 56.60] | 69.05 [55.07 to 83.03] | 61.67 [52.97 to 70.37]

22. Secondary Outcome: Percentage of Participants With PGA Response of Clear or Almost Clear During the Initial CP-690,550 Treatment (Period A)
Description: PGA response was defined as 0 (clear) or 1 (almost clear) on a 5-point scale where 0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe. 95% confidence interval is constructed using the normal approximation to the binomial distribution of one-sample proportion.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
percentage of participants
  Week 4 | 14.20 [10.44 to 17.96] | 37.91 [32.72 to 43.11]
  Week 8 | 30.51 [25.55 to 35.47] | 54.03 [48.69 to 59.37]
  Week 16 | 37.16 [31.95 to 42.37] | 58.81 [53.54 to 64.08]
  Week 24 | 37.16 [31.95 to 42.37] | 55.22 [49.90 to 60.55]

23. Secondary Outcome: Percentage of Participants With PGA Response of Clear or Almost Clear During Double-Blind Withdrawal Treatment (Period B)
Description: PGA response was defined as 0 (clear) or 1 (almost clear) on a 5-point scale where 0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe. 95% confidence interval is constructed using the normal approximation to the binomial distribution of two-sample proportion.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
percentage of participants
  Week 4 | 77.42 [1.90 to 38.30] | 57.32 [0.00 to 0.00] | 77.78 [14.84 to 44.48] | 48.12 [0.00 to 0.00]
  Week 8 | 74.19 [22.81 to 59.73] | 32.93 [0.00 to 0.00] | 82.22 [35.40 to 62.88] | 33.08 [0.00 to 0.00]
  Week 12 | 70.97 [24.21 to 61.62] | 28.05 [0.00 to 0.00] | 66.67 [24.68 to 56.09] | 26.32 [0.00 to 0.00]
  Week 16 | 58.06 [10.11 to 49.92] | 28.05 [0.00 to 0.00] | 62.22 [25.40 to 56.94] | 21.05 [0.00 to 0.00]

24. Secondary Outcome: Percentage of Participants With PGA Response of Clear or Almost Clear During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 22
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
percentage of participants
  Week 4 | 62.96 [44.75 to 81.18] | 40.00 [28.91 to 51.09] | 61.90 [47.22 to 76.59] | 59.17 [50.37 to 67.96]
  Week 8 | 62.96 [44.75 to 81.18] | 49.33 [38.02 to 60.65] | 54.76 [39.71 to 69.81] | 63.33 [54.71 to 71.96]
  Week 16 | 55.56 [36.81 to 74.30] | 49.33 [38.02 to 60.65] | 59.52 [44.68 to 74.37] | 55.00 [46.10 to 63.90]

25. Secondary Outcome: Mean Total Percent of Psoriatic Body Surface Area (BSA) During Initial CP-690,550 Treatment (Period A)
Description: Assessment of BSA with psoriasis performed separately for 4 body regions: head and neck, upper limbs, trunk (including axillae and groin), and lower limbs (including buttocks). The %surface area with psoriasis was estimated by means of the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumb together) represented approximately 1% of the total BSA. The number of handprints of psoriatic skin in a body region was used to determine the extent (%) to which a body region was involved with psoriasis.
Time Frame: Baseline and Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A; n equals the number of participants with an observation.
Measure: Mean (Standard Error); unit: percent psoriatic BSA
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
percent psoriatic BSA
  Baseline (n=331,335) | 27.5 (0.9) | 27.2 (0.9)
  Week 4 (n=326,331) | 22.3 (0.9) | 18.1 (0.8)
  Week 8 (n=322,323) | 17.2 (0.9) | 12.1 (0.8)
  Week 16 (n=311,306) | 13.3 (0.8) | 8.1 (0.7)
  Week 24 (n=277,279) | 12.0 (0.8) | 6.4 (0.7)

26. Secondary Outcome: Mean Total Percent of Psoriatic BSA During Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 25
Time Frame: Baseline and Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: percent psoriatic BSA
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
percent psoriatic BSA
  Baseline (n=31,82,45,133) | 1.9 (0.4) | 3.8 (0.8) | 2.0 (0.3) | 2.7 (0.4)
  Week 4 (n=30,82,43,128) | 1.9 (0.4) | 6.1 (0.8) | 1.8 (0.4) | 6.8 (0.9)
  Week 8 (n=30,70,43,104) | 2.2 (0.4) | 7.7 (1.2) | 2.0 (0.4) | 8.7 (1.2)
  Week 12 (n=28,53,42,84) | 2.0 (0.4) | 7.2 (1.0) | 2.3 (0.5) | 6.2 (0.9)
  Week 16 (n=28,45,38,70) | 2.2 (0.5) | 6.0 (0.9) | 2.6 (0.7) | 6.0 (0.8)

27. Secondary Outcome: Mean Total Percent of Psoriatic BSA During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 25
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: percent psoriatic BSA
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
percent psoriatic BSA
  Baseline (n=27,75,42,120) | 2.3 (0.5) | 11.4 (1.3) | 3.0 (0.8) | 12.0 (1.2)
  Week 4 (n=27,74,42,119) | 2.1 (0.4) | 10.6 (1.7) | 3.1 (0.9) | 7.2 (0.9)
  Week 8 (n=26,72,41,118) | 2.5 (0.5) | 9.0 (1.6) | 3.3 (1.0) | 6.1 (0.8)
  Week 16 (n=23,67,39,101) | 2.9 (0.5) | 7.1 (1.2) | 3.7 (1.3) | 4.5 (0.8)

28. Secondary Outcome: Mean Change From Baseline in Total Percent of Psoriatic BSA During Initial CP-690,550 Treatment (Period A)
Description: Baseline defined as the last observation up to first dosing date in Period A.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: percent change in psoriatic BSA
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 326 | 331
percent change in psoriatic BSA
  Week 4 (n=326,331) | -5.3 (0.5) | -9.0 (0.7)
  Week 8 (n=322,323) | -10.4 (0.7) | -14.5 (0.8)
  Week 16 (n=311,306) | -14.4 (0.8) | -18.5 (0.9)
  Week 24 (n=277,279) | -15.2 (0.9) | -19.4 (0.9)

29. Secondary Outcome: Mean Change From Baseline in Total Percent of Psoriatic BSA During Double-Blind Treatment Withdrawal (Period B)
Description: Baseline defined as the last observation up to first dosing date in Period B.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: percent change in psoriatic BSA
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 30 | 82 | 43 | 128
percent change in psoriatic BSA
  Week 4 (n=30,82,43,128) | 0.0 (0.4) | 2.3 (0.9) | -0.3 (0.3) | 4.1 (0.6)
  Week 8 (n=30,70,43,104) | 0.3 (0.4) | 4.1 (0.9) | -0.1 (0.4) | 6.3 (0.9)
  Week 12 (n=28,53,42,84) | 0.1 (0.5) | 4.8 (1.0) | 0.3 (0.6) | 4.7 (0.7)
  Week 16 (n=28,45,38,70) | 0.3 (0.5) | 3.7 (0.7) | 0.5 (0.7) | 4.5 (0.7)

30. Secondary Outcome: Mean Change From Baseline in Total Percent of Psoriatic BSA During CP-690,550 Re-Treatment (Period C)
Description: Baseline was defined as the last observation until first dosing date in Period C.
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: percent change in psoriatic BSA
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 74 | 42 | 119
percent change in psoriatic BSA
  Week 4 (n=27,74,42,119) | -0.2 (0.3) | -1.0 (1.0) | 0.1 (0.9) | -4.9 (0.8)
  Week 8 (n=26,72,41,118) | 0.1 (0.5) | -2.3 (1.0) | 0.3 (0.9) | -5.5 (0.8)
  Week 16 (n=23,67,39,101) | 0.5 (0.6) | -4.0 (1.1) | 0.6 (1.2) | -6.8 (0.8)

31. Secondary Outcome: Mean Percent of Psoriatic BSA by Body Region During Initial CP-690,550 Treatment (Period A)
Description: as for outcome 25
Time Frame: Baseline and Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: percent psoriatic BSA
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
percent psoriatic BSA
  Head/Neck, Baseline (n=331,335) | 28.7 (1.25) | 25.9 (1.17)
  Head/Neck, Week 4 (n=326,331) | 20.5 (1.20) | 14.3 (1.04)
  Head/Neck, Week 8 (n=322,323) | 14.8 (1.06) | 9.7 (0.96)
  Head/Neck, Week 16 (n=311,306) | 12.6 (1.05) | 7.5 (0.88)
  Head/Neck, Week 24 (n=277,279) | 12.8 (1.17) | 6.3 (0.89)
  Upper limbs, Baseline (n=331,335) | 26.5 (1.04) | 26.2 (1.06)
  Upper limbs, Week 4 (n=326,331) | 21.8 (1.02) | 17.3 (0.91)
  Upper limbs, Week 8 (n=322,323) | 17.0 (0.95) | 11.7 (0.83)
  Upper Limbs, Week 16 (n=311,306) | 13.6 (0.92) | 8.0 (0.70)
  Upper limbs, Week 24 (n=277,279) | 12.2 (0.98) | 6.5 (0.65)
  Trunk, Baseline (n=331,335) | 26.0 (1.23) | 25.9 (1.18)
  Trunk, Week 4 (n=326,331) | 20.8 (1.16) | 17.2 (1.02)
  Trunk, Week 8 (n=322,323) | 16.5 (1.11) | 11.4 (0.94)
  Trunk, Week 16 (n=311,306) | 13.5 (1.05) | 8.5 (0.95)
  Trunk, Week 24 (n=277,279) | 12.5 (1.05) | 6.9 (0.85)
  Lower limbs, Baseline (n=331,335) | 28.7 (1.14) | 28.9 (1.12)
  Lower limbs, Week 4 (n=326,331) | 24.1 (1.13) | 20.2 (0.99)
  Lower limbs, Week 8 (n=322,323) | 18.5 (1.05) | 13.4 (0.93)
  Lower limbs, Week 16 (n=311,306) | 13.1 (0.95) | 7.9 (0.79)
  Lower limbs, Week 24 (n=277,279) | 11.3 (0.90) | 6.1 (0.71)

32. Secondary Outcome: Mean Percent of Psoriatic BSA by Body Region During Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 25
Time Frame: Baseline and Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: percent psoriatic BSA
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
percent psoriatic BSA
  Head/Neck, Baseline (n=31,82,45,133) | 4.2 (1.53) | 3.3 (0.79) | 0.9 (0.34) | 2.8 (0.70)
  Head/Neck, Week 4 (n=30,82,43,128) | 4.1 (1.44) | 11.3 (1.99) | 1.5 (0.44) | 12.2 (1.59)
  Head/Neck, Week 8 (n=30,70,43,104) | 4.8 (1.80) | 13.0 (2.34) | 1.5 (0.46) | 15.1 (1.97)
  Head/Neck, Week 12 (n=28,53,42,84) | 3.8 (1.00) | 13.5 (2.96) | 2.8 (0.72) | 11.5 (2.03)
  Head/Neck, Week 16 (n=28,45,38,70) | 3.8 (1.19) | 9.2 (2.11) | 2.3 (0.80) | 9.6 (1.76)
  Upper limbs, Baseline (n=31,82,45,133) | 2.1 (0.42) | 5.1 (1.00) | 3.1 (0.55) | 3.1 (0.50)
  Upper limbs, Week 4 (n=30,82,43,128) | 2.4 (0.48) | 7.5 (1.19) | 3.0 (0.55) | 7.6 (0.97)
  Upper limbs, Week 8 (n=30,70,43,104) | 2.8 (0.58) | 8.9 (1.41) | 3.6 (0.68) | 8.9 (1.25)
  Upper limbs, Week 12 (n=28,53,42,84) | 3.1 (0.59) | 8.8 (1.38) | 3.3 (0.62) | 6.6 (1.00)
  Upper limbs, Week 16 (n=28,45,38,70) | 3.2 (0.70) | 6.5 (1.13) | 3.5 (0.66) | 6.9 (1.28)
  Trunk, Baseline (n=31,82,45,133) | 1.6 (0.52) | 3.2 (0.88) | 1.5 (0.53) | 2.6 (0.59)
  Trunk, Week 4 (n=30,82,43,128) | 1.8 (0.53) | 5.1 (1.00) | 1.6 (0.53) | 6.0 (1.05)
  Trunk, Week 8 (n=30,70,43,104) | 1.9 (0.56) | 7.4 (1.73) | 1.5 (0.37) | 7.9 (1.29)
  Trunk, Week 12 (n=28,53,42,84) | 1.7 (0.61) | 4.4 (0.67) | 1.4 (0.39) | 5.3 (1.04)
  Trunk, Week 16 (n=28,45,38,70) | 2.1 (0.74) | 4.8 (0.90) | 1.8 (0.91) | 5.5 (1.05)
  Lower limbs, Baseline (n=31,82,45,133) | 1.3 (0.37) | 3.8 (1.02) | 2.1 (0.44) | 2.4 (0.49)
  Lower limbs, Week 4 (n=30,82,43,128) | 1.2 (0.33) | 4.9 (0.75) | 1.4 (0.38) | 5.7 (0.90)
  Lower limbs, Week 8 (n=30,70,43,104) | 1.5 (0.36) | 6.1 (1.07) | 1.7 (0.53) | 7.5 (1.30)
  Lower limbs, Week 12 (n=28,53,42,84) | 1.2 (0.35) | 7.0 (1.24) | 2.4 (0.80) | 5.4 (0.95)
  Lower limbs, Week 16 (n=28,45,38,70) | 1.4 (0.42) | 6.0 (1.30) | 3.0 (1.03) | 5.1 (0.78)

33. Secondary Outcome: Mean Percent of Psoriatic BSA by Body Region During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 25
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: percent psoriatic BSA
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
percent psoriatic BSA
  Head/Neck, Baseline (n=27,75,42,120) | 4.0 (1.23) | 18.6 (2.62) | 2.0 (0.61) | 18.3 (1.95)
  Head/Neck, Week 4 (n=27,74,42,119) | 3.6 (1.33) | 12.5 (2.09) | 2.9 (0.76) | 7.5 (1.12)
  Head/Neck, Week 8 (n=26,72,41,118) | 3.9 (1.25) | 9.5 (2.01) | 3.3 (1.08) | 6.3 (1.02)
  Head/Neck, Week 16 (n=23,67,39,101) | 4.6 (1.50) | 9.8 (1.97) | 1.4 (0.46) | 6.1 (1.31)
  Upper limbs, Baseline (n=27,75,42,120) | 3.2 (0.72) | 12.5 (1.73) | 3.6 (0.63) | 13.2 (1.40)
  Upper limbs, Week 4 (n=27,74,42,119) | 3.4 (0.82) | 11.1 (1.92) | 4.1 (0.90) | 8.4 (1.23)
  Upper limbs, Week 8 (n=26,72,41,118) | 4.1 (0.99) | 8.9 (1.83) | 3.7 (0.92) | 6.7 (0.97)
  Upper limbs, Week 16 (n=23,67,39,101) | 4.0 (1.02) | 7.0 (1.33) | 4.6 (1.24) | 5.3 (1.02)
  Trunk, Baseline (n=27,75,42,120) | 2.2 (0.77) | 10.9 (1.73) | 2.0 (0.85) | 11.1 (1.35)
  Trunk, Week 4 (n=27,74,42,119) | 2.0 (0.68) | 11.1 (2.33) | 3.2 (1.72) | 6.7 (1.10)
  Trunk, Week 8 (n=26,72,41,118) | 2.4 (0.73) | 10.2 (2.16) | 3.5 (1.76) | 5.9 (1.15)
  Trunk, Week 16 (n=23,67,39,101) | 3.0 (0.96) | 7.1 (1.54) | 4.7 (2.34) | 4.8 (1.16)
  Lower limbs, Baseline (n=27,75,42,120) | 1.4 (0.44) | 9.4 (1.21) | 3.7 (1.15) | 10.4 (1.27)
  Lower limbs, Week 4 (n=27,74,42,119) | 1.1 (0.27) | 9.5 (1.81) | 2.6 (0.95) | 6.9 (1.06)
  Lower limbs, Week 8 (n=26,72,41,118) | 1.4 (0.38) | 8.0 (1.73) | 3.0 (1.10) | 5.8 (0.92)
  Lower limbs, Week 16 (n=23,67,39,101) | 1.8 (0.45) | 6.5 (1.26) | 3.0 (1.33) | 3.5 (0.64)

34. Secondary Outcome: Mean Change From Baseline in Percent of Psoriatic BSA by Body Region During Initial CP-690,550 Treatment (Period A)
Description: Baseline defined as the last observation up to first dosing date in Period A.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: percent change in psoriatic BSA
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 326 | 331
percent change in psoriatic BSA
  Head/Neck, Week 4 (n=326,331) | -7.9 (0.71) | -11.7 (0.86)
  Head/Neck, Week 8 (n=322,323) | -13.8 (0.98) | -16.0 (1.04)
  Head/Neck, Week 16 (n=311,306) | -15.4 (1.13) | -17.9 (1.07)
  Head/Neck, Week 24 (n=277,279) | -14.9 (1.21) | -18.6 (1.12)
  Upper limbs, Week 4 (n=326,331) | -4.9 (0.58) | -8.8 (0.80)
  Upper limbs, Week 8 (n=322,323) | -9.7 (0.77) | -14.1 (0.92)
  Upper limbs, Week 16 (n=311,306) | -13.1 (0.89) | -17.4 (1.03)
  Upper limbs, Week 24 (n=277,279) | -14.2 (0.98) | -18.5 (1.01)
  Trunk, Week 4 (n=326,331) | -5.5 (0.67) | -8.6 (0.86)
  Trunk, Week 8 (n=322,323) | -9.9 (0.87) | -13.8 (1.03)
  Trunk, Week 16 (n=311,306) | -12.9 (0.98) | -16.9 (1.17)
  Trunk, Week 24 (n=277,279) | -13.4 (1.12) | -17.8 (1.12)
  Lower limbs, Week 4 (n=326,331) | -4.8 (0.57) | -8.6 (0.85)
  Lower limbs, Week 8 (n=322,323) | -10.4 (0.82) | -14.8 (0.99)
  Lower limbs, Week 16 (n=311,306) | -15.9 (1.04) | -20.3 (1.10)
  Lower limbs, Week 24 (n=277,279) | -17.1 (1.09) | -21.2 (1.07)

35. Secondary Outcome: Mean Change From Baseline in Percent of Psoriatic BSA by Body Region During Double-Blind Treatment Withdrawal (Period B)
Description: Baseline defined as the last observation up to first dosing date in Period B.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: percent psoriatic BSA
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 30 | 82 | 43 | 128
percent psoriatic BSA
  Head/Neck, Week 4 (n=30,82,43,128) | -0.3 (0.98) | 8.0 (1.49) | 0.7 (0.44) | 9.3 (1.53)
  Head/Neck, Week 8 (n=30,70,43,104) | 0.4 (1.41) | 10.0 (1.87) | 0.6 (0.50) | 12.8 (1.86)
  Head/Neck, Week 12 (n=28,53,42,84) | -0.9 (1.58) | 11.8 (2.71) | 1.8 (0.69) | 10.4 (1.95)
  Head/Neck, Week 16 (n=28,45,38,70) | -0.8 (1.42) | 7.9 (1.70) | 1.2 (0.75) | 8.3 (1.66)
  Upper limbs, Week 4 (n=30,82,43,128) | 0.4 (0.33) | 2.3 (1.14) | -0.2 (0.29) | 4.5 (0.76)
  Upper limbs, Week 8 (n=30,70,43,104) | 0.8 (0.47) | 4.1 (0.99) | 0.4 (0.54) | 6.2 (0.96)
  Upper limbs, Week 12 (n=28,53,42,84) | 1.0 (0.51) | 4.8 (1.14) | 0.4 (0.50) | 4.7 (0.86)
  Upper limbs, Week 16 (n=28,45,38,70) | 1.1 (0.55) | 2.7 (0.75) | 0.6 (0.46) | 4.9 (0.95)
  Trunk, Week 4 (n=30,82,43,128) | 0.1 (0.50) | 1.9 (1.17) | 0.0 (0.51) | 3.3 (0.74)
  Trunk, Week 8 (n=30,70,43,104) | 0.3 (0.54) | 4.0 (1.34) | -0.2 (0.56) | 5.6 (0.97)
  Trunk, Week 12 (n=28,53,42,84) | 0.0 (0.68) | 2.9 (0.75) | -0.2 (0.63) | 3.8 (0.75)
  Trunk, Week 16 (n=28,45,38,70) | 0.4 (0.73) | 3.3 (0.81) | 0.0 (1.09) | 3.9 (0.71)
  Lower limbs, Week 4 (n=30,82,43,128) | -0.2 (0.42) | 1.1 (0.92) | -0.7 (0.39) | 3.2 (0.68)
  Lower limbs, Week 8 (n=30,70,43,104) | 0.2 (0.43) | 2.7 (0.83) | -0.5 (0.66) | 5.3 (0.98)
  Lower limbs, Week 12 (n=28,53,42,84) | -0.1 (0.47) | 4.6 (1.19) | 0.3 (0.84) | 3.9 (0.84)
  Lower limbs, Week 16 (n=28,45,38,70) | 0.0 (0.51) | 3.3 (0.94) | 0.7 (0.86) | 3.7 (0.76)

36. Secondary Outcome: Mean Change From Baseline in Percent of Psoriatic BSA by Body Region During CP-690,550 Re-Treatment (Period C)
Description: Baseline defined as the last observation up to first dosing date in Period C.
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: percent psoriatic BSA
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 74 | 42 | 119
percent psoriatic BSA
  Head/Neck, Week 4 (n=27,74,42,119) | -0.3 (0.92) | -6.4 (1.40) | 0.9 (0.81) | -10.8 (1.53)
  Head/Neck, Week 8 (n=26,72,41,118) | 0.0 (1.07) | -8.6 (1.68) | 1.2 (0.91) | -10.9 (1.51)
  Head/Neck, Week 16 (n=23,67,39,101) | 0.4 (1.41) | -8.1 (2.04) | -0.7 (0.77) | -11.6 (1.84)
  Upper limbs, Week 4 (n=27,74,42,119) | 0.1 (0.26) | -1.6 (0.90) | 0.5 (0.69) | -4.9 (0.94)
  Upper limbs, Week 8 (n=26,72,41,118) | 0.8 (0.50) | -3.0 (0.85) | 0.1 (0.53) | -6.3 (1.11)
  Upper limbs, Week 16 (n=23,67,39,101) | 0.7 (0.97) | -5.0 (1.15) | 1.0 (0.99) | -7.6 (1.20)
  Trunk, Week 4 (n=27,74,42,119) | -0.2 (0.20) | 0.1 (1.12) | 1.3 (1.87) | -4.6 (0.88)
  Trunk, Week 8 (n=26,72,41,118) | 0.1 (0.43) | -1.1 (1.04) | 1.5 (1.92) | -4.8 (0.88)
  Trunk, Week 16 (n=23,67,39,101) | 0.7 (0.82) | -4.1 (1.44) | 2.7 (2.46) | -5.6 (1.02)
  Lower limbs, Week 4 (n=27,74,42,119) | -0.3 (0.36) | -0.1 (1.44) | -1.1 (0.93) | -3.6 (0.97)
  Lower limbs, Week 8 (n=26,72,41,118) | -0.1 (0.52) | -1.3 (1.50) | -0.7 (0.78) | -4.3 (0.85)
  Lower limbs, Week 16 (n=23,67,39,101) | 0.2 (0.60) | -2.3 (1.15) | -0.9 (1.14) | -6.1 (0.93)

37. Secondary Outcome: Mean PASI Score During Initial CP-690,550 Treatment (Period A)
Description: Combined assessment of lesion severity and area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated:0(0%)-6(90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4). PASI score can vary in increments of 0.1; higher scores represent greater severity of psoriasis.
Time Frame: Baseline and Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
score on a scale
  Baseline (n=331,335) | 21.1 (0.5) | 20.9 (0.4)
  Week 4 (n=326,331) | 13.5 (0.5) | 10.4 (0.4)
  Week 8 (n=322,323) | 10.1 (0.4) | 6.5 (0.4)
  Week 16 (n=311,307) | 8.1 (0.4) | 5.0 (0.4)
  Week 24 (n=277,279) | 7.6 (0.4) | 4.4 (0.4)

38. Secondary Outcome: Mean PASI Score During Double-Blind Treatment Withdrawal (Period B)
Description: Combined assessment of lesion severity and area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated:0(0%)-6(90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4). PASI score can vary in increments of 0.1; higher scores represent greater severity of psoriasis. Baseline defined as last observation up to first dosing date in Period B.
Time Frame: Baseline and Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
score on a scale
  Baseline (n=31,82,45,133) | 1.6 (0.2) | 1.8 (0.2) | 1.7 (0.2) | 1.5 (0.1)
  Week 4 (n=30,82,43,128) | 2.0 (0.3) | 5.0 (0.6) | 1.8 (0.3) | 5.3 (0.6)
  Week 8 (n=30,70,43,104) | 2.4 (0.4) | 6.5 (0.7) | 2.0 (0.4) | 6.8 (0.7)
  Week 12 (n=28,53,42,84) | 2.3 (0.4) | 6.4 (0.7) | 2.5 (0.4) | 5.6 (0.6)
  Week 16 (n=28,45,38,70) | 2.7 (0.5) | 5.5 (0.7) | 2.9 (0.5) | 5.5 (0.6)

39. Secondary Outcome: Mean PASI Score During the CP-690,550 Re-Treatment (Period C)
Description: Combined assessment of lesion severity and area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated:0(0%)-6(90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4). PASI score can vary in increments of 0.1; higher scores represent greater severity of psoriasis. Baseline defined as last observation up to first dosing date in Period C.
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
score on a scale
  Baseline (n=27,75,42,120) | 2.7 (0.5) | 9.9 (0.9) | 3.4 (0.6) | 9.8 (0.8)
  Week 4 (n=27,74,42,119) | 2.5 (0.4) | 7.8 (1.0) | 3.3 (0.6) | 5.0 (0.5)
  Week 8 (n=26,72,41,118) | 2.6 (0.5) | 6.0 (0.9) | 3.2 (0.6) | 4.1 (0.5)
  Week 16 (n=23,67,39,101) | 2.9 (0.5) | 5.2 (0.8) | 3.5 (0.7) | 3.5 (0.5)

40. Secondary Outcome: Mean Change From Baseline-A in PASI Score During Initial CP-690,550 Treatment (Period A)
Description: Combined assessment of lesion severity and area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated:0(0%)-6(90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4). PASI score can vary in increments of 0.1; higher scores represent greater severity of psoriasis. Baseline-A defined as last observation up to first dosing date in Period A.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 326 | 331
scores on a scale
  Week 4 (n=326,331) | -7.6 (0.4) | -10.5 (0.4)
  Week 8 (n=322,323) | -11.1 (0.4) | -14.2 (0.5)
  Week 16 (n=311,307) | -13.1 (0.5) | -15.8 (0.5)
  Week 24 (n=277,279) | -13.4 (0.5) | -16.0 (0.5)

41. Secondary Outcome: Mean Change From Baseline-B in PASI Score During Double-Blind Treatment Withdrawal (Period B)
Description: Combined assessment of lesion severity and area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated:0(0%)-6(90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4). PASI score can vary in increments of 0.1; higher scores represent greater severity of psoriasis. Baseline-B defined as last observation up to first dosing date in Period B.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 30 | 82 | 43 | 128
scores on a scale
  Week 4 (n=30,82,43,128) | 0.4 (0.2) | 3.3 (0.6) | 0.2 (0.2) | 3.8 (0.5)
  Week 8 (n=30,70,43,104) | 0.9 (0.4) | 4.9 (0.7) | 0.3 (0.3) | 5.4 (0.6)
  Week 12 (n=28,53,42,84) | 0.7 (0.4) | 4.8 (0.7) | 0.9 (0.4) | 4.5 (0.6)
  Week 16 (n=28,45,38,70) | 1.0 (0.5) | 4.1 (0.6) | 1.4 (0.4) | 4.4 (0.5)

42. Secondary Outcome: Mean Change From Baseline-C in PASI Score During the CP-690,550 Re-Treatment (Period C)
Description: Combined assessment of lesion severity and area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated:0(0%)-6(90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4). PASI score can vary in increments of 0.1; higher scores represent greater severity of psoriasis. Baseline-C defined as last observation up to first dosing date in Period C.
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 74 | 42 | 119
scores on a scale
  Week 4 (n=27,74,42,119) | -0.2 (0.4) | -2.3 (0.7) | -0.1 (0.5) | -4.8 (0.6)
  Week 8 (n=26,72,41,118) | 0.0 (0.5) | -3.8 (0.7) | -0.2 (0.4) | -5.4 (0.6)
  Week 16 (n=23,67,39,101) | 0.1 (0.6) | -4.5 (0.9) | -0.0 (0.7) | -5.9 (0.6)

43. Secondary Outcome: Mean PASI Component Scores During Initial CP-690,550 Treatment (Period A)
Description: as for outcome 38
Time Frame: Baseline and Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- CP-690,550 10 mg BID (Period A): Participants received CP-690,550 10 mg tablets orally BID for 24 weeks in Period A (Initial Treatment)
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
score on a scale
  Erythema Head/Neck, Baseline (n=331,335) | 2.2 (0.1) | 2.2 (0.1)
  Erythema Head/Neck, Week 4 (n=326,331) | 1.4 (0.1) | 1.1 (0.1)
  Erythema Head/Neck, Week 8 (n=322,323) | 1.1 (0.1) | 0.7 (0.0)
  Erythema Head/Neck, Week 16 (n=311,307) | 1.0 (0.1) | 0.7 (0.1)
  Erythema Head/Neck, Week 24 (n=277,279) | 1.0 (0.1) | 0.6 (0.1)
  Induration Head/Neck, Baseline (n=331,335) | 2.0 (0.1) | 1.9 (0.1)
  Induration Head/Neck, Week 4 (n=326,331) | 1.2 (0.1) | 0.9 (0.1)
  Induration Head/Neck, Week 8 (n=322,323) | 0.9 (0.1) | 0.6 (0.0)
  Induration Head/Neck, Week 16 (n=311,307) | 0.8 (0.1) | 0.5 (0.0)
  Induration Head/Neck, Week 24 (n=277,279) | 0.8 (0.1) | 0.5 (0.0)
  Scaling Head/Neck, Baseline (n=331,335) | 2.2 (0.1) | 2.1 (0.1)
  Scaling Head/Neck, Week 4 (n=326,331) | 1.3 (0.1) | 1.0 (0.1)
  Scaling Head/Neck, Week 8 (n=322,323) | 1.0 (0.1) | 0.6 (0.0)
  Scaling Head/Neck, Week 16 (n=311,307) | 0.9 (0.1) | 0.6 (0.1)
  Scaling Head/Neck, Week 24 (n=277,279) | 0.9 (0.1) | 0.6 (0.1)
  Erythema Upper limbs, Baseline (n=331,335) | 2.8 (0.0) | 2.8 (0.0)
  Erythema Upper limbs, Week 4 (n=326,331) | 1.9 (0.0) | 1.6 (0.0)
  Erythema Upper limbs, Week 8 (n=322,323) | 1.6 (0.1) | 1.2 (0.0)
  Erythema Upper limbs, Week 16 (n=311,307) | 1.4 (0.1) | 1.1 (0.1)
  Erythema Upper limbs, Week 24 (n=277,279) | 1.4 (0.1) | 1.0 (0.1)
  Induration Upper limbs, Baseline (n=331,335) | 2.6 (0.0) | 2.6 (0.0)
  Induration Upper limbs, Week 4 (n=326,331) | 1.9 (0.0) | 1.5 (0.1)
  Induration Upper limbs, Week 8 (n=322,323) | 1.5 (0.1) | 1.1 (0.1)
  Induration Upper limbs, Week 16 (n=311,307 | 1.4 (0.1) | 1.0 (0.1)
  Induration Upper limbs, Week 24 (n=277,279) | 1.4 (0.1) | 1.0 (0.1)
  Scaling Upper limbs, Baseline (n=331,335) | 2.7 (0.0) | 2.6 (0.0)
  Scaling Upper limbs, Week 4 (n=326,331) | 1.9 (0.0) | 1.5 (0.1)
  Scaling Upper limbs, Week 8 (n=322,323) | 1.5 (0.1) | 1.1 (0.1)
  Scaling Upper limbs, Week 16 (n=311,307) | 1.4 (0.1) | 1.0 (0.1)
  Scaling Upper limbs, Week 24 (n=277,279) | 1.4 (0.1) | 1.0 (0.1)
  Erythema Trunk, Baseline (n=331,335) | 2.9 (0.0) | 2.8 (0.0)
  Erythema Trunk, Week 4 (n=326,331) | 1.9 (0.1) | 1.6 (0.1)
  Erythema Trunk, Week 8 (n=322,323) | 1.6 (0.1) | 1.1 (0.1)
  Erythema Trunk, Week 16 (n=311,307) | 1.4 (0.1) | 0.9 (0.1)
  Erythema Trunk, Week 24 (n=277,279) | 1.4 (0.1) | 0.8 (0.1)
  Induration Trunk, Baseline (n=331,335) | 2.6 (0.0) | 2.6 (0.0)
  Induration Trunk, Week 4 (n=326,331) | 1.8 (0.1) | 1.4 (0.1)
  Induration Trunk, Week 8 (n=322,323) | 1.4 (0.1) | 0.9 (0.1)
  Induration Trunk, Week 16 (n=311,307) | 1.2 (0.1) | 0.8 (0.1)
  Induration Trunk, Week 24 (n=277,279) | 1.2 (0.1) | 0.7 (0.1)
  Scaling Trunk, Baseline (n=331,335) | 2.6 (0.0) | 2.5 (0.0)
  Scaling Trunk, Week 4 (n=326,331) | 1.7 (0.1) | 1.4 (0.1)
  Scaling Trunk, Week 8 (n=322,323) | 1.3 (0.1) | 0.9 (0.1)
  Scaling Trunk, Week 16 (n=311,307) | 1.2 (0.1) | 0.7 (0.1)
  Scaling Trunk, Week 24 (n=277,279) | 1.1 (0.1) | 0.7 (0.1)
  Erythema Lower limbs, Baseline (n=331,335) | 3.1 (0.0) | 3.1 (0.0)
  Erythema Lower limbs, Week 4 (n=326,331) | 2.2 (0.0) | 1.9 (0.1)
  Erythema Lower limbs, Week 8 (n=322,323) | 1.9 (0.1) | 1.4 (0.1)
  Erythema Lower limbs, Week 16 (n=311,307) | 1.5 (0.1) | 1.1 (0.1)
  Erythema Lower limbs, Week 24 (n=277,279) | 1.4 (0.1) | 1.0 (0.1)
  Induration Lower limbs, Baseline (n=331,335) | 2.9 (0.0) | 2.9 (0.0)
  Induration Lower limbs, Week 4 (n=326,331) | 2.1 (0.0) | 1.6 (0.1)
  Induration Lwer limbs, Week 8 (n=322,323) | 1.6 (0.1) | 1.2 (0.1)
  Induration Lower limbs, Week 16 (n=311,307) | 1.3 (0.1) | 0.9 (0.1)
  Induration Lower limbs, Week 24 (n=277,279) | 1.3 (0.1) | 0.9 (0.1)
  Scaling Lower limbs, Baseline (n=331,335) | 2.9 (0.0) | 2.9 (0.0)
  Scaling Lower limbs, Week 4 (n=326,331) | 2.0 (0.1) | 1.8 (0.1)
  Scaling Lower limbs, Week 8 (n=322,323) | 1.6 (0.1) | 1.2 (0.1)
  Scaling Lower limbs, Week 16 (n=311,307) | 1.3 (0.1) | 1.0 (0.1)
  Scaling Lower limbs, Week 24 (n=277,279) | 1.3 (0.1) | 1.0 (0.1)

44. Secondary Outcome: Mean PASI Component Scores During Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 38
Time Frame: Baseline and Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo for CP-690,550 5 mg BID (Period B): Participants received CP-690,550 5 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
- Placebo for 10 mg CP-690,550 (Period B): Participants received CP-690,550 10 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal)
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for CP-690,550 5 mg BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
score on a scale
  Erythema Head/Neck, Baseline (n=31,82,45,133) | 0.5 (0.1) | 0.4 (0.1) | 0.3 (0.1) | 0.3 (0.0)
  Erythema Head/Neck, Week 4 (n=30,82,43,128) | 0.6 (0.1) | 1.1 (0.1) | 0.4 (0.1) | 1.1 (0.1)
  Erythema Head/Neck, Week 8 (n=30,70,43,104) | 0.7 (0.2) | 1.2 (0.1) | 0.3 (0.1) | 1.3 (0.1)
  Erythema Head/Neck, Week 12 (n=28,53,42,84) | 0.7 (0.2) | 1.1 (0.2) | 0.5 (0.1) | 1.1 (0.1)
  Erythema Head/Neck, Week 16 (n=28,45,38,70) | 0.7 (0.2) | 0.8 (0.1) | 0.5 (0.1) | 1.0 (0.1)
  Induration Head/Neck, Baseline (n=31,82,45,133) | 0.3 (0.1) | 0.4 (0.1) | 0.1 (0.1) | 0.2 (0.0)
  Induration Head/Neck, Week 4 (n=30,82,43,128) | 0.4 (0.1) | 0.9 (0.1) | 0.3 (0.1) | 0.9 (0.1)
  Induration Head/Neck, Week 8 (n=30,70,43,104) | 0.4 (0.1) | 1.0 (0.1) | 0.3 (0.1) | 1.1 (0.1)
  Induration Head/Neck, Week 12 (n=28,53,42,84) | 0.4 (0.1) | 0.9 (0.1) | 0.4 (0.1) | 0.9 (0.1)
  Induration Head/Neck, Week 16 (n=28,45,38,70) | 0.5 (0.1) | 0.7 (0.1) | 0.3 (0.1) | 0.8 (0.1)
  Scaling Head/Neck, Baseline (n=31,82,45,133) | 0.4 (0.1) | 0.4 (0.1) | 0.2 (0.1) | 0.3 (0.1)
  Scaling Head/Neck, Week 4 (n=30,82,43,128) | 0.4 (0.1) | 1.0 (0.1) | 0.3 (0.1) | 1.1 (0.1)
  Scaling Head/Neck, Week 8 (n=30,70,43,104) | 0.5 (0.1) | 1.1 (0.1) | 0.4 (0.1) | 1.3 (0.1)
  Scaling Head/Neck, Week 12 (n=28,53,42,84) | 0.6 (0.1) | 1.1 (0.1) | 0.5 (0.1) | 1.1 (0.1)
  Scaling Head/Neck, Week 16 (n=28,45,38,70) | 0.6 (0.2) | 0.8 (0.1) | 0.5 (0.1) | 0.9 (0.1)
  Erythema Upper limbs, Baseline (n=31,82,45,133) | 0.6 (0.1) | 0.6 (0.1) | 0.8 (0.1) | 0.5 (0.1)
  Erythema Upper limbs, Week 4 (n=30,82,43,128) | 0.8 (0.1) | 1.3 (0.1) | 0.8 (0.1) | 1.3 (0.1)
  Erythema Upper limbs, Week 8 (n=30,70,43,104) | 0.9 (0.2) | 1.5 (0.1) | 0.9 (0.1) | 1.4 (0.1)
  Erythema Upper limbs, Week 12 (n=28,53,42,84) | 1.0 (0.2) | 1.5 (0.1) | 0.9 (0.1) | 1.3 (0.1)
  Erythema Upper limbs, Week 16 (n=28,45,38,70) | 1.0 (0.2) | 1.4 (0.1) | 1.1 (0.1) | 1.3 (0.1)
  Induration Upper limbs, Baseline (n=31,82,45,133) | 0.7 (0.1) | 0.6 (0.1) | 0.6 (0.1) | 0.5 (0.1)
  Induration Upper limbs, Week 4 (n=30,82,43,128) | 0.8 (0.1) | 1.3 (0.1) | 0.7 (0.1) | 1.1 (0.1)
  Induration Upper limbs, Week 8 (n=30,70,43,104) | 0.8 (0.2) | 1.5 (0.1) | 0.8 (0.1) | 1.4 (0.1)
  Induration Upper limbs, Week 12 (n=28,53,42,84) | 1.0 (0.2) | 1.5 (0.1) | 1.0 (0.1) | 1.3 (0.1)
  Induration Upper limbs, Week 16 (n=28,45,38,70) | 1.1 (0.2) | 1.3 (0.2) | 1.1 (0.1) | 1.4 (0.1)
  Scaling Upper limbs, Baseline (n=31,82,45,133) | 0.8 (0.2) | 0.6 (0.1) | 0.7 (0.1) | 0.5 (0.1)
  Scaling Upper limbs, Week 4 (n=30,82,43,128) | 0.8 (0.2) | 1.3 (0.1) | 0.7 (0.1) | 1.2 (0.1)
  Scaling Upper limbs, Week 8 (n=30,70,43,104) | 0.9 (0.2) | 1.4 (0.1) | 0.8 (0.1) | 1.4 (0.1)
  Scaling Upper limbs, Week 12 (n=28,53,42,84) | 1.0 (0.2) | 1.4 (0.1) | 1.0 (0.1) | 1.4 (0.1)
  Scaling Upper limbs, Week 16 (n=28,45,38,70) | 1.1 (0.2) | 1.3 (0.2) | 1.3 (0.2) | 1.4 (0.1)
  Erythema Trunk, Baseline (n=31,82,45,133) | 0.5 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1)
  Erythema Trunk, Week 4 (n=30,82,43,128) | 0.7 (0.2) | 1.1 (0.1) | 0.4 (0.1) | 1.1 (0.1)
  Erythema Trunk, Week 8 (n=30,70,43,104) | 0.9 (0.2) | 1.5 (0.1) | 0.5 (0.1) | 1.4 (0.1)
  Erythema Trunk, Week 12 (n=28,53,42,84) | 0.7 (0.2) | 1.5 (0.2) | 0.5 (0.1) | 1.1 (0.1)
  Erythema Trunk, Week 16 (n=28,45,38,70) | 0.9 (0.2) | 1.3 (0.2) | 0.5 (0.1) | 1.1 (0.1)
  Induration Trunk, Baseline (n=31,82,45,133) | 0.4 (0.1) | 0.3 (0.1) | 0.3 (0.1) | 0.3 (0.0)
  Induration Trunk, Week 4 (n=30,82,43,128) | 0.4 (0.1) | 0.9 (0.1) | 0.3 (0.1) | 0.8 (0.1)
  Induration Trunk, Week 8 (n=30,70,43,104) | 0.5 (0.1) | 1.2 (0.1) | 0.4 (0.1) | 1.1 (0.1)
  Induration Trunk, Week 12 (n=28,53,42,84) | 0.5 (0.2) | 1.2 (0.1) | 0.5 (0.1) | 0.9 (0.1)
  Induration Trunk, Week 16 (n=28,45,38,70) | 0.6 (0.2) | 1.2 (0.2) | 0.6 (0.1) | 1.1 (0.1)
  Scaling Trunk, Baseline (n=31,82,45,133) | 0.3 (0.1) | 0.3 (0.1) | 0.3 (0.1) | 0.3 (0.0)
  Scaling Trunk, Week 4 (n=30,82,43,128) | 0.4 (0.1) | 0.9 (0.1) | 0.3 (0.1) | 0.8 (0.1)
  Scaling Trunk, Week 8 (n=30,70,43,104) | 0.5 (0.1) | 1.2 (0.1) | 0.4 (0.1) | 1.1 (0.1)
  Scaling Trunk, Week 12 (n=28,53,42,84) | 0.4 (0.1) | 1.2 (0.1) | 0.5 (0.1) | 0.9 (0.1)
  Scaling Trunk, Week 16 (n=28,45,38,70) | 0.6 (0.2) | 1.1 (0.2) | 0.6 (0.1) | 1.0 (0.1)
  Erythema Lower limbs, Baseline (n=31,82,45,133) | 0.5 (0.1) | 0.6 (0.1) | 0.8 (0.1) | 0.5 (0.1)
  Erythema Lower limbs, Week 4 (n=30,82,43,128) | 0.6 (0.1) | 1.3 (0.1) | 0.8 (0.1) | 1.3 (0.1)
  Erythema Lower limbs, Week 8 (n=30,70,43,104) | 0.8 (0.2) | 1.6 (0.1) | 0.8 (0.2) | 1.5 (0.1)
  Erythema Lower limbs, Week 12 (n=28,53,42,84) | 0.8 (0.2) | 1.6 (0.2) | 0.9 (0.2) | 1.4 (0.1)
  Erythema Lower limbs, Week 16 (n=28,45,38,70) | 0.8 (0.2) | 1.6 (0.2) | 1.0 (0.2) | 1.3 (0.1)
  Induration Lower limbs, Baseline (n=31,82,45,133) | 0.5 (0.1) | 0.5 (0.1) | 0.6 (0.1) | 0.3 (0.0)
  Induration Lower limbs, Week 4 (n=30,82,43,128) | 0.6 (0.1) | 1.0 (0.1) | 0.6 (0.1) | 1.0 (0.1)
  Induration Lower limbs, Week 8 (n=30,70,43,104) | 0.6 (0.2) | 1.4 (0.1) | 0.6 (0.1) | 1.3 (0.1)
  Induration Lower limbs, Week 12 (n=28,53,42,84) | 0.6 (0.2) | 1.4 (0.1) | 0.8 (0.1) | 1.2 (0.1)
  Induration Lower limbs, Week 16 (n=28,45,38,70) | 0.6 (0.1) | 1.4 (0.2) | 0.9 (0.2) | 1.2 (0.1)
  Scaling Lower limbs, Baseline (n=31,82,45,133) | 0.5 (0.1) | 0.4 (0.1) | 0.6 (0.1) | 0.4 (0.0)
  Scaling Lower limbs, Week 4 (n=30,82,43,128) | 0.5 (0.1) | 1.0 (0.1) | 0.6 (0.1) | 1.0 (0.1)
  Scaling Lower limbs, Week 8 (n=30,70,43,104) | 0.7 (0.2) | 1.3 (0.1) | 0.6 (0.1) | 1.3 (0.1)
  Scaling Lower limbs, Week 12 (n=28,53,42,84) | 0.6 (0.2) | 1.4 (0.1) | 0.7 (0.1) | 1.3 (0.1)
  Scaling Lower limbs, Week 16 (n=28,45,38,70) | 0.6 (0.2) | 1.4 (0.2) | 0.9 (0.2) | 1.3 (0.1)

45. Secondary Outcome: Mean PASI Component Scores During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 39
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
score on a scale
  Erythema Head/Neck, Baseline (n=27,75,42,120) | 0.7 (0.2) | 1.5 (0.1) | 0.5 (0.1) | 1.6 (0.1)
  Erythema Head/Neck, Week 4 (n=27,74,42,119) | 0.6 (0.1) | 1.1 (0.1) | 0.6 (0.1) | 0.7 (0.1)
  Erythema Head/Neck, Week 8 (n=26,72,41,118) | 0.8 (0.2) | 0.8 (0.1) | 0.5 (0.1) | 0.7 (0.1)
  Erythema Head/Neck, Week 16 (n=23,67,39,101) | 0.7 (0.2) | 1.0 (0.1) | 0.4 (0.1) | 0.6 (0.1)
  Induration Head/Neck, Baseline (n=27,75,42,120) | 0.5 (0.1) | 1.3 (0.1) | 0.4 (0.1) | 1.4 (0.1)
  Induration Head/Neck, Week 4 (n=27,74,42,119) | 0.3 (0.1) | 0.9 (0.1) | 0.4 (0.1) | 0.6 (0.1)
  Induration Head/Neck, Week 8 (n=26,72,41,118) | 0.4 (0.2) | 0.8 (0.1) | 0.3 (0.1) | 0.5 (0.1)
  Induration Head/Neck, Week 16 (n=23,67,39,101) | 0.4 (0.1) | 0.7 (0.1) | 0.2 (0.1) | 0.5 (0.1)
  Scaling Head/Neck, Baseline (n=27,75,42,120) | 0.6 (0.2) | 1.4 (0.1) | 0.5 (0.1) | 1.6 (0.1)
  Scaling Head/Neck, Week 4 (n=27,74,42,119) | 0.5 (0.2) | 1.0 (0.1) | 0.6 (0.1) | 0.7 (0.1)
  Scaling Head/Neck, Week 8 (n=26,72,41,118) | 0.7 (0.2) | 0.9 (0.1) | 0.5 (0.1) | 0.6 (0.1)
  Scaling Head/Neck, Week 16 (n=23,67,39,101) | 0.5 (0.2) | 0.9 (0.1) | 0.4 (0.1) | 0.5 (0.1)
  Erythema Upper limbs, Baseline (n=27,75,42,120) | 1.0 (0.2) | 1.9 (0.1) | 1.2 (0.2) | 1.8 (0.1)
  Erythema Upper limbs, Week 4 (n=27,74,42,119) | 0.9 (0.2) | 1.5 (0.1) | 1.1 (0.2) | 1.1 (0.1)
  Erythema Upper limbs, Week 8 (n=26,72,41,118) | 0.8 (0.2) | 1.2 (0.1) | 1.0 (0.1) | 1.0 (0.1)
  Erythema Upper limbs, Week 16 (n=23,67,39,101) | 1.0 (0.2) | 1.3 (0.1) | 1.1 (0.2) | 0.9 (0.1)
  Induration Upper limbs, Baseline (n=27,75,42,120) | 1.1 (0.2) | 1.9 (0.1) | 1.1 (0.1) | 1.7 (0.1)
  Induration Upper limbs, Week 4 (n=27,74,42,119) | 1.0 (0.2) | 1.4 (0.1) | 1.1 (0.1) | 1.1 (0.1)
  Induration Upper limbs, Week 8 (n=26,72,41,118) | 1.0 (0.2) | 1.2 (0.1) | 1.0 (0.1) | 1.0 (0.1)
  Induration Upper limbs, Week 16 (n=23,67,39,101) | 1.1 (0.2) | 1.2 (0.1) | 1.1 (0.2) | 0.9 (0.1)
  Scaling Upper limbs, Baseline (n=27,75,42,120) | 1.1 (0.2) | 1.8 (0.1) | 1.3 (0.2) | 1.8 (0.1)
  Scaling Upper limbs, Week 4 (n=27,74,42,119) | 1.1 (0.2) | 1.5 (0.1) | 1.1 (0.1) | 1.1 (0.1)
  Scaling Upper limbs, Week 8 (n=26,72,41,118) | 0.9 (0.2) | 1.2 (0.1) | 1.1 (0.1) | 1.0 (0.1)
  Scaling Upper limbs, Week 16 (n=23,67,39,101) | 1.2 (0.2) | 1.3 (0.1) | 1.1 (0.2) | 0.9 (0.1)
  Erythema Trunk, Baseline (n=27,75,42,120) | 0.9 (0.2) | 1.9 (0.1) | 0.7 (0.2) | 1.8 (0.1)
  Erythema Trunk, Week 4 (n=27,74,42,119) | 0.8 (0.2) | 1.4 (0.1) | 0.6 (0.1) | 1.0 (0.1)
  Erythema Trunk, Week 8 (n=26,72,41,118) | 0.8 (0.2) | 1.2 (0.1) | 0.7 (0.1) | 0.8 (0.1)
  Erythema Trunk, Week 16 (n=23,67,39,101) | 0.7 (0.2) | 1.1 (0.1) | 0.6 (0.2) | 0.8 (0.1)
  Induration Trunk, Baseline (n=27,75,42,120) | 0.7 (0.2) | 1.7 (0.1) | 0.7 (0.2) | 1.5 (0.1)
  Induration Trunk, Week 4 (n=27,74,42,119) | 0.6 (0.2) | 1.2 (0.1) | 0.6 (0.1) | 0.8 (0.1)
  Induration Trunk, Week 8 (n=26,72,41,118) | 0.5 (0.2) | 1.0 (0.1) | 0.6 (0.1) | 0.7 (0.1)
  Induration Trunk, Week 16 (n=23,67,39,101) | 0.5 (0.2) | 0.9 (0.1) | 0.6 (0.1) | 0.7 (0.1)
  Scaling Trunk, Baseline (n=27,75,42,120) | 0.7 (0.2) | 1.6 (0.1) | 0.7 (0.2) | 1.5 (0.1)
  Scaling Trunk, Week 4 (n=27,74,42,119) | 0.5 (0.1) | 1.3 (0.1) | 0.6 (0.1) | 0.9 (0.1)
  Scaling Trunk, Week 8 (n=26,72,41,118) | 0.5 (0.1) | 1.0 (0.1) | 0.6 (0.1) | 0.7 (0.1)
  Scaling Trunk, Week 16 (n=23,67,39,101) | 0.4 (0.1) | 0.9 (0.1) | 0.6 (0.1) | 0.7 (0.1)
  Erythema Lower limbs, Baseline (n=27,75,42,120) | 0.7 (0.2) | 2.1 (0.1) | 1.1 (0.2) | 1.9 (0.1)
  Erythema Lower limbs, Week 4 (n=27,74,42,119) | 0.7 (0.2) | 1.6 (0.1) | 1.0 (0.2) | 1.3 (0.1)
  Erythema Lower limbs, Week 8 (n=26,72,41,118) | 0.8 (0.2) | 1.3 (0.1) | 0.9 (0.2) | 1.0 (0.1)
  Erythema Lower limbs, Week 16 (n=23,67,39,101) | 1.0 (0.2) | 1.3 (0.1) | 0.9 (0.2) | 0.9 (0.1)
  Induration Lower limbs, Baseline (n=27,75,42,120) | 0.6 (0.1) | 1.9 (0.1) | 1.0 (0.2) | 1.7 (0.1)
  Induration Lower limbs, Week 4 (n=27,74,42,119) | 0.7 (0.2) | 1.5 (0.1) | 0.9 (0.2) | 1.0 (0.1)
  Induration Lower limbs, Week 8 (n=26,72,41,118) | 0.7 (0.2) | 1.3 (0.1) | 0.9 (0.2) | 0.9 (0.1)
  Induration Lower limbs, Week 16 (n=23,67,39,101) | 0.9 (0.2) | 1.1 (0.1) | 0.9 (0.2) | 0.8 (0.1)
  Scaling Lower limbs, Baseline (n=27,75,42,120) | 0.6 (0.2) | 1.8 (0.1) | 1.0 (0.2) | 1.8 (0.1)
  Scaling Lower limbs, Week 4 (n=27,74,42,119) | 0.7 (0.2) | 1.5 (0.1) | 0.9 (0.2) | 1.1 (0.1)
  Scaling Lower limbs, Week 8 (n=26,72,41,118) | 0.7 (0.2) | 1.2 (0.1) | 0.8 (0.2) | 1.0 (0.1)
  Scaling Lower limbs, Week 16 (n=23,67,39,101) | 1.0 (0.2) | 1.1 (0.1) | 0.8 (0.2) | 0.8 (0.1)

46. Secondary Outcome: Mean Change From Baseline in PASI Component Scores During Initial CP-690,550 Treatment (Period A)
Description: as for outcome 38
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 326 | 331
score on a scale
  Erythema Head/Neck, Week 4 (n=326,331) | -0.8 (0.1) | -1.2 (0.1)
  Erythema Head/Neck, Week 8 (n=322,323) | -1.1 (0.1) | -1.5 (0.1)
  Erythema Head/Neck, Week 16 (n=311,307) | -1.2 (0.1) | -1.6 (0.1)
  Erythema Head/Neck, Week 24 (n=277,279) | -1.2 (0.1) | -1.6 (0.1)
  Induration Head/Neck, Week 4 (n=326,331) | -0.8 (0.0) | -1.1 (0.1)
  Induration Head/Neck, Week 8 (n=322,323) | -1.1 (0.1) | -1.4 (0.1)
  Induration Head/Neck, Week 16 (n=311,307) | -1.2 (0.1) | -1.4 (0.1)
  Induration Head/Neck, Week 24 (n=277,279) | -1.1 (0.1) | -1.4 (0.1)
  Scaling Head/Neck, Week 4 (n=326,331) | -0.9 (0.1) | -1.1 (0.1)
  Scaling Head/Neck, Week 8 (n=322,323) | -1.2 (0.1) | -1.5 (0.1)
  Scaling Head/Neck, Week 16 (n=311,307) | -1.3 (0.1) | -1.5 (0.1)
  Scaling Head/Neck, Week 24 (n=277,279) | -1.2 (0.1) | -1.5 (0.1)
  Erythema Upper limbs, Week 4 (n=326,331) | -0.9 (0.0) | -1.2 (0.0)
  Erythema Upper limbs, Week 8 (n=322,323) | -1.3 (0.1) | -1.5 (0.1)
  Erythema Upper limbs, Week 16 (n=311,307) | -1.4 (0.1) | -1.7 (0.1)
  Erythema Upper limbs, Week 24 (n=277,279) | -1.5 (0.1) | -1.8 (0.1)
  Induration Upper limbs, Week 4 (n=326,331) | -0.8 (0.0) | -1.2 (0.1)
  Induration Upper limbs, Week 8 (n=322,323) | -1.1 (0.1) | -1.5 (0.1)
  Induration Upper limbs, Week 16 (n=311,307 | -1.2 (0.1) | -1.6 (0.1)
  Induration Upper limbs, Week 24 (n=277,279) | -1.2 (0.1) | -1.6 (0.1)
  Scaling Upper limbs, Week 4 (n=326,331) | -0.7 (0.0) | -1.1 (0.1)
  Scaling Upper limbs, Week 8 (n=322,323) | -1.1 (0.1) | -1.5 (0.1)
  Scaling Upper limbs, Week 16 (n=311,307) | -1.2 (0.1) | -1.6 (0.1)
  Scaling Upper limbs, Week 24 (n=277,279) | -1.3 (0.1) | -1.6 (0.1)
  Erythema Trunk, Week 4 (n=326,331) | -0.9 (0.0) | -1.3 (0.1)
  Erythema Trunk, Week 8 (n=322,323) | -1.3 (0.1) | -1.7 (0.1)
  Erythema Trunk, Week 16 (n=311,307) | -1.5 (0.1) | -1.9 (0.1)
  Erythema Trunk, Week 24 (n=277,279) | -1.5 (0.1) | -2.0 (0.1)
  Induration Trunk, Week 4 (n=326,331) | -0.8 (0.0) | -1.2 (0.1)
  Induration Trunk, Week 8 (n=322,323) | -1.2 (0.1) | -1.7 (0.1)
  Induration Trunk, Week 16 (n=311,307) | -1.4 (0.1) | -1.8 (0.1)
  Induration Trunk, Week 24 (n=277,279) | -1.4 (0.1) | -1.9 (0.1)
  Scaling Trunk, Week 4 (n=326,331) | -0.8 (0.1) | -1.1 (0.1)
  Scaling Trunk, Week 8 (n=322,323) | -1.2 (0.1) | -1.6 (0.1)
  Scaling Trunk, Week 16 (n=311,307) | -1.4 (0.1) | -1.8 (0.1)
  Scaling Trunk, Week 24 (n=277,279) | -1.4 (0.1) | -1.8 (0.1)
  Erythema Lower limbs, Week 4 (n=326,331) | -0.9 (0.0) | -1.2 (0.0)
  Erythema Lower limbs, Week 8 (n=322,323) | -1.3 (0.1) | -1.7 (0.1)
  Erythema Lower limbs, Week 16 (n=311,307) | -1.6 (0.1) | -2.0 (0.1)
  Erythema Lower limbs, Week 24 (n=277,279) | -1.7 (0.1) | -2.1 (0.1)
  Induration Lower limbs, Week 4 (n=326,331) | -0.8 (0.0) | -1.3 (0.1)
  Induration Lower limbs, Week 8 (n=322,323) | -1.2 (0.1) | -1.7 (0.1)
  Induration Lower limbs, Week 16 (n=311,307) | -1.5 (0.1) | -2.0 (0.1)
  Induration Lower limbs, Week 24 (n=277,279) | -1.6 (0.1) | -2.0 (0.1)
  Scaling Lower limbs, Week 4 (n=326,331) | -0.9 (0.0) | -1.2 (0.1)
  Scaling Lower limbs, Week 8 (n=322,323) | -1.3 (0.1) | -1.8 (0.1)
  Scaling Lower limbs, Week 16 (n=311,307) | -1.6 (0.1) | -2.0 (0.1)
  Scaling Lower limbs, Week 24 (n=277,279) | -1.6 (0.1) | -2.0 (0.1)

47. Secondary Outcome: Mean Change From Baseline in PASI Component Scores During Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 38
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for CP-690,550 5 mg BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 (Period B)
Number analyzed (Participants) | 30 | 82 | 45 | 128
score on a scale
  Erythema Head/Neck, Week 4 (n=30,82,43,128) | 0.1 (0.1) | 0.8 (0.1) | 0.2 (0.1) | 0.8 (0.1)
  Erythema Head/Neck, Week 8 (n=30,70,43,104) | 0.2 (0.2) | 0.9 (0.1) | 0.1 (0.1) | 1.1 (0.1)
  Erythema Head/Neck, Week 12 (n=28,53,42,84) | 0.2 (0.1) | 0.8 (0.1) | 0.2 (0.1) | 0.9 (0.1)
  Erythema Head/Neck, Week 16 (n=28,45,38,70) | 0.1 (0.1) | 0.6 (0.1) | 0.2 (0.1) | 0.8 (0.1)
  Induration Head/Neck, Week 4 (n=30,82,43,128) | 0.1 (0.1) | 0.5 (0.1) | 0.1 (0.1) | 0.7 (0.1)
  Induration Head/Neck, Week 8 (n=30,70,43,104) | 0.1 (0.1) | 0.7 (0.1) | 0.2 (0.1) | 0.9 (0.1)
  Induration Head/Neck, Week 12 (n=28,53,42,84) | 0.1 (0.1) | 0.6 (0.1) | 0.3 (0.1) | 0.8 (0.1)
  Induration Head/Neck, Week 16 (n=28,45,38,70) | 0.1 (0.1) | 0.5 (0.1) | 0.2 (0.1) | 0.7 (0.1)
  Scaling Head/Neck, Week 4 (n=30,82,43,128) | 0.0 (0.1) | 0.6 (0.1) | 0.2 (0.1) | 0.8 (0.1)
  Scaling Head/Neck, Week 8 (n=30,70,43,104) | 0.1 (0.1) | 0.8 (0.1) | 0.2 (0.1) | 1.0 (0.1)
  Scaling Head/Neck, Week 12 (n=28,53,42,84) | 0.1 (0.1) | 0.7 (0.1) | 0.3 (0.1) | 1.0 (0.1)
  Scaling Head/Neck, Week 16 (n=28,45,38,70) | 0.1 (0.1) | 0.7 (0.1) | 0.3 (0.1) | 0.8 (0.1)
  Erythema Upper limbs, Week 4 (n=30,82,43,128) | 0.1 (0.1) | 0.7 (0.1) | 0.1 (0.1) | 0.7 (0.1)
  Erythema Upper limbs, Week 8 (n=30,70,43,104) | 0.3 (0.1) | 0.9 (0.1) | 0.2 (0.1) | 0.9 (0.1)
  Erythema Upper limbs, Week 12 (n=28,53,42,84) | 0.4 (0.2) | 0.9 (0.1) | 0.2 (0.1) | 0.9 (0.1)
  Erythema Upper limbs, Week 16 (n=28,45,38,70) | 0.4 (0.1) | 0.8 (0.1) | 0.4 (0.1) | 0.9 (0.1)
  Induration Upper limbs, Week 4 (n=30,82,43,128) | 0.1 (0.1) | 0.6 (0.1) | 0.1 (0.1) | 0.6 (0.1)
  Induration Upper limbs, Week 8 (n=30,70,43,104) | 0.2 (0.1) | 0.9 (0.1) | 0.2 (0.1) | 0.9 (0.1)
  Induration Upper limbs, Week 12 (n=28,53,42,84) | 0.4 (0.2) | 0.9 (0.1) | 0.4 (0.1) | 0.9 (0.1)
  Induration Upper limbs, Week 16 (n=28,45,38,70) | 0.4 (0.2) | 0.9 (0.1) | 0.5 (0.1) | 0.9 (0.1)
  Scaling Upper limbs, Week 4 (n=30,82,43,128) | 0.1 (0.1) | 0.7 (0.1) | 0.1 (0.1) | 0.7 (0.1)
  Scaling Upper limbs, Week 8 (n=30,70,43,104) | 0.1 (0.1) | 0.9 (0.1) | 0.1 (0.1) | 0.9 (0.1)
  Scaling Upper limbs, Week 12 (n=28,53,42,84) | 0.3 (0.1) | 0.9 (0.1) | 0.3 (0.1) | 1.0 (0.1)
  Scaling Upper limbs, Week 16 (n=28,45,38,70) | 0.3 (0.2) | 0.9 (0.1) | 0.6 (0.1) | 1.1 (0.1)
  Erythema Trunk, Week 4 (n=30,82,43,128) | 0.2 (0.1) | 0.7 (0.1) | 0.0 (0.1) | 0.7 (0.1)
  Erythema Trunk, Week 8 (n=30,70,43,104) | 0.4 (0.1) | 1.0 (0.1) | 0.1 (0.1) | 1.0 (0.1)
  Erythema Trunk, Week 12 (n=28,53,42,84) | 0.1 (0.1) | 1.2 (0.2) | 0.2 (0.1) | 0.8 (0.1)
  Erythema Trunk, Week 16 (n=28,45,38,70) | 0.3 (0.2) | 1.0 (0.2) | 0.2 (0.1) | 0.8 (0.1)
  Induration Trunk, Week 4 (n=30,82,43,128) | -0.0 (0.1) | 0.6 (0.1) | 0.0 (0.1) | 0.5 (0.1)
  Induration Trunk, Week 8 (n=30,70,43,104) | 0.1 (0.1) | 0.9 (0.1) | 0.2 (0.1) | 0.8 (0.1)
  Induration Trunk, Week 12 (n=28,53,42,84) | 0.1 (0.1) | 1.0 (0.1) | 0.3 (0.1) | 0.7 (0.1)
  Induration Trunk, Week 16 (n=28,45,38,70) | 0.2 (0.1) | 1.0 (0.2) | 0.3 (0.1) | 0.8 (0.1)
  Scaling Trunk, Week 4 (n=30,82,43,128) | 0.1 (0.1) | 0.6 (0.1) | -0.0 (0.1) | 0.5 (0.1)
  Scaling Trunk, Week 8 (n=30,70,43,104) | 0.2 (0.1) | 0.9 (0.1) | 0.2 (0.1) | 0.9 (0.1)
  Scaling Trunk, Week 12 (n=28,53,42,84) | 0.1 (0.1) | 0.9 (0.1) | 0.2 (0.1) | 0.6 (0.1)
  Scaling Trunk, Week 16 (n=28,45,38,70) | 0.4 (0.2) | 0.9 (0.2) | 0.3 (0.2) | 0.8 (0.1)
  Erythema Lower limbs, Week 4 (n=30,82,43,128) | 0.1 (0.1) | 0.7 (0.1) | 0.0 (0.1) | 0.8 (0.1)
  Erythema Lower limbs, Week 8 (n=30,70,43,104) | 0.3 (0.2) | 1.0 (0.1) | -0.0 (0.1) | 1.1 (0.1)
  Erythema Lower limbs, Week 12 (n=28,53,42,84) | 0.3 (0.2) | 1.0 (0.1) | 0.1 (0.2) | 1.0 (0.1)
  Erythema Lower limbs, Week 16 (n=28,45,38,70) | 0.3 (0.2) | 1.1 (0.2) | 0.3 (0.2) | 0.9 (0.1)
  Induration Lower limbs, Week 4 (n=30,82,43,128) | 0.1 (0.1) | 0.5 (0.1) | 0.0 (0.1) | 0.7 (0.1)
  Induration Lower limbs, Week 8 (n=30,70,43,104) | 0.1 (0.2) | 0.9 (0.1) | 0.0 (0.1) | 1.0 (0.1)
  Induration Lower limbs, Week 12 (n=28,53,42,84) | 0.1 (0.2) | 0.9 (0.1) | 0.2 (0.1) | 0.9 (0.1)
  Induration Lower limbs, Week 16 (n=28,45,38,70) | 0.1 (0.1) | 0.9 (0.1) | 0.4 (0.2) | 0.9 (0.1)
  Scaling Lower limbs, Week 4 (n=30,82,43,128) | 0.1 (0.1) | 0.6 (0.1) | -0.0 (0.1) | 0.6 (0.1)
  Scaling Lower limbs, Week 8 (n=30,70,43,104) | 0.3 (0.2) | 0.9 (0.1) | -0.0 (0.1) | 0.9 (0.1)
  Scaling Lower limbs, Week 12 (n=28,53,42,84) | 0.2 (0.2) | 0.9 (0.1) | 0.0 (0.1) | 0.9 (0.1)
  Scaling Lower limbs, Week 16 (n=28,45,38,70) | 0.2 (0.2) | 1.0 (0.1) | 0.3 (0.2) | 1.0 (0.1)

48. Secondary Outcome: Mean Change From Baseline in PASI Component Scores During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 39
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 74 | 42 | 119
score on a scale
  Erythema Head/Neck, Week 4 (n=27,74,42,119) | -0.1 (0.1) | -0.4 (0.1) | 0.1 (0.1) | -0.9 (0.1)
  Erythema Head/Neck, Week 8 (n=26,72,41,118) | 0.1 (0.1) | -0.7 (0.1) | -0.0 (0.1) | -0.9 (0.1)
  Erythema Head/Neck, Week 16 (n=23,67,39,101) | -0.1 (0.1) | -0.4 (0.1) | -0.1 (0.1) | -0.9 (0.1)
  Induration Head/Neck, Week 4 (n=27,74,42,119) | -0.2 (0.1) | -0.4 (0.1) | 0.0 (0.1) | -0.8 (0.1)
  Induration Head/Neck, Week 8 (n=26,72,41,118) | -0.0 (0.2) | -0.5 (0.1) | -0.0 (0.1) | -0.8 (0.1)
  Induration Head/Neck, Week 16 (n=23,67,39,101) | -0.1 (0.1) | -0.6 (0.1) | -0.2 (0.1) | -0.9 (0.1)
  Scaling Head/Neck, Week 4 (n=27,74,42,119) | -0.1 (0.1) | -0.4 (0.1) | 0.0 (0.1) | -0.9 (0.1)
  Scaling Head/Neck, Week 8 (n=26,72,41,118) | 0.1 (0.1) | -0.5 (0.1) | -0.0 (0.1) | -0.9 (0.1)
  Scaling Head/Neck, Week 16 (n=23,67,39,101) | -0.1 (0.1) | -0.5 (0.1) | -0.2 (0.1) | -1.0 (0.1)
  Erythema Upper limbs, Week 4 (n=27,74,42,119) | -0.0 (0.1) | -0.4 (0.1) | -0.0 (0.1) | -0.6 (0.1)
  Erythema Upper limbs, Week 8 (n=26,72,41,118) | -0.1 (0.1) | -0.7 (0.1) | -0.1 (0.1) | -0.8 (0.1)
  Erythema Upper limbs, Week 16 (n=23,67,39,101) | 0.0 (0.2) | -0.6 (0.1) | -0.2 (0.2) | -0.8 (0.1)
  Induration Upper limbs, Week 4 (n=27,74,42,119) | -0.0 (0.1) | -0.5 (0.1) | -0.0 (0.1) | -0.6 (0.1)
  Induration Upper limbs, Week 8 (n=26,72,41,118) | -0.0 (0.1) | -0.7 (0.1) | -0.1 (0.1) | -0.8 (0.1)
  Induration Upper limbs, Week 16 (n=23,67,39,101) | -0.0 (0.2) | -0.6 (0.1) | -0.1 (0.2) | -0.8 (0.1)
  Scaling Upper limbs, Week 4 (n=27,74,42,119) | 0.0 (0.1) | -0.3 (0.1) | -0.2 (0.1) | -0.7 (0.1)
  Scaling Upper limbs, Week 8 (n=26,72,41,118) | -0.0 (0.2) | -0.6 (0.1) | -0.1 (0.1) | -0.8 (0.1)
  Scaling Upper limbs, Week 16 (n=23,67,39,101) | 0.0 (0.2) | -0.5 (0.1) | -0.2 (0.2) | -0.8 (0.1)
  Erythema Trunk, Week 4 (n=27,74,42,119) | -0.1 (0.1) | -0.5 (0.1) | -0.1 (0.1) | -0.8 (0.1)
  Erythema Trunk, Week 8 (n=26,72,41,118) | -0.1 (02) | -0.7 (01) | 0.0 (0.2) | -1.0 (0.1)
  Erythema Trunk, Week 16 (n=23,67,39,101) | -0.2 (0.2) | -0.8 (0.1) | -0.1 (0.2) | -1.0 (0.1)
  Induration Trunk, Week 4 (n=27,74,42,119) | -0.1 (0.1) | -0.5 (0.1) | -0.1 (0.1) | -0.7 (0.1)
  Induration Trunk, Week 8 (n=26,72,41,118) | -0.1 (0.1) | -0.7 (0.1) | -0.2 (0.1) | -0.8 (0.1)
  Induration Trunk, Week 16 (n=23,67,39,101) | -0.2 (0.2) | -0.8 (0.1) | -0.2 (0.2) | -0.8 (0.1)
  Scaling Trunk, Week 4 (n=27,74,42,119) | -0.2 (0.2) | -0.4 (0.1) | -0.1 (0.1) | -0.6 (0.1)
  Scaling Trunk, Week 8 (n=26,72,41,118) | 0.0 (0.1) | -0.6 (0.1) | -0.1 (0.1) | -0.8 (0.1)
  Scaling Trunk, Week 16 (n=23,67,39,101) | -0.3 (0.2) | -0.7 (0.1) | -0.1 (0.1) | -0.8 (0.1)
  Erythema Lower limbs, Week 4 (n=27,74,42,119) | 0.0 (0.1) | -0.5 (0.1) | -0.1 (0.1) | -0.7 (0.1)
  Erythema Lower limbs, Week 8 (n=26,72,41,118) | 0.1 (0.1) | -0.7 (0.1) | -0.2 (0.1) | -0.9 (0.1)
  Erythema Lower limbs, Week 16 (n=23,67,39,101) | 0.2 (0.2) | -0.7 (0.1) | -0.2 (0.2) | -1.0 (0.1)
  Induration Lower limbs, Week 4 (n=27,74,42,119) | 0.2 (0.1) | -0.4 (0.1) | -0.1 (0.1) | -0.7 (0.1)
  Induration Lower limbs, Week 8 (n=26,72,41,118) | 0.1 (0.2) | -0.6 (0.1) | -0.1 (0.1) | -0.8 (0.1)
  Induration Lower limbs, Week 16 (n=23,67,39,101) | 0.3 (0.2) | -0.7 (0.1) | -0.1 (0.2) | -0.9 (0.1)
  Scaling Lower limbs, Week 4 (n=27,74,42,119) | 0.1 (0.1) | -0.3 (0.1) | -0.1 (0.1) | -0.7 (0.1)
  Scaling Lower limbs, Week 8 (n=26,72,41,118) | 0.1 (0.2) | -0.6 (0.1) | -0.1 (0.1) | -0.8 (0.1)
  Scaling Lower limbs, Week 16 (n=23,67,39,101) | 0.3 (0.2) | -0.6 (0.1) | -0.2 (0.2) | -0.9 (0.1)

49. Secondary Outcome: Percentage of Participants Achieving at Least a 50% Reduction in PASI Relative to Baseline-A (PASI50) During Period A
Description: PASI quantifies the severity of psoriasis based on both lesion severity and the percent of BSA) affected. PASI is a composite score by the investigator of degree of erythema, induration, and scaling (scored separately) for each of 4 body regions (head and neck, upper limbs, trunk, and lower limbs), with adjustment for percent of BSA involved for each body region and for proportion of the body region to the whole body. PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A; NRI
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
percentage of participants
  Week 4 | 28.70 [23.83 to 33.57] | 54.63 [49.30 to 59.96]
  Week 8 | 55.29 [49.93 to 60.64] | 75.52 [70.92 to 80.13]
  Week 16 | 65.26 [60.13 to 70.39] | 79.40 [75.07 to 83.73]
  Week 24 | 59.52 [54.23 to 64.80] | 73.13 [68.39 to 77.88]

50. Secondary Outcome: Percentage of Participants Achieving at Least a 90% Reduction in PASI Relative to Baseline-A (PASI90) During Period A
Description: as for outcome 49
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
percentage of participants
  Week 4 | 1.21 [0.03 to 2.39] | 6.27 [3.67 to 8.86]
  Week 8 | 8.76 [5.72 to 11.81] | 24.78 [20.15 to 29.40]
  Week 16 | 18.73 [14.53 to 22.93] | 36.72 [31.55 to 41.88]
  Week 24 | 20.24 [15.91 to 24.57] | 37.31 [32.13 to 42.49]

51. Secondary Outcome: Percentage of Participants Achieving at Least a 100% Reduction in PASI Relative to Baseline-A (PASI100) During Period A
Description: as for outcome 49
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
percentage of participants
  Week 4 | 0.91 [0.0 to 1.93] | 2.09 [0.56 to 3.62]
  Week 8 | 2.72 [0.97 to 4.47] | 7.46 [4.65 to 10.28]
  Week 16 | 7.25 [4.46 to 10.04] | 15.82 [11.91 to 19.73]
  Week 24 | 8.16 [5.21 to 11.11] | 17.31 [13.26 to 21.37]

52. Secondary Outcome: Percentage of Participants Achieving at Least a 50% Reduction in PASI Relative to Baseline-A (PASI50) During the CP-690,550 Re-Treatment (Period C)
Description: PASI quantifies severity of psoriasis based on both lesion severity and percent of BSA affected. PASI is a composite score by investigator of degree of erythema, induration, and scaling (scored separately) for each of 4 body regions (head/neck, upper limbs, trunk, lower limbs), with adjustment for percent of BSA involved for each body region and for proportion of body region to the whole body. PASI score can vary in increments of 0.1 and range from 0.0-72.0; higher scores representing greater severity of psoriasis. Baseline-A defined as last observation up to first dosing date in Period A.
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
percentage of participants
  Baseline | 96.30 [89.17 to 100.00] | 42.67 [31.47 to 53.86] | 92.86 [85.07 to 100.00] | 49.17 [40.22 to 58.11]
  Week 4 | 100.00 [100.00 to 100.00] | 69.33 [58.90 to 79.77] | 92.86 [85.07 to 100.00] | 84.17 [77.64 to 90.70]
  Week 8 | 92.59 [82.71 to 100.00] | 81.33 [72.52 to 90.15] | 95.24 [88.80 to 100.00] | 89.17 [83.61 to 94.73]
  Week 16 | 85.19 [71.79 to 98.58] | 82.67 [74.10 to 91.23] | 85.71 [75.13 to 96.30] | 79.17 [71.90 to 86.43]

53. Secondary Outcome: Percentage of Participants Achieving at Least a 90% Reduction in PASI Relative to Baseline-A (PASI90) During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 52
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
percentage of participants
  Baseline | 48.15 [29.30 to 66.99] | 12.00 [4.65 to 19.35] | 45.24 [30.19 to 60.29] | 15.83 [9.30 to 22.36]
  Week 4 | 48.15 [29.30 to 66.99] | 17.33 [8.77 to 25.90] | 47.62 [32.51 to 62.72] | 35.00 [26.47 to 43.53]
  Week 8 | 48.15 [29.3 to 66.99] | 21.33 [12.06 to 30.60] | 47.62 [32.51 to 62.72] | 42.50 [33.66 to 51.34]
  Week 16 | 33.33 [15.55 to 51.11] | 21.33 [12.06 to 30.60] | 45.24 [30.19 to 60.29] | 44.17 [35.28 to 53.05]

54. Secondary Outcome: Percentage of Participants Achieving 100% Reduction in PASI Relative to Baseline-A (PASI100) During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 52
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
percentage of participants
  Baseline | 18.52 [3.87 to 33.17] | 5.33 [0.25 to 10.42] | 23.81 [10.93 to 36.69] | 5.00 [1.10 to 8.90]
  Week 4 | 18.52 [3.87 to 33.17] | 9.33 [2.75 to 15.92] | 21.43 [9.02 to 33.84] | 15.00 [8.61 to 21.39]
  Week 8 | 18.52 [3.87 to 33.17] | 13.33 [5.64 to 21.03] | 21.43 [9.02 to 33.84] | 19.17 [12.12 to 26.21]
  Week 16 | 14.81 [1.42 to 28.21] | 10.67 [3.68 to 17.65] | 26.19 [12.89 to 39.49] | 20.83 [13.57 to 28.10]

55. Secondary Outcome: Percentage of Participants With a PASI Score ≥125% of the Baseline-A PASI Score During Initial CP-690,550 Treatment (Period A)
Description: PASI quantifies the severity of psoriasis based on both lesion severity and percent of BSA affected. PASI is a composite score by the investigator of degree of erythema, induration, and scaling (scored separately) for each of 4 body regions (head and neck, upper limbs, trunk, and lower limbs), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0-72.0; higher scores representing greater severity of psoriasis.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 329 | 333
percentage of participants
  Week 4 (n=326,331) | 0.92 [0.00 to 1.96] | 0.60 [0.00 to 1.44]
  Week 8 (n=322,323) | 0.62 [0.00 to 1.48] | 0.62 [0.00 to 1.47]
  Week 16 (n=311,307) | 0.96 [0.00 to 2.05] | 0.98 [0.00 to 2.08]
  Week 24 (n=277,279) | 1.08 [0.00 to 2.30] | 0.36 [0.00 to 1.06]
  Overall (n=329,333) | 2.13 [0.57 to 3.69] | 2.10 [0.56 to 3.64]

56. Secondary Outcome: Percentage of Participants With a PASI Score ≥125% of the Baseline-A PASI Score During Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 52
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 132
percentage of participants
  Week 4 (n=30,82,43,128) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 8 (n=30,70,43,104) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 12 (n=28,53,42,84) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [-3.51 to 1.13] | 1.19
  Week 16 (n=28,45,38,70) | 0.00 | 0.00 | 0.00 | 0.00
  Overall (n=31,82,45,132) | 0.00 | 0.00 | 0.00 | 0.76

57. Secondary Outcome: Percentage of Participants With a PASI Score ≥125% of the Baseline-A PASI Score During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 52
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
percentage of participants
  Week 4 (n=27,74,42,119) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 8 (n=26,72,41,118) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 16 (n=23,67,39,101) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 2.56 [0.00 to 7.52] | 0.00 [0.00 to 0.00]
  Overall (n=27,75,42,120) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 2.38 [0.00 to 6.99] | 0.00 [0.00 to 0.00]

58. Secondary Outcome: Mean Itch Severity Item (ISI) Score During the Initial CP-690,550 Treatment (Period A)
Description: The severity of itch (pruritus) due to psoriasis was assessed using the ISI, a single item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends.
Time Frame: Baseline and Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
score on a scale
  Baseline (n=331,335) | 6.7 (0.1) | 6.9 (0.1)
  Week 4 (n=326,331) | 3.2 (0.1) | 2.2 (0.1)
  Week 8 (n=322,321) | 2.8 (0.1) | 1.6 (0.1)
  Week 16 (n=310,307) | 2.9 (0.2) | 1.7 (0.1)
  Week 24 (n=274,278) | 2.9 (0.2) | 1.6 (0.1)

59. Secondary Outcome: Mean ISI Score During the Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 58
Time Frame: Baseline and Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
score on a scale
  Baseline (n=31,82,45,133) | 1.5 (0.4) | 1.2 (0.2) | 0.6 (0.2) | 0.8 (0.1)
  Week 4 (n=30,82,43,127) | 1.7 (0.4) | 3.6 (0.3) | 0.7 (0.2) | 4.1 (0.3)
  Week 8 (n=30,69,43,104) | 1.5 (0.4) | 4.0 (0.4) | 1.2 (0.3) | 4.1 (0.3)
  Week 12 (n=29,53,41,84) | 1.9 (0.4) | 4.0 (0.4) | 1.3 (0.3) | 3.8 (0.3)
  Week 16 (n=28,45,38,70) | 2.2 (0.5) | 3.7 (0.4) | 1.6 (0.4) | 4.0 (0.4)

60. Secondary Outcome: Mean ISI Score During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 58
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
score on a scale
  Baseline (n=27,75,42,120) | 2.3 (0.5) | 4.9 (0.3) | 1.7 (0.4) | 5.2 (0.3)
  Week 4 (n=27,74,42,119) | 2.6 (0.5) | 2.6 (0.2) | 1.7 (0.4) | 2.1 (0.2)
  Week 8 (n=26,72,41,118) | 2.4 (0.5) | 2.3 (0.2) | 1.5 (0.3) | 1.8 (0.2)
  Week 16 (n=23,67,39,100) | 2.3 (0.5) | 2.2 (0.3) | 1.4 (0.4) | 1.6 (0.2)

61. Secondary Outcome: Mean Change From Baseline-A in ISI Score During the Initial CP-690,550 Treatment (Period A)
Description: The severity of itch (pruritus) due to psoriasis was assessed using the ISI, a single item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends. Baseline-A defined as the last observation up to first dosing date in Period A.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 326 | 331
score on a scale
  Week 4 (n=326,331) | -3.6 (0.1) | -4.6 (0.2)
  Week 8 (n=322,321) | -3.9 (0.2) | -5.3 (0.2)
  Week 16 (n=310,307) | -3.8 (0.2) | -5.2 (0.2)
  Week 24 (n=274,278) | -3.7 (0.2) | -5.3 (0.2)

62. Secondary Outcome: Mean Change From Baseline-B in ISI Score During the Double-Blind Treatment Withdrawal (Period B)
Description: The severity of itch (pruritus) due to psoriasis was assessed using the ISI, a single item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends. Baseline-B defined as the last observation up to first dosing date in Period B.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 30 | 82 | 43 | 127
score on a scale
  Week 4 (n=30,82,43,127) | 0.2 (0.3) | 2.4 (0.3) | 0.1 (0.2) | 3.3 (0.3)
  Week 8 (n=30,69,43,104) | -0.0 (0.3) | 2.9 (0.3) | 0.6 (0.2) | 3.4 (0.3)
  Week 12 (n=29,53,41,84) | 0.3 (0.2) | 2.8 (0.3) | 0.7 (0.2) | 3.2 (0.3)
  Week 16 (n=28,45,38,70) | 0.6 (0.3) | 2.7 (0.4) | 0.9 (0.3) | 3.6 (0.4)

63. Secondary Outcome: Mean Change From Baseline-C in ISI Score During the CP-690,550 Re-Treatment (Period C)
Description: The severity of itch (pruritus) due to psoriasis was assessed using the ISI, a single item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends. Baseline-C defined as the last observation up to first dosing date in Period C.
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 74 | 42 | 119
score on a scale
  Week 4 (n=27,74,42,119) | 0.3 (0.4) | -2.3 (0.3) | 0.0 (0.2) | -3.1 (0.3)
  Week 8 (n=26,72,41,118) | 0.1 (0.4) | -2.6 (0.3) | -0.2 (0.2) | -3.4 (0.3)
  Week 16 (n=23,67,39,100) | 0.4 (0.4) | -2.6 (0.4) | -0.3 (0.3) | -3.6 (0.3)

64. Secondary Outcome: Percentage of Participants With ISI Score of 0 During the Initial CP-690,550 Treatment (Period A)
Description: as for outcome 58
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A participants with a Baseline-A ISI greater than (>) 0, where Baseline-A is defined as the last observation up to first dosing date in Period A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 325 | 327
percentage of participants
  Week 4 | 12.92 [9.28 to 16.57] | 25.69 [20.95 to 30.42]
  Week 8 | 16.92 [12.85 to 21.00] | 41.28 [35.95 to 46.62]
  Week 16 | 20.00 [15.65 to 24.35] | 37.92 [32.66 to 43.18]
  Week 24 | 19.38 [15.09 to 23.68] | 37.31 [32.07 to 42.55]

65. Secondary Outcome: Percentage of Participants With ISI Score of 0 During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 58
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C participants with a Baseline-C ISI greater than (>) 0, where Baseline-C is defined as the last observation up to first dosing date in Period C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 18 | 71 | 27 | 104
percentage of participants
  Baseline | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 4 | 0.00 [0.00 to 0.00] | 11.27 [3.91 to 18.62] | 7.41 [0.00 to 17.29] | 23.08 [14.98 to 31.17]
  Week 8 | 5.56 [0.00 to 16.14] | 18.31 [9.31 to 27.31] | 18.52 [3.87 to 33.17] | 38.46 [29.11 to 47.81]
  Week 16 | 11.11 [0.00 to 25.63] | 15.49 [7.08 to 23.91] | 25.93 [9.40 to 42.46] | 28.85 [20.14 to 37.55]

66. Secondary Outcome: Percentage of Participants Achieving ISI Score of ≤1 During the Initial CP-690,550 Treatment (Period A)
Description: as for outcome 58
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A participants with a Baseline-A ISI >1, where Baseline-A is defined as the last observation up to first dosing date in Period A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 315 | 315
percentage of participants
  Week 4 | 27.62 [22.68 to 32.56] | 46.03 [40.53 to 51.54]
  Week 8 | 34.29 [29.04 to 39.53] | 60.00 [54.59 to 65.41]
  Week 16 | 34.92 [29.66 to 40.19] | 60.00 [54.59 to 65.41]
  Week 24 | 31.11 [26.00 to 36.22] | 55.24 [49.75 to 60.73]

67. Secondary Outcome: Percentage of Participants Achieving an ISI Score of ≤1 During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 58
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C participants with a Baseline-C ISI >1, where Baseline-C is defined as the last observation up to first dosing date in Period C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 14 | 62 | 14 | 95
percentage of participants
  Baseline | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 4 | 14.29 [0.00 to 32.62] | 22.58 [12.17 to 32.99] | 14.29 [0.00 to 32.62] | 41.05 [31.16 to 50.94]
  Week 8 | 21.43 [0.00 to 42.92] | 33.87 [22.09 to 45.65] | 21.43 [0.00 to 42.92] | 55.79 [45.80 to 65.78]
  Week 16 | 21.43 [0.00 to 42.92] | 41.94 [29.65 to 54.22] | 35.71 [10.61 to 60.81] | 50.53 [40.47 to 60.58]

68. Secondary Outcome: Percentage of Participants Achieving ISI ≥2-Point Reduction During the Initial CP-690,550 Treatment (Period A)
Description: as for outcome 58
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A participants with a Baseline-A ISI ≥2, where Baseline-A is defined as the last observation up to first dosing date in Period A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 315 | 315
percentage of participants
  Week 4 | 81.59 [77.31 to 85.87] | 88.89 [85.42 to 92.36]
  Week 8 | 80.32 [75.93 to 84.71] | 87.94 [84.34 to 91.53]
  Week 16 | 73.97 [69.12 to 78.81] | 84.76 [80.79 to 88.73]
  Week 24 | 65.71 [60.47 to 70.96] | 74.92 [70.13 to 79.71]

69. Secondary Outcome: Percentage of Participants Achieving ISI ≥2-Point Reduction During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 58
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C participants with a Baseline-C ISI ≥2, where Baseline-C is defined as the last observation up to first dosing date in Period C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 14 | 62 | 14 | 95
percentage of participants
  Week 4 | 28.57 [4.91 to 52.24] | 61.29 [49.17 to 73.41] | 14.29 [0.00 to 32.62] | 80.00 [71.96 to 88.04]
  Week 8 | 28.57 [4.91 to 52.24] | 64.52 [52.61 to 76.43] | 28.57 [4.91 to 52.24] | 78.95 [70.75 to 87.15]
  Week 16 | 21.43 [0.00 to 42.92] | 62.90 [50.88 to 74.93] | 28.57 [4.91 to 52.24] | 69.47 [60.21 to 78.73]

70. Secondary Outcome: ISI Score of ≤1 During the Initial CP-690,550 Treatment (Period A) - Percentage of Participants With a Response
Description: as for outcome 58
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A participants with Baseline-A ISI >1, where Baseline-A was defined as the last observation before the first dosing date in Period A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 315 | 315
percentage of participants
  Week 4 | 27.8 [23.2 to 33.2] | 47.2 [41.8 to 52.9]
  Week 8 | 41.2 [36.0 to 46.9] | 67.8 [62.5 to 72.9]
  Week 16 | 52.4 [46.8 to 58.2] | 78.6 [73.7 to 83.1]
  Week 24 | 72.4 [55.1 to 87.3] | 83.4 [77.9 to 88.2]

71. Secondary Outcome: Median Time to ISI Score of ≤1 During the Initial CP-690,550 Treatment (Period A)
Description: as for outcome 58
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: as for outcome 70
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 313 | 313
weeks | 16.4 [16.1 to 24.6] | 8.0 [5.1 to 8.1]

72. Secondary Outcome: ISI Score of ≤1 During CP-690,550 Re-Treatment (Period C) - Percentage of Participants With a Response
Description: as for outcome 58
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: as for outcome 67
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 14 | 62 | 14 | 95
percentage of participants
  Week 4 | 14.3 [3.8 to 46.1] | 22.8 [14.2 to 35.5] | 14.3 [3.8 to 46.1] | 41.3 [32.1 to 51.9]
  Week 8 | 28.6 [11.8 to 59.4] | 37.9 [27.0 to 51.4] | 21.4 [7.5 to 52.8] | 59.8 [50.0 to 69.7]
  Week 16 | 40.5 [18.3 to 73.5] | 79.1 [46.8 to 98.0] | 49.5 [21.8 to 85.0] | 90.3 [69.9 to 98.9]

73. Secondary Outcome: Median Time to ISI Score of ≤1 During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 58
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C participants with Baseline-C ISI >1, where Baseline-C defined as the last observation up to first dosing date in Period C.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 14 | 62 | 14 | 95
weeks | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 16.1 [10.1 to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 8.3 [6.0 to 12.4]

74. Secondary Outcome: ISI Reduction (2-point Decrease in ISI Score) During the Initial CP-690,550 Treatment (Period A) - Percentage of Participants With a Response
Description: as for outcome 58
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A participants with Baseline-A ISI ≥2, where Baseline-A was defined as the last observation before the first dosing date in Period A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 315 | 315
percentage of participants
  Week 4 | 82.2 [77.8 to 86.2] | 90.3 [86.7 to 93.3]
  Week 8 | 89.5 [85.8 to 92.6] | 96.5 [94.0 to 98.2]
  Week 16 | 93.6 [90.5 to 96.0] | 97.8 [95.5 to 99.1]
  Week 24 | 96.2 [92.5 to 98.4] | 97.8 [95.5 to 99.1]

75. Secondary Outcome: Median Time to ISI Reduction (2-point Decrease in ISI Score) During the Initial CP-690,550 Treatment (Period A)
Description: as for outcome 58
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: as for outcome 74
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 313 | 313
weeks | 4.1 [NA to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 4.1 [NA to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue.

76. Secondary Outcome: ISI Reduction (2-point Decrease in ISI Score) During the CP-690,550 Re-Treatment (Period C) - Percentage of Participant With a Response
Description: as for outcome 58
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C participants with Baseline-C ISI ≥2, where Baseline-C defined as the last observation up to first dosing date in Period C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 14 | 62 | 14 | 95
percentage of participants
  Week 4 | 28.6 [11.8 to 59.4] | 61.8 [49.9 to 73.8] | 14.3 [3.8 to 46.1] | 80.0 [71.5 to 87.3]
  Week 8 | 35.7 [16.7 to 65.7] | 75.1 [63.8 to 85.1] | 28.6 [11.8 to 59.4] | 86.7 [78.9 to 92.6]
  Week 16 | 57.1 [25.6 to 91.1] | 100.0 [NA to NA] — 95% confidence interval could not be estimated due to censoring. | 36.5 [17.0 to 66.9] | 91.0 [83.6 to 95.9]

77. Secondary Outcome: Median Time to ISI Reduction (2-point Decrease in ISI Score) During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 58
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: as for outcome 73
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 14 | 62 | 14 | 95
weeks | 16.6 [4.4 to NA] — 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 4.9 [4.3 to 7.1] | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 4.3 [4.1 to 4.4]

78. Secondary Outcome: Mean Dermatology Life Quality Index (DLQI) Score During the Initial CP-690,550 Treatment (Period A)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life.
Time Frame: Baseline and Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 330 | 333
score on a scale
  Baseline (n=330,333) | 12.6 (0.4) | 12.6 (0.4)
  Week 4 (n=326,330) | 6.8 (0.3) | 4.8 (0.3)
  Week 8 (n=321,319) | 5.4 (0.3) | 3.4 (0.3)
  Week 16 (n=310,303) | 4.7 (0.3) | 2.9 (0.3)
  Week 24 (n=273,277) | 5.1 (0.4) | 2.6 (0.3)

79. Secondary Outcome: Mean DLQI Score During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 78
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
score on a scale
  Baseline (n=27,75,42,120) | 3.6 (1.0) | 7.0 (0.8) | 2.2 (0.5) | 8.8 (0.7)
  Week 4 (n=27,74,42,119) | 3.4 (1.0) | 4.3 (0.5) | 2.2 (0.5) | 3.9 (0.4)
  Week 8 (n=26,71,41,118) | 3.9 (1.3) | 3.1 (0.4) | 2.2 (0.5) | 2.7 (0.4)
  Week 16 (n=22,66,39,101) | 3.0 (1.0) | 3.4 (0.5) | 2.1 (0.7) | 2.4 (0.4)

80. Secondary Outcome: Mean DLQI Score During the Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 78
Time Frame: Baseline and Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
score on a scale
  Baseline (n=31,82,45,133) | 2.6 (0.7) | 1.8 (0.3) | 1.2 (0.3) | 1.2 (0.2)
  Week 4 (n=30,82,43,127) | 3.4 (0.9) | 4.7 (0.5) | 1.3 (0.4) | 5.9 (0.6)
  Week 8 (n=30,68,43,104) | 3.1 (0.9) | 5.9 (0.8) | 1.6 (0.5) | 6.4 (0.7)
  Week 12 (n=28,52,41,83) | 3.3 (1.1) | 4.7 (0.6) | 1.9 (0.4) | 5.3 (0.7)
  Week 16 (n=28,44,38,68) | 3.5 (1.0) | 5.0 (0.7) | 2.0 (0.4) | 6.2 (0.8)

81. Secondary Outcome: Mean Change From Baseline-A in DLQI Score During the Initial CP-690,550 Treatment (Period A)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life. The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline. Baseline-A defined as the last observation up to first dosing date in Period A.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 325 | 328
scores on a scale
  Week 4 (n=325,328) | -5.8 (0.3) | -7.6 (0.3)
  Week 8 (n=320,317) | -7.1 (0.3) | -9.1 (0.4)
  Week 16 (n=309,301) | -7.6 (0.4) | -9.4 (0.4)
  Week 24 (n=272,275) | -7.1 (0.4) | -9.7 (0.4)

82. Secondary Outcome: Mean Change From Baseline-B in DLQI Score During the Double-Blind Treatment Withdrawal (Period B)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life. The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline. Baseline-B defined as the last observation up to first dosing date in Period B.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 30 | 82 | 43 | 127
scores on a scale
  Week 4 (n=30,82,43,127) | 0.8 (0.7) | 3.0 (0.5) | 0.1 (0.3) | 4.6 (0.5)
  Week 8 (n=30,68,43,104) | 0.5 (0.3) | 4.1 (0.7) | 0.3 (0.5) | 5.4 (0.6)
  Week 12 (n=28,52,41,83) | 0.9 (0.5) | 3.4 (0.5) | 0.6 (0.4) | 4.5 (0.7)
  Week 16 (n=28,44,38,68) | 1.1 (0.5) | 3.6 (0.6) | 0.5 (0.3) | 5.4 (0.8)

83. Secondary Outcome: Mean Change From Baseline-C in DLQI Score During the CP-690,550 Re-Treatment (Period C)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life. The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline. Baseline-C defined as the last observation up to first dosing date in Period C.
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals number of participants with an observation
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 74 | 42 | 119
scores on a scale
  Week 4 (n=27,74,42,119) | -0.2 (0.2) | -2.9 (0.5) | 0.0 (0.4) | -4.9 (0.6)
  Week 8 (n=26,71,41,118) | 0.2 (0.4) | -3.4 (0.5) | -0.0 (0.5) | -5.9 (0.6)
  Week 16 (n=22,66,39,101) | 0.5 (0.8) | -3.3 (0.8) | -0.0 (0.7) | -6.3 (0.7)

84. Secondary Outcome: Mean DLQI Subscale Scores During the Initial CP-690,550 Treatment (Period A)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much); higher scores indicate poor quality of life. The DLQI can be analyzed under 6 subscales by combining questions and is categorized as follows: symptoms and feelings (maximum score=6); daily activities (maximum score=6); leisure (maximum score=6); work and school (maximum score=3); personal relationships (maximum score=6); and treatment (maximum score=3).
Time Frame: Baseline and Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 330 | 333
score on a scale
  Daily Activities, Baseline (n=330,333) | 2.7 (0.10) | 2.7 (0.10)
  Daily Activities, Week 4 (n=326,330) | 1.5 (0.09) | 1.1 (0.07)
  Daily Activities, Week 8 (n=321,320) | 1.2 (0.08) | 0.8 (0.07)
  Daily Activities, Week 16 (n=310,303) | 1.0 (0.08) | 0.6 (0.07)
  Daily Activities, Week 24 (n=273,277) | 1.1 (0.09) | 0.6 (0.07)
  Personal Relationships, Baseline (n=331,332) | 1.7 (0.10) | 1.7 (0.10)
  Personal Relationships, Week 4 (n=326,330) | 1.0 (0.08) | 0.6 (0.07)
  Personal Relationships, Week 8 (n=321,318) | 0.7 (0.06) | 0.4 (0.06)
  Personal Relationships, Week 16 (n=310,302) | 0.6 (0.06) | 0.3 (0.06)
  Personal Relationships, Week 24 (n=271,276) | 0.6 (0.07) | 0.3 (0.05)
  Symptoms and Feelings, Baseline (n=331,333) | 3.9 (0.09) | 3.9 (0.08)
  Symptoms and Feelings, Week 4 (n=326,330) | 2.1 (0.07) | 1.6 (0.07)
  Symptoms and Feelings, Week 8 (n=321,319) | 1.8 (0.08) | 1.2 (0.07)
  Symptoms and Feelings, Week 16 (n=310,303) | 1.7 (0.08) | 1.1 (0.08)
  Symptoms and Feelings, Week 24 (n=273,277) | 1.7 (0.09) | 1.0 (0.08)
  Leisure, Baseline (n=331,333) | 2.1 (0.11) | 2.2 (0.11)
  Leisure, Week 4 (n=326,330) | 1.1 (0.09) | 0.8 (0.07)
  Leisure, Week 8 (n=321,320) | 0.9 (0.08) | 0.5 (0.06)
  Leisure, Week 16 (n=310,303) | 0.7 (0.07) | 0.4 (0.06)
  Leisure, Week 24 (n=272,277) | 0.8 (0.08) | 0.4 (0.05)
  Work and School, Baseline (n=330,333) | 0.9 (0.06) | 0.9 (0.06)
  Work and School, Week 4 (n=326,330) | 0.5 (0.05) | 0.3 (0.04)
  Work and School, Week 8 (n=321,319) | 0.3 (0.04) | 0.2 (0.03)
  Work and School, Week 16 (n=309,303) | 0.3 (0.04) | 0.2 (0.03)
  Work and School, Week 24 (n=273,277) | 0.4 (0.04) | 0.1 (0.03)
  Treatment, Baseline (n=331,332) | 1.1 (0.06) | 1.2 (0.06)
  Treatment, Week 4 (n=326,330) | 0.6 (0.04) | 0.5 (0.04)
  Treatment, Week 8 (n=321,320) | 0.5 (0.04) | 0.4 (0.03)
  Treatment, Week 16 (n=310,303) | 0.5 (0.04) | 0.3 (0.04)
  Treatment, Week 24 (n=272,277) | 0.6 (0.05) | 0.2 (0.03)

85. Secondary Outcome: Mean DLQI Subscale Scores During the Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 84
Time Frame: Baseline and Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
score on a scale
  Daily Activities, Baseline (n=31,82,45,133) | 0.5 (0.18) | 0.3 (0.07) | 0.2 (0.07) | 0.3 (0.07)
  Daily Activities, Week 4 (n=30,82,43,127) | 0.8 (0.30) | 0.8 (0.14) | 0.3 (0.09) | 1.2 (0.14)
  Daily Activities, Week 8 (n=30,68,43,104) | 0.6 (0.25) | 1.1 (0.19) | 0.4 (0.13) | 1.2 (0.17)
  Daily Activities, Week 12 (n=28,52,41,83) | 0.6 (0.23) | 0.9 (0.15) | 0.3 (0.10) | 1.1 (0.17)
  Daily Activities, Week 16 (n=28,44,38,68) | 0.6 (0.22) | 1.2 (0.21) | 0.4 (0.12) | 1.3 (0.21)
  Personal Relationships, Baseline (n=31,82,45,133) | 0.3 (0.13) | 0.2 (0.06) | 0.2 (0.08) | 0.1 (0.04)
  Personal Relationships, Week 4 (n=30,82,43,126) | 0.4 (0.19) | 0.6 (0.11) | 0.1 (0.05) | 0.6 (0.10)
  Personal Relationships, Week 8 (n=30,68,43,103) | 0.4 (0.22) | 0.8 (0.17) | 0.1 (0.07) | 0.9 (0.14)
  Personal Relationships, Week 12 (n=28,52,41,83) | 0.4 (0.23) | 0.6 (0.15) | 0.1 (0.05) | 0.7 (0.13)
  Personal Relationships, Week 16 (n=28,44,38,68) | 0.4 (0.23) | 0.5 (0.16) | 0.2 (0.07) | 0.8 (0.17)
  Symptoms and Feelings, Baseline (n=31,82,45,133) | 1.1 (0.25) | 0.8 (0.10) | 0.5 (0.10) | 0.6 (0.08)
  Symptoms and Feelings, Week 4 (n=30,82,43,127) | 1.3 (0.30) | 2.0 (0.19) | 0.5 (0.13) | 2.2 (0.16)
  Symptoms and Feelings, Week 8 (n=30,68,43,104) | 1.1 (0.24) | 2.2 (0.19) | 0.7 (0.16) | 2.3 (0.18)
  Symptoms and Feelings, Week 12 (n=28,52,41,83) | 1.1 (0.28) | 2.1 (0.19) | 1.0 (0.19) | 2.0 (0.18)
  Symptoms and Feelings, Week 16 (n=28,44,38,68) | 1.4 (0.31) | 1.9 (0.19) | 1.0 (0.16) | 2.2 (0.21)
  Leisure, Baseline (n=31,82,45,133) | 0.3 (0.12) | 0.2 (0.07) | 0.2 (0.08) | 0.2 (0.05)
  Leisure, Week 4 (n=30,82,42,127) | 0.5 (0.23) | 0.6 (0.11) | 0.1 (0.08) | 0.9 (0.13)
  Leisure, Week 8 (n=30,68,43,104) | 0.5 (0.15) | 0.8 (0.18) | 0.2 (0.11) | 0.9 (0.15)
  Leisure, Week 12 (n=28,52,41,83) | 0.5 (0.18) | 0.5 (0.14) | 0.2 (0.07) | 0.7 (0.14)
  Leisure, Week 16 (n=28,44,37,68) | 0.5 (0.17) | 0.5 (0.15) | 0.1 (0.07) | 0.9 (0.17)
  Work and School, Baseline (n=31,82,45,133) | 0.1 (0.04) | 0.1 (0.05) | 0.0 (0.02) | 0.1 (0.02)
  Work and School, Week 4 (n=30,82,43,127) | 0.1 (0.06) | 0.3 (0.07) | 0.0 (0.02) | 0.5 (0.09)
  Work and School, Week 8 (n=30,68,43,104) | 0.2 (0.08) | 0.3 (0.09) | 0.0 (0.03) | 0.5 (0.09)
  Work and School, Week 12 (n=28,52,41,83) | 0.2 (0.13) | 0.2 (0.06) | 0.1 (0.05) | 0.4 (0.09)
  Work and School, Week 16 (n=28,44,38,68) | 0.3 (0.13) | 0.3 (0.08) | 0.0 (0.03) | 0.4 (0.10)
  Treatment, Baseline (n=31,82,45,133) | 0.3 (0.10) | 0.1 (0.04) | 0.2 (0.05) | 0.1 (0.03)
  Treatment, Week 4 (n=30,82,43,127) | 0.3 (0.10) | 0.4 (0.07) | 0.2 (0.06) | 0.5 (0.08)
  Treatment, Week 8 (n=30,68,43,104) | 0.3 (0.10) | 0.5 (0.09) | 0.1 (0.05) | 0.6 (0.09)
  Treatment, Week 12 (n=28,52,41,83) | 0.4 (0.14) | 0.4 (0.09) | 0.2 (0.09) | 0.5 (0.08)
  Treatment, Week 16 (n=28,44,38,68) | 0.3 (0.12) | 0.6 (0.11) | 0.2 (0.07) | 0.6 (0.11)

86. Secondary Outcome: Mean DLQI Subscale Scores During the CP-690,550 Re-Treatment (Period C)
Description: as for outcome 84
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
score on a scale
  Daily Activities, Baseline (n=27,75,42,120) | 0.7 (0.23) | 1.5 (0.19) | 0.4 (0.12) | 1.8 (0.17)
  Daily Activities, Week 4 (n=27,74,42,119) | 0.6 (0.24) | 0.9 (0.14) | 0.5 (0.14) | 0.8 (0.11)
  Daily Activities, Week 8 (n=26,71,41,118) | 0.9 (0.33) | 0.7 (0.12) | 0.4 (0.14) | 0.5 (0.09)
  Daily Activities, Week 16 (n=22,65,39,101) | 0.7 (0.27) | 0.8 (0.14) | 0.4 (0.15) | 0.5 (0.10)
  Personal Relationships, Baseline (n=27,75,42,120) | 0.4 (0.23) | 0.9 (0.16) | 0.1 (0.06) | 1.2 (0.15)
  Personal Relationships, Week 4 (n=27,74,42,119) | 0.4 (0.24) | 0.5 (0.10) | 0.2 (0.09) | 0.5 (0.10)
  Personal Relationships, Week 8 (n=26,71,41,118) | 0.4 (0.25) | 0.2 (0.07) | 0.3 (0.12) | 0.3 (0.09)
  Personal Relationships, Week 16 (n=22,66,39,101) | 0.2 (0.16) | 0.3 (0.09) | 0.1 (0.11) | 0.2 (0.06)
  Symptoms and Feelings, Baseline (n=27,75,42,120) | 1.4 (0.32) | 2.6 (0.19) | 1.1 (0.20) | 2.9 (0.18)
  Symptoms and Feelings, Week 4 (n=27,74,42,119) | 1.4 (0.27) | 1.6 (0.15) | 1.0 (0.20) | 1.4 (0.11)
  Symptoms and Feelings, Week 8 (n=26,71,41,118) | 1.5 (0.36) | 1.5 (0.14) | 1.0 (0.18) | 1.0 (0.12)
  Symptoms and Feelings, Week 16 (n=22,66,39,101) | 1.2 (0.27) | 1.5 (0.15) | 0.9 (0.22) | 1.0 (0.12)
  Leisure, Baseline (n=27,75,42,120) | 0.5 (0.18) | 0.9 (0.18) | 0.1 (0.06) | 1.4 (0.16)
  Leisure, Week 4 (n=27,74,41,119) | 0.4 (0.17) | 0.6 (0.13) | 0.2 (0.09) | 0.6 (0.10)
  Leisure, Week 8 (n=26,71,41,118) | 0.5 (0.22) | 0.4 (0.08) | 0.3 (0.10) | 0.4 (0.09)
  Leisure, Week 16 (n=22,66,39,101) | 0.4 (0.24) | 0.4 (0.10) | 0.3 (0.13) | 0.4 (0.09)
  Work and School, Baseline (n=27,75,42,120) | 0.3 (0.14) | 0.5 (0.09) | 0.1 (0.04) | 0.6 (0.09)
  Work and School, Week 4 (n=27,74,42,119) | 0.2 (0.12) | 0.2 (0.08) | 0.1 (0.04) | 0.2 (0.05)
  Work and School, Week 8 (n=26,71,41,118) | 0.2 (0.14) | 0.1 (0.04) | 0.0 (0.03) | 0.2 (0.05)
  Work and School, Week 16 (n =22,66,39,101) | 0.2 (0.14) | 0.2 (0.05) | 0.2 (0.09) | 0.1 (0.05)
  Treatment, Baseline (n=27,75,42,120) | 0.3 (0.13) | 0.7 (0.10) | 0.3 (0.09) | 0.9 (0.09)
  Treatment, Week 4 (n=27,74,42,119) | 0.3 (0.10) | 0.4 (0.08) | 0.2 (0.09) | 0.4 (0.05)
  Treatment, Week 8 (n=26,71,41,118) | 0.3 (0.14) | 0.3 (0.06) | 0.1 (0.05) | 0.3 (0.05)
  Treatment, Week 16 (n=22,66,39,101) | 0.2 (0.09) | 0.2 (0.06) | 0.2 (0.08) | 0.3 (0.05)

87. Secondary Outcome: Mean Change From Baseline-A in DLQI Subscale Scores During the Initial CP-690,550 Treatment (Period A)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much); higher scores indicate poor quality of life. The DLQI can be analyzed under 6 subscales by combining questions and is categorized as follows: symptoms and feelings (maximum score=6); daily activities (maximum score=6); leisure (maximum score=6); work and school (maximum score=3); personal relationships (maximum score=6); and treatment (maximum score=3). The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline. Baseline-A defined as the last observation up to first dosing date in Period A.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 325 | 328
scores on a scale
  Daily Activities, Week 4 (n=325,328) | -1.2 (0.09) | -1.6 (0.09)
  Daily Activities, Week 8 (n=320,318) | -1.5 (0.10) | -1.9 (0.10)
  Daily Activities, Week 16 (n=309,301) | -1.7 (0.10) | -2.0 (0.10)
  Daily Activities, Week 24 (n=272,275) | -1.6 (0.11) | -2.0 (0.11)
  Personal Relationships, Week 4 (n=326,327) | -0.8 (0.08) | -1.0 (0.09)
  Personal Relationships, Week 8 (n=321,316) | -1.0 (0.08) | -1.3 (0.09)
  Personal Relationships, Week 16 (n=310,300) | -1.1 (0.09) | -1.3 (0.10)
  Personal Relationships, Week 24 (n=271,274) | -1.0 (0.10) | -1.3 (0.10)
  Symptoms and Feelings, Week 4 (n=326,328) | -1.9 (0.08) | -2.3 (0.08)
  Symptoms and Feelings, Week 8 (n=321,317) | -2.2 (0.09) | -2.7 (0.09)
  Symptoms and Feelings, Week 18 (n=310,301) | -2.2 (0.09) | -2.8 (0.10)
  Symptoms and Feelings, Week 24 (n=273,275) | -2.1 (0.11) | -2.9 (0.10)
  Leisure, Week 4 (n=326,328) | -1.0 (0.10) | -1.4 (0.10)
  Leisure, Week 16 (n=310,301) | -1.4 (0.11) | -1.7 (0.11)
  Leisure, Week 8 (n=321,318) | -1.2 (0.10) | -1.7 (0.10)
  Leisure, Week 24 (n=272,275) | -1.3 (0.12) | -1.8 (0.12)
  Work and School, Week 4 (n=325,328) | -0.4 (0.05) | -0.6 (0.06)
  Work and School, Week 8 (n=320,317) | -0.6 (0.05) | -0.7 (0.06)
  Work and School, Week 16 (n=308,301) | -0.6 (0.06) | -0.7 (0.06)
  Work and School, Week 24 (n=272,275) | -0.5 (0.06) | -0.7 (0.06)
  Treatment, Week 4 (n=326,327) | -0.5 (0.06) | -0.7 (0.05)
  Treatment, Week 8 (n=321,317) | -0.6 (0.06) | -0.8 (0.06)
  Treatment, Week 16 (n=310,300) | -0.6 (0.06) | -0.9 (0.06)
  Treatment, Week 24 (n=272,274) | -0.5 (0.06) | -1.0 (0.06)

88. Secondary Outcome: Mean Change From Baseline-B in DLQI Subscale Scores During the Double-Blind Treatment Withdrawal (Period B)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much); higher scores indicate poor quality of life. The DLQI can be analyzed under 6 subscales by combining questions and is categorized as follows: symptoms and feelings (maximum score=6); daily activities (maximum score=6); leisure (maximum score=6); work and school (maximum score=3); personal relationships (maximum score=6); and treatment (maximum score=3). The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline. Baseline-B defined as the last observation up to first dosing date in Period B.
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 30 | 82 | 43 | 127
scores on a scale
  Daily Activities, Week 4 (n=30,82,43,127) | 0.3 (0.22) | 0.5 (0.14) | 0.1 (0.08) | 0.9 (0.13)
  Daily Activities, Week 8 (n=30,68,43,104) | 0.1 (0.09) | 0.8 (0.17) | 0.2 (0.13) | 1.0 (0.17)
  Daily Activities, Week 12 (n=28,52,41,83) | 0.2 (0.13) | 0.7 (0.14) | 0.1 (0.11) | 0.9 (0.17)
  Daily Activities, Week 16 (n=28,44,38,68) | 0.2 (0.12) | 0.9 (0.19) | 0.2 (0.10) | 1.1 (0.22)
  Personal Relationships, Week 4 (n=30,82,43,126) | 0.0 (0.11) | 0.4 (0.10) | -0.1 (0.08) | 0.5 (0.09)
  Personal Relationships, Week 8 (n=30,68,43,103) | 0.1 (0.15) | 0.6 (0.15) | -0.1 (0.09) | 0.8 (0.13)
  Personal Relationships, Week 12 (n=28,52,41,83) | 0.1 (0.14) | 0.4 (0.14) | -0.1 (0.09) | 0.6 (0.13)
  Personal Relationships, Week 16 (n=28,44,38,68) | 0.1 (0.15) | 0.3 (0.15) | -0.1 (0.10) | 0.8 (0.17)
  Symptoms and Feelings, Week 4 (n=30,82,43,127) | 0.2 (0.25) | 1.3 (0.17) | 0.1 (0.13) | 1.7 (0.14)
  Symptoms and Feelings, Week 8 (n=30,68,43,104) | 0.0 (0.13) | 1.5 (0.17) | 0.2 (0.17) | 1.8 (0.16)
  Symptoms and Feelings, Week 12 (n=28,52,41,83) | 0.1 (0.19) | 1.4 (0.18) | 0.5 (0.19) | 1.6 (0.18)
  Symptoms and Feelings, Week 16 (n=28,44,38,68) | 0.4 (0.21) | 1.3 (0.22) | 0.5 (0.14) | 1.8 (0.21)
  Leisure, Week 4 (n=30,82,42,127) | 0.2 (0.22) | 0.3 (0.11) | -0.1 (0.09) | 0.7 (0.12)
  Leisure, Week 8 (n=30,68,43,104) | 0.1 (0.10) | 0.5 (0.16) | 0.0 (0.10) | 0.8 (0.15)
  Leisure, Week 12 (n=28,52,41,83) | 0.2 (0.12) | 0.4 (0.11) | 0.0 (0.09) | 0.6 (0.15)
  Leisure, Week 16 (n=28,44,37,68) | 0.2 (0.12) | 0.4 (0.12) | -0.1 (0.08) | 0.8 (0.18)
  Work and School, Week 4 (n=30,82,43,127) | 0.0 (0.6) | 0.2 (0.07) | 0.0 (0.00) | 0.5 (0.08)
  Work and School, Week 8 (n=30,68,43,104) | 0.1 (0.06) | 0.2 (0.09) | 0.0 (0.02) | 0.4 (0.08)
  Work and School, Week 12 (n=28,52,41,83) | 0.1 (0.08) | 0.1 (0.07) | 0.1 (0.04) | 0.3 (0.09)
  Work and School, Week 16 (n=28,44,38,68) | 0.2 (0.10) | 0.2 (0.09) | 0.0 (0.00) | 0.4 (0.10)
  Treatment, Week 4 (n=30,82,43,127) | 0.0 (0.07) | 0.2 (0.06) | 0.1 (0.06) | 0.4 (0.07)
  Treatment, Week 8 (n=30,68,43,104) | 0.0 (0.06) | 0.4 (0.09) | 0.0 (0.06) | 0.6 (0.08)
  Treatment, Week 12 (n=28,52,41,83) | 0.1 (0.11) | 0.3 (0.7) | 0.0 (0.09) | 0.4 (0.09)
  Treatment, Week 16 (n=28,44,38,68) | 0.0 (0.10) | 0.5 (0.11) | 0.1 (0.05) | 0.5 (0.10)

89. Secondary Outcome: Mean Change From Baseline-C in DLQI Subscale Scores During the CP-690,550 Re-Treatment (Period C)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much); higher scores indicate poor quality of life. The DLQI can be analyzed under 6 subscales by combining questions and is categorized as follows: symptoms and feelings (maximum score=6); daily activities (maximum score=6); leisure (maximum score=6); work and school (maximum score=3); personal relationships (maximum score=6); and treatment (maximum score=3). The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline. Baseline-C defined as the last observation up to first dosing date in Period C.
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 74 | 42 | 119
scores on a scale
  Daily Activities, Week 4 (n=27,74,42,119) | 0.0 (0.06) | -0.7 (0.12) | 0.1 (0.11) | -1.0 (0.13)
  Daily Activities, Week 8 (n=26,71,41,118) | 0.2 (0.15) | -0.7 (0.13) | 0.0 (0.14) | -1.3 (0.15)
  Daily Activities, Week 16 (n=22,65,39,101) | 0.4 (0.23) | -0.7 (0.20) | -0.1 (0.18) | -1.3 (0.18)
  Personal Relationships, Week 4 (n=27,74,42,119) | 0.0 (0.05) | -0.4 (0.11) | 0.1 (0.08) | -0.7 (0.13)
  Personal Relationships, Week 8 (n=26,71,41,118) | 0.0 (0.07) | -0.6 (0.13) | 0.1 (0.13) | -0.8 (0.14)
  Personal Relationships, Week 16 (n=22,66,39,101) | 0.0 (0.11) | -0.6 (0.14) | 0.1 (0.12) | -0.9 (0.15)
  Symptoms and Feelings, Week 4 (n=27,74,42,119) | 0.0 (0.14) | -1.0 (0.13) | -0.1 (0.13) | -1.5 (0.15)
  Symptoms and Feelings, Week 8 (n=26,71,41,118) | 0.0 (0.14) | -1.1 (0.17) | -0.1 (0.18) | -1.8 (0.18)
  Symptoms and Feelings, Week 16 (n=22,66,39,101) | 0.0 (0.20) | -1.0 (0.20) | -0.2 (0.21) | -1.9 (0.19)
  Leisure, Week 4 (n=27,74,41,119) | -0.1 (0.08) | -0.3 (0.14) | 0.1 (0.06) | -0.8 (0.13)
  Leisure, Week 8 (n=26,71,41,118) | 0.0 (0.13) | -0.4 (0.13) | 0.1 (0.10) | -1.0 (0.15)
  Leisure, Week 16 (n=22,66,39,101) | 0.0 (0.28) | -0.4 (0.17) | 0.2 (0.12) | -1.1 (0.18)
  Work and School, Week 4 (n=27,74,42,119) | 0.0 (0.06) | -0.2 (0.07) | 0.0 (0.03) | -0.4 (0.08)
  Work and School, Week 8 (n=26,71,41,118) | 0.0 (0.7) | -0.3 (0.09) | 0.0 (0.06) | -0.4 (0.09)
  Work and School, Week 16 (n=22,66,39,101) | 0.0 (0.07) | -0.3 (0.10) | 0.1 (0.09) | -0.5 (0.09)
  Treatment, Week 4 (n=27,74,42,119) | 0.0 (0.08) | -0.2 (0.08) | 0.0 (0.07) | -0.6 (0.07)
  Treatment, Week 8 (n=26,71,41,118) | 0.0 (0.07) | -0.3 (0.08) | -0.2 (0.09) | -0.07 (0.09)
  Treatment, Week 16 (n=22,66,39,101) | 0.0 (0.08) | -0.3 (0.09) | -0.1 (0.11) | -0.7 (0.10)

90. Secondary Outcome: Percentage of Participants Achieving DLQI ≥5 Point Reduction From Baseline-A Response During Initial CP-690,550 Treatment (Period A)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life. The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A participants with a Baseline-A DLQI ≥5, where Baseline-A is defined as the last observation up to first dosing date in Period A. n=participants with an observation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 284 | 281
percentage of participants
  Week 4 | 59.86 [54.16 to 65.56] | 75.44 [70.41 to 80.48]
  Week 8 | 70.42 [65.11 to 75.73] | 80.78 [76.18 to 85.39]
  Week 16 | 70.77 [65.49 to 76.06] | 79.00 [74.24 to 83.77]
  Week 24 | 59.86 [54.16 to 65.56] | 72.95 [67.76 to 78.15]

91. Secondary Outcome: Percentage of Participants Achieving DLQI ≥5 Point Reduction From Baseline-B Response During Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 90
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B participants with Baseline-B DLQI ≥5.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 9 | 12 | 3 | 9
percentage of participants
  Week 4 | 0.00 | 16.67 | 33.33 | 0.00
  Week 8 | 0.00 | 0.00 | 0.00 | 11.11
  Week 12 | 11.11 | 0.00 | 66.67 | 11.11
  Week 16 | 0.00 | 8.33 | 33.33 | 11.11

92. Secondary Outcome: Percentage of Participants Achieving DLQI ≥5 Point Reduction From Baseline-C Response During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 83
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C participants with Baseline-C DLQI ≥5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 8 | 40 | 8 | 76
percentage of participants
  Week 4 | 0.00 [0.00 to 0.00] | 47.50 [32.02 to 62.98] | 0.00 [0.00 to 0.00] | 65.79 [55.12 to 76.46]
  Week 8 | 12.50 [0.00 to 35.42] | 55.00 [39.58 to 70.42] | 25.00 [0.00 to 55.01] | 77.63 [68.26 to 87.00]
  Week 16 | 12.50 [0.00 to 35.42] | 47.50 [32.02 to 62.98] | 12.50 [0.00 to 35.42] | 64.47 [53.71 to 75.23]

93. Secondary Outcome: Percentage of Participants Achieving DLQI ≤1 Response During the Initial CP-690,550 Treatment (Period A)
Description: as for outcome 90
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A participants with a Baseline-A DLQI ≤1, where Baseline-A is defined as the last observation up to first dosing date in Period A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 320 | 320
percentage of participants
  Week 4 | 13.44 [9.70 to 17.17] | 26.88 [22.02 to 31.73]
  Week 8 | 25.94 [21.14 to 30.74] | 41.88 [36.47 to 47.28]
  Week 16 | 30.94 [25.87 to 36.00] | 53.13 [47.66 to 58.59]
  Week 24 | 30.63 [25.57 to 35.68] | 50.00 [44.52 to 55.48]

94. Secondary Outcome: Percentage of Participants Achieving DLQI ≤1 Response During Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 90
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B participants with Baseline-B DLQI >1 where Baseline-B defined as last observation up to first dosing date in Period B.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 13 | 25 | 12 | 31
percentage of participants
  Baseline | 0.00 | 0.00 | 0.00 | 0.00
  Week 4 | 7.69 | 4.00 | 41.67 | 12.90
  Week 8 | 7.69 | 0.00 | 33.33 | 9.68
  Week 12 | 7.69 | 0.00 | 8.33 | 9.68
  Week 16 | 7.69 | 0.00 | 16.67 | 9.68

95. Secondary Outcome: Percentage of Participants Achieving DLQI ≤1 Response During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 90
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C participants with a Baseline-C DLQI >1, where Baseline-C is defined as the last observation up to first dosing date in Period C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 12 | 61 | 16 | 93
percentage of participants
  Baseline | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 4 | 16.67 [0.00 to 37.75] | 24.59 [13.78 to 35.40] | 37.50 [13.78 to 61.22] | 24.73 [15.96 to 33.50]
  Week 8 | 16.67 [0.00 to 37.75] | 26.23 [15.19 to 37.27] | 31.25 [8.54 to 53.96] | 40.86 [30.87 to 50.85]
  Week 16 | 16.67 [0.00 to 37.75] | 29.51 [18.06 to 40.95] | 37.50 [13.78 to 61.22] | 40.86 [30.87 to 50.85]

96. Secondary Outcome: Percentage of Participants by DLQI Severity Category During the Initial CP-690,550 Treatment (Period A)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). Severity is measured using the following categories of scores: 0-1=no effect on patients' lives; 2-5=small effect; 6-10=moderate effect; 11-20=very large effect; 21-30=extremely large effect.
Time Frame: Baseline and Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 330 | 333
percentage of participants
  Baseline, No effect (0-1) (n=330,333) | 3.0 (3.0) | 3.9 (3.9)
  Baseline, Small effect (2-5;n=330,333) | 15.2 (15.2) | 17.1 (17.1)
  Baseline, Moderate effect (6-10;n=330,333) | 27.0 (27.0) | 21.3 (21.3)
  Baseline, Very large effect (11-20;n=330,333) | 39.1 (39.1) | 41.7 (41.7)
  Baseline, Extremely large effect (21-30;n=330,333) | 15.8 (15.8) | 15.9 (15.9)
  Week 4, No effect (0-1) (n=326,330) | 15.6 (15.6) | 29.4 (29.4)
  Week 4, Small effect (2-5;n=326,330) | 35.9 (35.9) | 37.3 (37.3)
  Week 4, Moderate effect (6-10;n=326,330) | 25.8 (25.8) | 22.1 (22.1)
  Week 4, Very large effect (11-20;n=326,330) | 18.7 (18.7) | 9.7 (9.7)
  Week 4, Extremely large effect (21-30;n=326,330) | 4.0 (4.0) | 1.5 (1.5)
  Week 8, No effect (0-1) (n=321,319) | 28.0 (28.0) | 45.5 (45.5)
  Week 8, Small effect (2-5;n=321,319) | 34.0 (34.0) | 34.8 (34.8)
  Week 8, Moderate effect (6-10;n=321,319) | 23.7 (23.7) | 12.5 (12.5)
  Week 8, Very large effect (11-20;n=321,319) | 11.8 (11.8) | 5.0 (5.0)
  Week 8, Extremely large effect (21-30;n=321,319) | 2.5 (2.5) | 2.2 (2.2)
  Week 16, No effect (0-1) (n=310,303) | 34.2 (34.2) | 59.4 (59.4)
  Week 16, Small effect (2-5;n=310,303) | 34.5 (34.5) | 22.1 (22.1)
  Week 16, Moderate effect (6-10;n=310,303) | 18.4 (18.4) | 10.6 (10.6)
  Week 16, Very large effect (11-20;n=310,303) | 11.0 (11.0) | 6.3 (6.3)
  Week 16, Extremely large effect (21-30;n=310,303) | 1.9 (1.9) | 1.7 (1.7)
  Week 24, No effect (0-1) (n=273,277) | 38.1 (38.1) | 61.0 (61.0)
  Week 24, Small effect (2-5;n=273,277) | 27.1 (27.1) | 24.9 (24.9)
  Week 24, Moderate effect (6-10;n=273,277) | 19.0 (19.0) | 9.0 (9.0)
  Week 24, Very large effect (11-20;n=273,277) | 12.8 (12.8) | 3.2 (.32)
  Week 24, Extremely large effect (21-30;n=273,277) | 2.9 (2.9) | 1.8 (1.8)

97. Secondary Outcome: Percentage of Participants With DLQI ≥5-Point Reduction From Baseline-A Response During Initial CP-690,550 Treatment (Period A)
Description: as for outcome 90
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A participants with Baseline-A DLQI ≥5, where Baseline-A was defined as the last observation before the first dosing date in Period A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 283 | 279
percentage of participants
  Week 4 | 60.1 [54.5 to 65.9] | 76.6 [71.5 to 81.4]
  Week 8 | 77.4 [72.4 to 82.2] | 88.7 [84.6 to 92.2]
  Week 16 | 85.7 [81.3 to 89.6] | 94.9 [91.6 to 97.2]
  Week 24 | 91.9 [83.2 to 97.1] | 96.1 [92.9 to 98.1]

98. Secondary Outcome: Median Time to DLQI ≥5-Point Reduction From Baseline-A Response During Initial CP-690,550 Treatment (Period A)
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: as for outcome 97
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 283 | 279
weeks | 4.4 [4.3 to 4.7] | 4.1 [4.1 to 4.3]

99. Secondary Outcome: Percentage of Participants With DLQI ≥5-Point Reduction From Baseline-A Response During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 90
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: FAS-C participants with Baseline-C DLQI ≥5, where Baseline-C defined as the last observation up to first dosing date in Period C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 8 | 40 | 8 | 76
percentage of participants
  Week 4 | 0.0 [0.0 to 0.0] | 47.5 [33.5 to 63.9] | 0.0 [0.0 to 0.0] | 65.8 [55.2 to 76.2]
  Week 8 | 12.5 [1.9 to 61.3] | 72.5 [58.3 to 85.1] | 25.0 [6.9 to 68.5] | 80.9 [71.3 to 88.9]
  Week 16 | 12.5 [1.9 to 61.3] | 81.3 [67.3 to 91.9] | 25.0 [6.9 to 68.5] | 88.4 [79.1 to 94.8]

100. Secondary Outcome: Median Time to DLQI ≥5-Point Reduction From Baseline-A Response During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 98
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: as for outcome 99
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 8 | 40 | 8 | 76
weeks | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 8.1 [4.7 to 8.6] | NA [NA to NA] — Median and 95% confidence interval cannot be estimated due to <50% of events occurring and/or censoring issue. | 4.4 [4.3 to 5.7]

101. Secondary Outcome: Mean Short-Form 36 (SF-36) Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores During the Initial CP-690,550 Treatment (Period A)
Description: The SF-36 is a general health status questionnaire that assesses 8 domains of functional health and well being: Physical Functioning, Role Limitations due to Physical Health Problems, Bodily Pain, Social Functioning, Mental Health, Role Limitations due to Emotional Problems, Vitality, and General Health Perceptions. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). A PCS score and MCS score are based on a normalized sum of the 8 scale scores; PCS/MCS summary concept score = (raw score*10) plus 50. Linear transformations were performed to transform scores to a mean of 50 and standard deviations (SDs) of 10, in the general population. In norm-based scoring, each scale is scored to have same average (50)/SD (10). With this method anytime a scale score is below 50, health status is below average, and each point is one-tenth of a SD. Higher scores indicate a better health related quality of life.
Time Frame: Baseline and Week 24 (Period A)
Population: FAS-A; n=number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 330 | 334
score on a scale
  Baseline Physical Health Score (n=330,334) | 48.1 (0.5) | 47.8 (0.5)
  Week 24 Physical Health Score (n=273,276) | 50.5 (0.5) | 52.9 (0.5)
  Baseline Mental Health Score (n=330,334) | 45.2 (0.7) | 46.1 (0.6)
  Week 24 Mental Health Score (n=273,276) | 48.9 (0.6) | 51.2 (0.6)

102. Secondary Outcome: Mean SF-36 PCS and MCS Scores During CP-690,550 Re-Treatment (Period C)
Description: The SF-36 is a general health status questionnaire that assesses 8 domains of functional health and well being: Physical Functioning, Role Limitations due to Physical Health Problems, Bodily Pain, Social Functioning, Mental Health, Role Limitations due to Emotional Problems, Vitality, and General Health Perceptions. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). A PCS score and MCS score are based on a normalized sum of the 8 scale scores; PCS/MCS summary concept score = (raw score*10) plus 50. Linear transformations were performed to transform scores to a mean of 50 and SDs of 10, in the general population. In norm-based scoring, each scale is scored to have same average (50)/SD (10). With this method anytime a scale score is below 50, health status is below average, and each point is one-tenth of a SD. Higher scores indicate a better health related quality of life.
Time Frame: Baseline and Week 56 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
score on a scale
  Baseline Physical Health Score (n=27,75,42,120) | 51.8 (1.8) | 49.9 (1.1) | 53.8 (1.1) | 49.7 (0.8)
  Week 56 Physical Health Score (n=22,65,34,98) | 52.9 (1.8) | 52.7 (1.0) | 52.9 (1.4) | 51.2 (0.9)
  Baseline Mental Health Score (n=27,75,42,120) | 51.7 (1.9) | 51.0 (1.1) | 50.8 (1.9) | 48.3 (1.0)
  Week 56 Mental Health Score (n=22,65,34,98) | 50.8 (1.8) | 50.9 (1.2) | 52.4 (1.5) | 53.7 (0.8)

103. Secondary Outcome: Mean Change From Baseline-A in SF-36 PCS and MCS Scores During the Initial CP-690,550 Treatment (Period A)
Description: as for outcome 102
Time Frame: Week 24 (Period A)
Population: FAS-A
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 273 | 275
scores on a scale
  Physical Health Score | 1.9 (0.5) | 5.2 (0.5)
  Mental Health Score | 3.2 (0.6) | 4.9 (0.6)

104. Secondary Outcome: Mean Change From Baseline-C in SF-36 PCS and MCS Scores During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 102
Time Frame: Week 56 (Period C)
Population: FAS-C
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 22 | 65 | 34 | 98
scores on a scale
  Physical Health Score | -0.9 (1.2) | 2.7 (0.8) | -1.0 (0.8) | 1.8 (0.9)
  Mental Health Score | -1.6 (1.2) | 0.1 (1.0) | 0.5 (1.9) | 4.9 (1.0)

105. Secondary Outcome: Mean SF-36 Domain Scores During the Initial CP-690,550 Treatment (Period A)
Description: The SF-36 is a general health status questionnaire that assesses 8 domains of functional health and well being: Physical Functioning, Role Limitations due to Physical Health Problems, Bodily Pain, Social Functioning, Mental Health, Role Limitations due to Emotional Problems, Vitality, and General Health Perceptions. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Higher scores indicate a better health related quality of life.
Time Frame: Baseline and Week 24 (Period A)
Population: FAS-A; n=number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
score on a scale
  Baseline Physical Functioning (n=331,335) | 48.3 (0.6) | 48.0 (0.6)
  Week 24 Physical Functioning (n=273,276) | 50.7 (0.6) | 52.7 (0.5)
  Baseline Role Physical (n=331,335) | 47.2 (0.6) | 47.6 (0.6)
  Week 24 Role Physical (n=273,276) | 50.2 (0.6) | 53.1 (0.5)
  Baseline Bodily Pain (n=331,334) | 44.7 (0.6) | 44.2 (0.7)
  Week 24 Bodily Pain (n=273,276) | 50.0 (0.6) | 53.2 (0.5)
  Baseline General Health (n=330,335) | 48.1 (0.5) | 48.9 (0.5)
  Week 24 General Health (n=273,276) | 49.0 (0.6) | 50.3 (0.5)
  Baseline Vitality (n=331,334) | 49.2 (0.6) | 49.3 (0.5)
  Week 24 Vitality (n=273,276) | 51.0 (0.6) | 54.2 (0.5)
  Baseline Social Functioning (n=331,334) | 44.6 (0.7) | 44.6 (0.7)
  Week 24 Social Functioning (n=273,276) | 48.9 (0.6) | 51.7 (0.5)
  Baseline Role Emotional (n=331,335) | 45.5 (0.7) | 45.8 (0.7)
  Week 24 Role Emotional (n=273,276) | 49.2 (0.6) | 51.2 (0.5)
  Baseline Mental Health (n=331,334) | 45.0 (0.6) | 46.4 (0.6)
  Week 24 Mental Health (n=273,276) | 48.8 (0.6) | 51.0 (0.6)
  Baseline Health Transition Score (n=331,334) | 3.0 (0.0) | 3.1 (0.0)
  Week 24 Health Transition Score (n=272, 276) | 2.8 (0.0) | 2.8 (0.0)

106. Secondary Outcome: Mean SF-36 Domain Scores During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 105
Time Frame: Baseline and Week 56 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
score on a scale
  Baseline Physical Functioning (n=27,75,42,120) | 50.7 (1.8) | 51.3 (1.0) | 52.7 (1.3) | 51.1 (0.8)
  Week 56 Physical Functioning (n=22,65,34,98) | 51.7 (1.9) | 52.4 (1.1) | 52.3 (1.6) | 51.3 (0.9)
  Baseline Role Physical (n=27,75,42,120) | 51.2 (1.6) | 50.5 (1.0) | 53.3 (1.1) | 49.1 (0.9)
  Week 56 Role Physical (n=22,65,34,98) | 52.5 (1.6) | 51.4 (1.2) | 54.2 (1.1) | 51.9 (0.8)
  Baseline Bodily Pain (n=27,75,42,120) | 52.8 (1.9) | 48.8 (1.2) | 54.1 (1.5) | 47.1 (1.1)
  Week 56 Bodily Pain (n=22,65,34,98) | 53.9 (2.1) | 52.7 (1.0) | 53.5 (1.8) | 52.7 (0.9)
  Baseline General Health (n=27,75,42,120) | 52.0 (1.7) | 49.6 (1.1) | 51.9 (1.4) | 48.7 (0.9)
  Week 56 General Health (n=22,65,34,98) | 51.5 (1.8) | 51.8 (1.0) | 51.1 (1.4) | 50.7 (0.8)
  Baseline Vitality (n=27,75,42,120) | 53.8 (2.2) | 52.2 (1.1) | 54.1 (1.5) | 51.3 (0.9)
  Week 56 Vitality (n=22,65,34,98) | 52.2 (2.2) | 53.2 (1.1) | 54.8 (1.7) | 54.3 (0.9)
  Baseline Social Functioning (n=27,75,42,120) | 51.2 (1.8) | 49.7 (1.0) | 51.5 (1.4) | 48.1 (1.0)
  Week 56 Social Functioning (n=22,65,34,98) | 52.2 (1.6) | 52.4 (1.0) | 51.3 (1.7) | 53.2 (0.6)
  Baseline Role Emotional (n=27,75,42,120) | 51.1 (1.8) | 51.6 (0.8) | 50.3 (1.7) | 48.0 (1.0)
  Week 56 Role Emotional (n=22,65,34,98) | 50.5 (1.8) | 50.0 (1.3) | 52.9 (1.1) | 53.0 (0.6)
  Baseline Mental Health (n=27,75,42,120) | 51.2 (2.0) | 50.2 (1.1) | 51.6 (1.8) | 48.4 (1.0)
  Week 56 Mental Health (n=22,65,34,98) | 51.1 (1.8) | 51.1 (1.2) | 52.2 (1.5) | 52.7 (0.8)
  Baseline Health Transition (n=27,75,42,120) | 2.9 (0.1) | 3.1 (0.1) | 2.8 (0.1) | 3.0 (0.1)
  Week 56 Health Transition (n=22,65,34,98) | 3.0 (0.1) | 2.7 (0.1) | 2.8 (0.1) | 2.8 (0.1)

107. Secondary Outcome: Mean Change From Baseline-A in SF-36 Domain Scores During the Initial CP-690,550 Treatment (Period A)
Description: The SF-36 is a general health status questionnaire that assesses 8 domains of functional health and well being: Physical Functioning, Role Limitations due to Physical Health Problems, Bodily Pain, Social Functioning, Mental Health, Role Limitations due to Emotional Problems, Vitality, and General Health Perceptions. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Higher scores indicate a better health related quality of life. Baseline-A defined as the last observation up to first dosing date in Period A.
Time Frame: Week 24 (Period A)
Population: FAS-A; n=number of participants with an observation
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 273 | 276
scores on a scale
  Physical Functioning (n=273,276) | 1.8 (0.5) | 4.6 (0.5)
  Role Physical (n=273,276) | 2.6 (0.7) | 5.6 (0.6)
  Bodily Pain (n=273,275) | 4.5 (0.7) | 9.0 (0.7)
  General Health (n=273,276) | 0.7 (0.5) | 1.7 (0.4)
  Vitality (n=273,275) | 1.3 (0.5) | 4.8 (0.5)
  Social Functioning (n=273,275) | 3.7 (0.7) | 6.6 (0.7)
  Role Emotional (n=273,276) | 3.2 (0.8) | 5.6 (0.7)
  Mental Health (n=273,275) | 3.4 (0.6) | 4.4 (0.6)
  Health Transition (n=272,275) | -0.2 (0.1) | -0.2 (0.0)

108. Secondary Outcome: Mean Change From Baseline-C in SF-36 Domain Scores During CP-690,550 Re-Treatment (Period C)
Description: The SF-36 is a general health status questionnaire that assesses 8 domains of functional health and well being: Physical Functioning, Role Limitations due to Physical Health Problems, Bodily Pain, Social Functioning, Mental Health, Role Limitations due to Emotional Problems, Vitality, and General Health Perceptions. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Higher scores indicate a better health related quality of life. Baseline-C defined as the last observation up to first dosing date in Period C.
Time Frame: Week 56 (Period C)
Population: FAS-C
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 22 | 65 | 34 | 98
scores on a scale
  Physical Functioning | -0.4 (0.7) | 1.2 (0.7) | -0.5 (0.7) | 0.7 (0.9)
  Role Physical | -0.7 (0.9) | 1.2 (1.1) | 0.2 (0.8) | 2.7 (0.9)
  Bodily Pain | -1.6 (1.6) | 3.8 (1.1) | -1.1 (1.4) | 6.0 (1.2)
  General Health | -0.7 (0.9) | 1.9 (0.8) | -1.1 (0.9) | 1.6 (0.8)
  Vitality | -3.5 (1.3) | 1.1 (0.9) | 0.2 (1.6) | 3.1 (1.0)
  Social Functioning | -1.5 (0.7) | 2.6 (1.1) | -1.3 (1.9) | 4.7 (1.0)
  Role Emotional | -1.4 (1.0) | -1.3 (1.2) | 1.9 (1.6) | 4.6 (1.0)
  Mental Health | -0.1 (1.5) | 1.1 (0.9) | -0.5 (1.5) | 4.1 (1.0)
  Health Transition Score | -0.0 (0.1) | -0.3 (0.1) | 0.1 (0.1) | -0.2 (0.1)

109. Secondary Outcome: Percentage of Participants in Each Patient Global Assessment (PtGA) of Psoriasis Category During the Initial CP-690,550 Treatment (Period A)
Description: The PtGA asks the participant to evaluate the overall cutaneous disease at that point in time on a single item, 5 point scale. The scale is scored as follows: 0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe
Time Frame: Baseline and Weeks 4, 8, 16 and 24 (Period A)
Population: FAS-A
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 330 | 335
percentage of participants
  Baseline, Clear (n=330,335) | 0.0 | 0.0
  Baseline, Almost clear (n=330,335) | 0.0 | 0.3
  Baseline, Mild (n=330,335) | 3.6 | 1.2
  Baseline, Moderate (n=330,335) | 30.3 | 34.6
  Baseline Severe (n=330,335) | 66.1 | 63.9
  Week 4, Clear (n=325,331) | 0.3 | 1.2
  Week 4, Almost Clear (n=325,331) | 11.7 | 20.2
  Week 4, Mild (n=325,331) | 24.9 | 30.5
  Week 4, Moderate (n=325,331) | 40.6 | 37.8
  Week 4, Severe (n=325,331) | 22.5 | 10.3
  Week 8, Clear (n=320,321) | 1.9 | 5.9
  Week 8, Almost Clear (n=320,321) | 21.3 | 41.4
  Week 8, Mild (n=320,321) | 31.9 | 25.2
  Week 8, Moderate (n=320,321) | 30.0 | 22.4
  Week 8, Severe (n=320,321) | 15.0 | 5.0
  Week 16, Clear (n=310,303) | 5.5 | 16.8
  Week 16, Almost Clear (n=310,303) | 27.1 | 43.6
  Week 16, Mild (n=310,303) | 30.6 | 20.8
  Week 16, Moderate (n=310,303) | 27.7 | 11.9
  Week 16, Severe (n=310,303) | 9.0 | 6.9
  Week 24, Clear (n=273,277) | 8.1 | 20.9
  Week 24, Almost Clear (n=273,277) | 27.8 | 41.5
  Week 24, Mild (n=273,277) | 23.8 | 20.2
  Week 24, Moderate (n=273,277) | 30.0 | 13.4
  Week 24, Severe (n=273,277) | 10.3 | 4.0

110. Secondary Outcome: Percentage of Participants in Each PtGA of Psoriasis Category During Double-Blind Treatment Withdrawal (Period B)
Description: as for outcome 109
Time Frame: Baseline and Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B; n equals the number of participants with observations
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
percentage of participants
  Baseline, Clear (n=31,82,45,133) | 16.1 | 19.5 | 24.4 | 35.3
  Baseline, Almost Clear (n=31,82,45,133) | 45.2 | 61.0 | 62.2 | 46.6
  Baseline, Mild (n=31,82,45,133) | 25.8 | 12.2 | 11.1 | 15.0
  Baseline, Moderate (n=31,82,45,133) | 12.9 | 7.3 | 2.2 | 3.0
  Baseline, Severe (n=31,82,45,133) | 0.0 | 0.0 | 0.0 | 0.0
  Week 4, Clear (n=30,82,43,126) | 23.3 | 8.5 | 23.3 | 11.1
  Week 4, Almost Clear (n=30,82,43,126) | 43.3 | 34.1 | 58.1 | 33.3
  Week 4, Mild (n=30,82,43,126) | 23.3 | 30.5 | 11.6 | 17.5
  Week 4, Moderate (n=30,82,43,126) | 6.7 | 15.9 | 7.0 | 27.0
  Week 4, Severe (n=30,82,43,126) | 3.3 | 11.0 | 0.0 | 11.1
  Week 8, Clear (n=30,68,43,104) | 23.3 | 7.4 | 20.9 | 5.8
  Week 8, Almost Clear (n=30,68,43,104) | 30.0 | 27.9 | 48.8 | 29.8
  Week 8, Mild (n=30,68,43,104) | 36.7 | 23.5 | 23.3 | 26.0
  Week 8, Moderate (n=30,68,43,104) | 10.0 | 26.5 | 7.0 | 23.1
  Week 8, Severe (n=30,68,43,104) | 0.0 | 14.7 | 0.0 | 15.4
  Week 12, Clear (n=28,52,41,83) | 17.9 | 1.9 | 14.6 | 4.8
  Week 12, Almost Clear (n=28,52,41,83) | 35.7 | 19.2 | 58.5 | 32.5
  Week 12, Mild (n=28,52,41,83) | 32.1 | 36.5 | 22.0 | 24.1
  Week 12, Moderate (n=28,52,41,83) | 10.7 | 28.8 | 4.9 | 24.1
  Week 12, Severe (n=28,52,41,83) | 3.6 | 13.5 | 0.0 | 14.5
  Week 16, Clear (n=27,45,38,68) | 22.2 | 4.4 | 18.4 | 7.4
  Week 16, Almost Clear (n=27,45,38,68) | 33.3 | 28.9 | 52.6 | 25.0
  Week 16, Mild (n=27,45,38,68) | 18.5 | 22.2 | 21.1 | 25.0
  Week 16, Moderate (n=27,45,38,68) | 25.9 | 33.3 | 7.9 | 30.9
  Week 16, Severe (n=27,45,38,68) | 0.0 | 11.1 | 0.0 | 11.8

111. Secondary Outcome: Percentage of Participants in Each PtGA of Psoriasis Category During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 109
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
percentage of participants
  Baseline, Clear (n=27,75,42,120) | 22.2 | 2.7 | 19.0 | 5.0
  Baseline, Almost Clear (n=27,75,42,120) | 33.3 | 18.7 | 50.0 | 18.3
  Baseline, Mild (n=27,75,42,120) | 18.5 | 18.7 | 16.7 | 17.5
  Baseline, Moderate (n=27,75,42,120) | 25.9 | 37.3 | 14.3 | 33.3
  Baseline, Severe (n=27,75,42,120) | 0.0 | 22.7 | 0.0 | 25.8
  Week 4, Clear (n=27,74,42,118) | 18.5 | 5.4 | 19.0 | 10.2
  Week 4, Almost Clear (n=27,74,42,118) | 37.0 | 23.0 | 50.0 | 41.5
  Week 4, Mild (n=27,74,42,118) | 33.3 | 41.9 | 11.9 | 23.7
  Week 4, Moderate (n=27,74,42,118) | 11.1 | 25.7 | 14.3 | 20.3
  Week 4, Severe (n=27,74,42,118) | 0.0 | 4.1 | 4.8 | 4.2
  Week 8, Clear (n=26,71,41,118) | 19.2 | 7.0 | 19.5 | 15.3
  Week 8, Almost Clear (n=26,71,41,118) | 26.9 | 36.6 | 51.2 | 46.6
  Week 8, Mild (n=26,71,41,118) | 30.8 | 38.0 | 19.5 | 24.6
  Week 8, Moderate (n=26,71,41,118) | 19.2 | 16.9 | 7.3 | 9.3
  Week 8, Severe (n=26,71,41,118) | 3.8 | 1.4 | 2.4 | 4.2
  Week 16, Clear (n=22,65,38,101) | 13.6 | 10.8 | 18.4 | 20.8
  Week 16, Almost Clear (n=22,65,38,101) | 31.8 | 43.1 | 57.9 | 47.5
  Week 16, Mild (n=22,65,38,101) | 36.4 | 27.7 | 10.5 | 18.8
  Week 16, Moderate (n=22,65,38,101) | 13.6 | 13.8 | 5.3 | 10.9
  Week 16, Severe (n=22,65,38,101) | 4.5 | 4.6 | 7.9 | 2.0

112. Secondary Outcome: Percentage of Participants With PtGA Response of Clear or Almost Clear During the Initial CP-690,550 Treatment (Period A)
Description: The PtGA asks the participant to evaluate the overall cutaneous disease at that point in time on a single item, 5 point scale. The scale is scored as follows: 0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe. Response defined as score of 0 or 1.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
percentage of participants
  Week 4 | 11.78 [8.31 to 15.26] | 21.19 [16.82 to 25.57]
  Week 8 | 22.36 [17.87 to 26.84] | 45.37 [40.04 to 50.70]
  Week 16 | 30.51 [25.55 to 35.47] | 54.63 [49.30 to 59.96]
  Week 24 | 29.61 [24.69 to 34.53] | 51.64 [46.29 to 56.99]

113. Secondary Outcome: Percentage of Participants With PtGA Response of Clear or Almost Clear During CP-690,550 Re-Treatment (Period C) Among Participants Who Had a PtGA of Mild, Moderate or Severe During CP-690,550 Treatment Withdrawal (Period B)
Description: as for outcome 112
Time Frame: Baseline and Weeks 4, 8, and 16 (Period C)
Population: FAS-C
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 14 | 63 | 17 | 100
percentage of participants
  Baseline (n=14,63,17,100) | 14.29 [0.00 to 32.62] | 6.35 [0.33 to 12.37] | 23.53 [3.37 to 43.69] | 8.00 [2.68 to 13.32]
  Week 4 (n=14,63,17,100) | 21.43 [0.00 to 42.92] | 19.05 [9.35 to 28.74] | 35.29 [12.58 to 58.01] | 42.00 [32.33 to 51.67]
  Week 8 (n=14,63,17,100) | 21.43 [0.00 to 42.92] | 34.92 [23.15 to 46.69] | 41.18 [17.78 to 64.57] | 54.00 [44.23 to 63.77]
  Week 16 (n=14,63,17,100) | 21.43 [0.00 to 42.92] | 41.27 [29.11 to 53.43] | 58.82 [35.43 to 82.22] | 53.00 [43.22 to 62.78]

114. Secondary Outcome: Percentage of Participants Maintaining PtGA Response of Clear or Almost Clear During the Double-Blind Treatment Withdrawal (Period B) Among Participants Who Had a Response of Clear or Almost Clear at Beginning of Period B
Description: as for outcome 112
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: FAS-B
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 19 | 66 | 39 | 107
percentage of participants
  Week 4 | 94.7 [68.1 to 99.2] | 50.7 [38.0 to 62.0] | 82.0 [65.9 to 91.0] | 55.5 [45.5 to 64.4]
  Week 8 | 89.2 [63.1 to 97.2] | 32.8 [21.6 to 44.4] | 71.4 [54.3 to 83.0] | 33.3 [24.5 to 42.4]
  Week 12 | 77.3 [50.1 to 90.8] | 21.3 [12.2 to 32.2] | 68.8 [51.6 to 80.9] | 24.2 [16.4 to 32.9]
  Week 16 | 77.3 [50.1 to 90.8] | 16.0 [7.5 to 27.3] | 0.0 [NA to NA] — 95% CI could not be estimated due to censoring. | 0.0 [NA to NA] — 95% CI could not be estimated due to censoring.

115. Secondary Outcome: Mean EuroQol 5 Dimensions (EQ-5D) Health State Profile Utility Score and VAS Scores During the Initial CP-690,550 Treatment Period (Period A)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: FAS-A; n=number of participants with an observation.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 329 | 332
score on a scale
  Utility Score, Baseline (n=329,332) | 0.7 (0.0) | 0.7 (0.0)
  Utility Score, Week 24 (n=270,272) | 0.8 (0.0) | 0.9 (0.0)
  VAS, Baseline (n=329,332) | 69.9 (1.3) | 70.6 (1.3)
  VAS, Week 24 (n=269,274) | 75.6 (1.2) | 80.3 (1.0)

116. Secondary Outcome: Mean EQ-5D Utility Score and VAS Scores During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 115
Time Frame: Baseline and Week 56 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
score on a scale
  Baseline Utility Score (n=27,75,42,120) | 0.8 (0.0) | 0.8 (0.0) | 0.9 (0.0) | 0.8 (0.0)
  Week 56 Utility Score (n=22,65,34,96) | 0.9 (0.0) | 0.9 (0.0) | 0.9 (0.0) | 0.9 (0.0)
  Baseline VAS (n=27,75,42,120) | 79.6 (3.4) | 76.5 (2.2) | 76.8 (3.5) | 75.3 (1.8)
  Week 56 VAS (n=22,65,34,96) | 82.0 (2.5) | 82.3 (1.7) | 82.7 (2.7) | 83.8 (1.2)

117. Secondary Outcome: Mean Change From Baseline-A in EQ-5D Utility Score and VAS Scores During the Initial CP-690,550 Treatment Period (Period A)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state. Baseline-A defined as the last observation up to first dosing date in Period A.
Time Frame: Week 24 (Period A)
Population: FAS-A; n=number of participants with an observation
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 269 | 271
scores on a scale
  Week 24 Utility Score (n=269,269) | 0.1 (0.0) | 0.2 (0.0)
  Week 24 VAS (n=268, 271) | 5.3 (1.5) | 9.3 (1.4)

118. Secondary Outcome: Mean Change From Baseline-C in EQ-5D Utility Score and VAS Scores During CP-690,550 Re-Treatment (Period C)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state. Baseline-C defined as the last observation up to first dosing date in Period C.
Time Frame: Week 56 (Period C)
Population: FAS-C
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 22 | 65 | 34 | 96
scores on a scale
  Week 56 Utility Score | 0.0 (0.0) | 0.1 (0.0) | -0.0 (0.0) | 0.1 (0.0)
  Week 56 Visual Analogue Score | -1.0 (1.6) | 4.2 (1.7) | 6.4 (3.8) | 6.4 (1.5)

119. Secondary Outcome: Mean EQ-5D Domain Scores During the Initial CP-690,550 Treatment Period (Period A)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. The score for each of the 5 dimensions can range from 1 to 3; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed").
Time Frame: Baseline and Week 24 (Period A)
Population: FAS-A; n=number of participants with an observation.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 329 | 332
score on a scale
  Mobility, Baseline (n=329,332) | 1.3 (0.0) | 1.3 (0.0)
  Mobility, Week 24 (n=270,274) | 1.2 (0.0) | 1.2 (0.0)
  Self-Care, Baseline (n=330,332) | 1.1 (0.0) | 1.1 (0.0)
  Self-Care, Week 24 (n=270,272) | 1.1 (0.0) | 1.0 (0.0)
  Usual Activities Baseline (n=330,332) | 1.4 (0.0) | 1.4 (0.0)
  Usual Activities Week 24 (n=270,273) | 1.2 (0.0) | 1.1 (0.0)
  Pain/Discomfort Baseline (n=330,332) | 1.8 (0.0) | 1.9 (0.0)
  Pain/Discomfort Week 24 (n=270,274) | 1.5 (0.0) | 1.4 (0.0)
  Anxiety/Depression Baseline (n=330,332) | 1.4 (0.0) | 1.4 (0.0)
  Anxiety/Depression Week 24 (n=270,274) | 1.3 (0.0) | 1.3 (0.0)

120. Secondary Outcome: Mean EQ-5D Domain Scores During CP-690,550 Re-Treatment (Period C)
Description: as for outcome 119
Time Frame: Baseline and Week 56 (Period C)
Population: FAS-C; n equals the number of participants with an observation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
score on a scale
  Baseline Mobility (n=27,75,42,120) | 1.2 (0.1) | 1.2 (0.0) | 1.1 (0.1) | 1.2 (0.0)
  Week 56 Mobility (n=22,65,34,96) | 1.2 (0.1) | 1.1 (0.0) | 1.1 (0.1) | 1.2 (0.0)
  Baseline Self-Care (n=27,75,42,120) | 1.1 (0.1) | 1.1 (0.0) | 1.0 (0.0) | 1.1 (0.0)
  Week 56 Self-Care (n=22,65,34,96) | 1.1 (0.1) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0)
  Baseline Usual Activities (n=27,75,42,120) | 1.3 (0.1) | 1.2 (0.1) | 1.1 (0.1) | 1.3 (0.0)
  Week 56 Usual Activities (n=22,65,34,96) | 1.1 (0.1) | 1.1 (0.0) | 1.1 (0.1) | 1.1 (0.0)
  Baseline Pain/Discomfort (n=27,75,42,120) | 1.5 (0.1) | 1.6 (0.1) | 1.3 (0.1) | 1.7 (0.1)
  Week 56 Pain/Discomfort (n=22,65,34,96) | 1.4 (0.1) | 1.5 (0.1) | 1.3 (0.1) | 1.4 (0.1)
  Baseline Anxiety/Depression (n=27,75,42,120) | 1.3 (0.1) | 1.3 (0.1) | 1.2 (0.1) | 1.3 (0.0)
  Week 56 Anxiety/Depression (n=22,65,34,96) | 1.2 (0.1) | 1.3 (0.1) | 1.2 (0.1) | 1.2 (0.0)

121. Secondary Outcome: Mean Change From Baseline-A in EQ-5D Domain Scores During the Initial CP-690,550 Treatment Period (Period A)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. The score for each of the 5 dimensions can range from 1 to 3; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Baseline-A defined as the last observation up to first dosing date in Period A.
Time Frame: Week 24 (Period A)
Population: FAS-A; n=number of participants with an observation
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 269 | 271
scores on a scale
  Mobility (n=269,271) | -0.1 (0.0) | -0.1 (0.0)
  Self-Care (n=270,269) | 0.0 (0.0) | -0.1 (0.0)
  Usual Activities (n=270,270) | -0.1 (0.0) | -0.2 (0.0)
  Pain / Discomfort (n=270,271) | -0.3 (0.0) | -0.5 (0.0)
  Anxiety / Depression (n=270,271) | -0.1 (0.0) | -0.2 (0.0)

122. Secondary Outcome: Mean Change From Baseline-C in EQ-5D Domain Scores During CP-690,550 Re-Treatment (Period C)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. The score for each of the 5 dimensions can range from 1 to 3; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Baseline-C defined as the last observation up to first dosing date in Period C.
Time Frame: Week 56 (Period C)
Population: FAS-C
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 22 | 65 | 34 | 96
scores on a scale
  Mobility | 0.0 (0.1) | -0.0 (0.0) | 0.0 (0.0) | -0.0 (0.0)
  Self-Care | 0.0 (0.1) | -0.1 (0.0) | 0.0 (0.0) | -0.1 (0.0)
  Usual Activities | -0.0 (0.0) | -0.1 (0.0) | 0.0 (0.0) | -0.2 (0.0)
  Pain / Discomfort | 0.0 (0.1) | -0.1 (0.1) | 0.0 (0.1) | -0.3 (0.1)
  Anxiety / Depression | -0.1 (0.1) | -0.1 (0.1) | 0.1 (0.1) | -0.1 (0.1)

123. Secondary Outcome: Percentage of Participants With Pustular, Erythrodermic, or Guttate Psoriasis During the Initial CP-690,550 Treatment (Period A)
Time Frame: Weeks 4, 8, 16, and 24 (Period A)
Population: Safety-A
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A)
Number analyzed (Participants) | 331 | 335
percentage of participants
  Erythrodermic psoriasis | 0.0 | 0.6
  Guttate psoriasis | 0.0 | 0.0
  Pustular psoriasis | 0.0 | 0.3

124. Secondary Outcome: Percentage of Participants With Pustular, Erythrodermic, or Guttate Psoriasis During Double-Blind Treatment Withdrawal (Period B)
Time Frame: Weeks 4, 8, 12, and 16 (Period B)
Population: Safety-B
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID (Period B) | Placebo for 5 mg CP-690,550 BID (Period B) | CP-690,550 10 mg BID (Period B) | Placebo for 10 mg CP-690,550 BID (Period B)
Number analyzed (Participants) | 31 | 82 | 45 | 133
percentage of participants
  Erythrodermic psoriasis | 0.0 | 0.0 | 0.0 | 0.0
  Guttate psoriasis | 0.0 | 0.0 | 0.0 | 0.8
  Pustular psoriasis | 0.0 | 0.0 | 0.0 | 0.0

125. Secondary Outcome: Percentage of Participants With Pustular, Erythrodermic, or Guttate Psoriasis During CP-690,550 Re-Treatment (Period C)
Time Frame: Weeks 4, 8, and 16 (Period C)
Population: Safety-C
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID / CP-690,550 5 mg BID | Placebo BID / CP-690,550 5 mg BID | CP-690,550 10 mg BID / CP-690,550 10 mg BID | Placebo BID / CP-690,550 10 mg BID
Number analyzed (Participants) | 27 | 75 | 42 | 120
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- CP-690,550 5 mg/CP-690,550 5 mg/CP-690,550 5 mg: Participants received CP-690,550 5 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by CP-690,550 5 mg tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 5 mg for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- CP-690,550 5 mg/Placebo/CP-690,550 5 mg: Participants received CP-690,550 5 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 5 mg for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- CP-690,550 10 mg/CP-690,550 10 mg/CP-690,550 10 mg: Participants received CP-690,550 10 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by CP-690,550 10 mg tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 10 mg for up to 28 weeks in Period C (Double-Blind Re-Treatment)
- CP-690,550 10 mg / Placebo / CP-690,550 10 mg: Participants received CP-690,550 10 mg tablets orally BID for 24 weeks in Period A (Initial Treatment) followed by placebo tablets orally BID for 4, 8, 12 or 16 weeks during Period B (Double-Blind Treatment Withdrawal) followed by CP-690,550 10 mg for up to 28 weeks in Period C (Double-Blind Re-Treatment)
Arm/Group | CP-690,550 5 mg BID (Period A) | CP-690,550 10 mg BID (Period A) | CP-690,550 5 mg/CP-690,550 5 mg/CP-690,550 5 mg | CP-690,550 5 mg/Placebo/CP-690,550 5 mg | CP-690,550 10 mg/CP-690,550 10 mg/CP-690,550 10 mg | CP-690,550 10 mg / Placebo / CP-690,550 10 mg
Serious Adverse Events (participants affected / at risk) | 6/218 | 9/157 | 1/31 | 3/82 | 4/45 | 4/133
Other Adverse Events (participants affected / at risk) | 101/218 | 94/157 | 25/31 | 65/82 | 41/45 | 108/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg BID (Period A) (N=218) | CP-690,550 10 mg BID (Period A) (N=157) | CP-690,550 5 mg/CP-690,550 5 mg/CP-690,550 5 mg (N=31) | CP-690,550 5 mg/Placebo/CP-690,550 5 mg (N=82) | CP-690,550 10 mg/CP-690,550 10 mg/CP-690,550 10 mg (N=45) | CP-690,550 10 mg / Placebo / CP-690,550 10 mg (N=133)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Drug ineffective (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster multi-dermatomal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Pregnancy test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypomania (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg BID (Period A) (N=218) | CP-690,550 10 mg BID (Period A) (N=157) | CP-690,550 5 mg/CP-690,550 5 mg/CP-690,550 5 mg (N=31) | CP-690,550 5 mg/Placebo/CP-690,550 5 mg (N=82) | CP-690,550 10 mg/CP-690,550 10 mg/CP-690,550 10 mg (N=45) | CP-690,550 10 mg / Placebo / CP-690,550 10 mg (N=133)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 1 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 1 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 5 | 2 | 0 | 5 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 5 | 0 | 3 | 4 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 0 | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 1
Nausea (Gastrointestinal disorders) | 10 | 5 | 1 | 3 | 2 | 6
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 0 | 1 | 2 | 2
Fatigue (General disorders) | 2 | 3 | 1 | 2 | 0 | 3
Influenza like illness (General disorders) | 1 | 3 | 1 | 2 | 0 | 3
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 2 | 1 | 2 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 3 | 0 | 0 | 1 | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3 | 0 | 2 | 2 | 10
Ear infection (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0
Folliculitis (Infections and infestations) | 1 | 2 | 1 | 1 | 0 | 7
Gastroenteritis viral (Infections and infestations) | 2 | 4 | 0 | 1 | 1 | 4
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 3
Hordeolum (Infections and infestations) | 0 | 2 | 0 | 0 | 2 | 1
Influenza (Infections and infestations) | 1 | 4 | 2 | 6 | 1 | 3
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 18 | 15 | 3 | 15 | 8 | 23
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 2 | 0 | 2 | 3 | 4
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 3 | 1 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 2 | 2 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 7 | 2 | 14 | 5 | 18
Urinary tract infection (Infections and infestations) | 7 | 5 | 1 | 6 | 4 | 9
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 2 | 1 | 2 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 1 | 2
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 2 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 1 | 3
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3 | 2 | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1 | 2 | 0 | 0
Bacterial test positive (Investigations) | 1 | 0 | 0 | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 3 | 3 | 0 | 2 | 4 | 4
Blood creatine phosphokinase increased (Investigations) | 10 | 5 | 1 | 6 | 12 | 14
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Blood glucose fluctuation (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 3 | 1 | 2 | 2 | 3
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 2 | 0 | 1 | 2 | 5
Haemoglobin decreased (Investigations) | 2 | 2 | 0 | 1 | 1 | 1
Low density lipoprotein increased (Investigations) | 0 | 1 | 0 | 1 | 4 | 1
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 3 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 7 | 1 | 0 | 4 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 5 | 1 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 2 | 0 | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 0 | 0 | 1 | 3 | 6
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 3 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tongue neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 2 | 2 | 5
Headache (Nervous system disorders) | 6 | 6 | 2 | 5 | 4 | 17
Paraesthesia (Nervous system disorders) | 1 | 2 | 1 | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 2 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 3 | 0 | 0 | 1 | 2
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 3 | 1 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 5 | 1 | 3 | 2
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 1 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2 | 0 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 6 | 0 | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 5 | 5 | 1 | 5 | 2 | 7
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Clinical interpretation regarding sub-phenotypes of psoriasis (e.g., scalp psoriasis) should not be made based on the reported assessments by body regions. For example, the body region of head does not reflect solely scalp psoriasis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.